#### **Statistical Analysis Plan**

**Study ID: 207497** 

Official Title of Study: Reporting and Analysis Plan for A Phase I/II, Open-label, Dose Escalation and Expansion Study to Evaluate Safety, Tolerability, and Clinical Activity of the Antibody-Drug Conjugate GSK2857916 Administered in Combination with Lenalidomide Plus Dexamethasone (Arm A), or Bortezomib Plus Dexamethasone (Arm B) in Participants with Relapsed /Refractory Multiple Myeloma – (DREAMM 6)

**NCT ID**: NCT03544281

Date of Document: 25 April 2023

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A Phase I/II, Open-label, Dose Escalation and Expansion Study to Evaluate Safety, Tolerability, and Clinical Activity of the Antibody-Drug Conjugate GSK2857916 Administered in Combination with Lenalidomide Plus Dexamethasone (Arm A), or Bortezomib Plus Dexamethasone (Arm B) in Participants with Relapsed / Refractory Multiple Myeloma – (DREAMM 6) |
|---|---|---|
| <b>Compound Number</b> | : | GSK2857916 |
| Effective Date | : | Refer to Document Date |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 207497 (DREAMM 6) [GSK Document No. TMF-14624358, Dated: 2022-JUN-30].
- This RAP is intended to describe the efficacy, safety, pharmacokinetic (PK), pharmacodynamic (PD), and patient reported outcome (PRO) analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Interim Analysis (IA) and Statistical Analysis Complete (SAC) deliverables.

#### RAP Author(s):

| Author | Approval Method |
|---|---|
| PPD Statistics Leader (Oncology, Clinical Statistics) | Email |
| PPD (Clinical Pharmacology Modeling & Simulations Complimentary Worker, Accuro for GSK) | Email |

Copyright 2023 the GSK group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Approvals**

| Reviewers | Approval Method |
|---|---|
| PPD | Email |
| Principal Programmer/Analyst (Oncology, Clinical Programming) | Ellian |
| PPD | E |
| , Clinical Development | Email |
| PPD | E |
| Clinical Scientist (Oncology, Clinical Development) | Email |
| PPD | Email |
| PPD , SMG Pharma Safety (SERM Dev Oncology Scientists) | Email |
| PPD | Email |
| PPD (R&D GCSD) | Ellian |
| PPD | |
| PPD , PCO Strategy and Engagement | Email |
| (Development – Global Med – VEO – VE Oncology) | |
| PPD | |
| PPD (Dev-GCO-Rx GCD-Medical | Email |
| Writing & Clin Submission) | |
| PPD | |
| PPD – Precision Medicine and Companion Diagnostics, | Email |
| Oncology-EMU-MTT Precision Med & Comp Diagnostics | |

# Clinical Statistics and Clinical Programming Line Approvals (Method: Veeva Vault TMF eSignature):



## **TABLE OF CONTENTS**

| | | PAGE |
|----|----------------------------------------------------------------|------|
| 1. | INTRODUCTION | 7 |
| | 1.1. RAP Amendments | |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 11 |
| | 2.1. Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. Study Objective(s) and Endpoint(s) | |
| | 2.3. Study Design | |
| | 2.3.1. Overall Design | 15 |
| | 2.4. Statistical Hypotheses / Statistical Analyses | 20 |
| | 2.4.1. Arm A - Belantamab Mafodotin with Len/Dex | 20 |
| | 2.4.2. Arm B - Belantamab Mafodotin with Bor/Dex | 20 |
| 3. | PLANNED ANALYSES | 21 |
| | 3.1. Interim Analyses | |
| | 3.1.1. Arm A – Belantamab Mafodotin with Len/Dex | |
| | 3.1.2. Arm B- Belantamab Mafodotin with Bor/Dex | 27 |
| | 3.2. Final Analyses | 31 |
| 4. | ANALYSIS POPULATIONS | 32 |
| | 4.1. Protocol Deviations | |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONVENTIONS | |
| | 5.1. Study Treatment & Sub-group Display Descriptors | |
| | 5.2. Baseline Definitions | |
| | 5.3. Examination of Covariates, Other Strata and Subgroups | |
| | 5.3.1. Examination of Subgroups | 35 |
| | Conventions | 36 |
| | Conventions | |
| 6. | STUDY POPULATION ANALYSES | 37 |
| | 6.1. Overview of Planned Study Population Analyses | 37 |
| | 6.2. Disposition of Participants | 37 |
| | 6.3. Demographic and Baseline Characteristics | 37 |
| | 6.4. Treatment Compliance | 38 |
| | 6.5. Extent of Exposure | |
| | 6.6. Concomitant Medications | 40 |
| 7. | EFFICACY ANALYSES | 42 |
| | 7.1. Primary Efficacy Analyses | 42 |
| | 7.1.1. Endpoint/Variables | 42 |
| | 7.1.2. Summary Measure | |
| | 7.1.3. Population of Interest | |
| _ | 7.1.4. Statistical Analyses / Methods | 45 |


| 8. | SAFE | TY ANALYSES | 51 |
|---|---|---|---|
| | 8.1. | Adverse Events Analyses | |
| | 8.2. | Adverse Events of Special Interest Analyses | |
| | | 8.2.1. Belantamab Mafodotin | |
| | | 8.2.2. Corneal events (GSK scale) | 55 |
| | | 8.2.3. Eye Disorder (CTCAE) | |
| | 8.3. | Deaths and Serious Adverse Events | |
| | 8.4. | Adverse Events Leading to Discontinuation and Dose Modification | 57 |
| | 8.5. | Ocular findings from ophthalmic exam | 57 |
| | 8.6. | Pregnancies | 58 |
| | 8.7. | Clinical Laboratory Analyses | |
| | 8.8. | Other Safety Analyses | |
| | | 8.8.1. ECG | 59 |
| | | 8.8.2. Anti-Drug Antibody Analyses | |
| | | 8.8.3. Profile Plot | 59 |
| _ | | | |
| 9. | | MACOKINETIC ANALYSES | |
| | 9.1. | Drug Concentration Measures | |
| | 9.2. | Derived Pharmacokinetic Parameters | |
| | | 9.2.1. Belantamab Mafodotin, Total mAb, and Cys-mcMMAF | |
| | 0.0 | 9.2.2. Lenalidomide and Bortezomib | |
| | 9.3. | Summary Measure | |
| | 9.4. | Population of Interest | |
| | 9.5. | Statistical Analyses / Methods | 63 |
| 10 | DHAR | MACOKINETIC AND PHARMACODYNAMIC ANALYSES | 64 |
| 10. | 10.1. | | |
| | 10.1. | Exposure-response for Emeday and Oalety Emapoints | 04 |
| 11 | POPU | LATION PHARMACOKINETIC (POPPK) ANALYSIS | 64 |
| • • • • | | | 0 . |
| CI | | | |
| 13. | PATIE | NT REPORTED OUTCOMES ANALYSES | |
| | 13.1. | Compliance of PRO-CTCAE, OSDI, and EORTC QLQ-C30 | 67 |
| | 13.2. | Patient Reported Outcome Version of the Common Term Criteria | |
| | | for Adverse Events (PRO-CTCAE) | |
| | 13.3. | Visual Function Questionnaires | 68 |
| | | 13.3.1. National Eye Institute Function Questionnaire-25 (NEI- | |
| | | VFQ-25) | |
| | | 13.3.2. Ocular Surface Disease Index | |
| | 13.4. | Value Evidence and Outcome | 69 |
| | | 13.4.1. European Organization for Research and Treatment of | |
| | | Cancer Quality of Life Questionnaire 30-item Core module | |
| | | (EORTC QLQ-C30) | 69 |

| | | 13.4.2. | European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 20-item Multiple Myeloma module (EORTC QLQ-MY20) | 70 |
|---|---|---|---|---|
| 11 | DEEE | DENICES | | |
| 14. | REFER | RENCES. | | / 1 |
| 15. | APPE | NDICES | | 73 |
| | 15.1. | Appendix | ( 1: Assessment Windows | 73 |
| | 15.2. | Appendix | c 2: Study Phases and Treatment Emergent Adverse | |
| | | 15.2.1. | | |
| | | 15.2.2. | | 75 |
| | | 15.2.3. | Treatment Emergent and On-treatment Flag for Adverse | |
| | | | Events | 75 |
| | 15.3. | | 3: Data Display Standards & Handling Conventions | |
| | | 15.3.1. | Reporting Process | |
| | | 15.3.2. | Reporting Standards | |
| | | 15.3.3. | Reporting Standards for Pharmacokinetic Data | 78 |
| | | 15.3.4. | Extended Loss to Follow-up or Extended Time without an | 70 |
| | | 15.3.5. | Additional Cuidance on Crading Record on Changes in | 79 |
| | | 15.5.5. | Additional Guidance on Grading Based on Changes in Visual Acuity | 90 |
| | 15.4. | Annendi | ∨isual Actity | |
| | 10.4. | 15.4.1. | General | |
| | | 15.4.2. | Study Population | |
| | | 15.4.3. | Safety | |
| | | 15.4.4. | Biomarker and/or Pharmacodynamic Data | 83 |
| | 15.5. | | s 5: Reporting Standards for Missing Data | |
| | | | Premature Withdrawals | |
| | | 15.5.2. | | |
| | 15.6. | Appendix | c 6: Values of Potential Clinical Importance | |
| | 15.7. | Appendix | د 7: Pharmacokinetic / Pharmacodynamic Analyses | 89 |
| | | 15.7.1. | · | |
| | | | Specification | |
| | | | Pharmacokinetic / Pharmacodynamic Methodology | |
| | 15.8. | | κ 8: Population Pharmacokinetic (PopPK) Analyses | |
| | | 15.8.1. | Systems | |
| | | 15.8.2. | Data Assembly | |
| | | 15.8.3. | Model Development | |
| | 45.0 | 15.8.4. | Model Qualification | |
| | 15.9. | | ( 9: Patient Reported Outcomes | |
| | | | EORTC QLQ-C30 | |
| | | 15.9.2.<br>15.9.3. | NEI-VFQ-25 | |
| | 15 10 | | ( 10: COVID-19 Impact | |
| | | | (11: Abbreviations & Trademarks | |
| | 10.11. | | Abbreviations | |
| | | | Trademarks | |
| | 15.12 | | 12: List of Data Displays | |
| | | | Data Display Numbering | |
| | | | Deliverables | |
| | | | Study Population Tables | |


| | 207497 |
|-----------------------------------------------------------|--------|
| 15.12.4. Efficacy Tables | 124 |
| 15.12.5. Efficacy Figures | 129 |
| 15.12.6. Safety Tables | 132 |
| 15.12.7. Safety Figures | 161 |
| 15.12.8. Pharmacokinetic Tables | 163 |
| 15.12.9. Pharmacokinetic Figures | 167 |
| 15.12.10. Biomarker Tables | 173 |
| 15.12.11.Biomarker Figures | 174 |
| 15.12.12.Patient Reported Outcomes Tables | 176 |
| 15.12.13. Patient Reported Outcomes Figures | 185 |
| 15.12.14.ICH Listings | 200 |
| 15.12.15. Non-ICH Listings | 206 |
| 15.13. Appendix 13: Example Mock Shells for Data Displays | 210 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the safety, tolerability, and efficacy analyses required for interim and final analyses and to describe the analyses to be included in the Clinical Study Report for Protocol 207497:

| Protocol Revision Chronology: | | |
|---|---|---|
| 2017N330850_00 | 2018-FEB-28 | Original |
| 2017N330850_01 | 2018-MAY-07 | Amendment 01 The protocol has been amended to include the following: additional authors were added, change in the Primary Medical Monitor, changes made in the Schedule of Activities tables, minor correction made in the participants' eligibility criteria, clarification made on dose delays of study drugs by giving examples of different scenarios, all routine and disease evaluation related blood and urine tests now will be done locally; centrally only if unable to perform locally, and administrative changes made throughout the document. |
| 2017N330850_02 | 2018-MAY-14 | Amendment 01 (republished) Republishing of protocol amendment 1 2017N330850_01. |
| 2017N330850_03 | 2019-APR-26 | Amendment 02 The protocol has been amended to change ECOG eligibility criteria in Arm A from 0-2 to 0-1, b) to include additional guidance for management of neutropenia / prophylaxis of infections to be implemented across the study on resuming Arm A and c) more stringent hematological monitoring for both Arm A and Arm B. Also, regulatory feedback encouraged generation of additional data (safety, PK, PD, clinical activity) at lower dose levels of GSK2857916 to support dose selection for future Phase 3 studies with GSK2857916 in combination with standard of care (SoC) agents. Protocol Amendment 2 also incorporates the Protocol Clarification letter (dated 28-Feb-2019) previously issued to study sites, that provided updated guidance on grading corneal events and dosing participants with GSK2857916. Administrative corrections and general program updates are also included in Amendment 2. |
| 2017N330850_04 | 2020-JUL-13 | Amendment 03 The protocol has been amended to include updated duration of contraception for female participants to align with this guidance of childbearing potential based on review of guidelines on aneugens. Additionally, upon review of safety data from Study 205678 (DREAMM-2), it was determined that ocular changes associated with belantamab mafodotin treatment were mostly limited to the corneal epithelium [GSK Document Number 2013N175128 V08, 2020]. Therefore, further collection of ocular safety |

| | | data in belantamab mafodotin studies will be focused on corneal changes. Preclinical data from xenograft mouse models and emerging clinical data from Arm A in Amendment 2 suggests greater activity of belantamab mafodotin in combination with lenalidomide. Given this, doses higher than 2.5 mg/kg of belantamab mafodotin will not be evaluated in combination with lenalidomide/ dexamethasone in Arm A in Amendment 3. Furthermore, in order to reduce increased exposure of belantamab mafodotin over time and potentially improve the benefit/risk for participants, reduced dose levels and extended dosing schedules for belantamab mafodotin will be evaluated in Amendment 3. |
|---|---|---|
| TMF-14624358 | 2022-JUN-30 | Amendment 04 |
| | | The protocol has been amended to allow continued treatment of study participants who continue to derive clinical benefit post the final analysis, update for changes made per the latest IB, match plans for final statistical analysis, and support deliverables for final CSR and to implement PACT. |

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology"

# 1.1. RAP Amendments

# **Revision chronology:**

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis Plan_Study207497_Final_V1 [18-NOV-2020] | |
| Statistical Analysis Plan RA | AP Amendment 1 [30-AUG-2021] |
| Various sections | Updated use of the word "participants" instead of "subjects," except within Appendix 12 and sections referring to the list of data displays. |
| Section 2.1 | Added activity. Added activity. Added activity. |
| Section 3.1. Interim<br>Analyses | Edited paragraph and page break formatting. |
| Section 5.1 Study<br>Treatment & Sub-group<br>Display Descriptors | Updated "Data Display" labelling, as per interim 1 review, adding combination name. |
| Section 6.3 Demographic and Baseline Characteristics | Added clarifying statements stating summaries "may be summarized." |
| | Added description of "Relative Dose Intensity" |
| Section 6.5 Extent of Exposure | Updated definition of "Duration of Delays" to account for calculation of SPLIT and STRETCH dosing schedules. |
| | Added description of "duration of follow-up" |

| RAP Section | Amendment Details |
|---|---|
| | Added wording on summarizing columns |
| Section 7.1 Primary<br>Efficacy Analyses | <ul> <li>Deleted option to create ORR display at interim, based on unconfirmed<br/>responses in certain cases. ORR at interim analyses will be analyzed<br/>based on confirmed responses if available.</li> </ul> |
| , , | Updated "Derivation of Confirmed Response", and "Assignments for Progression and Censoring Dates for Collaboration and Censoring Dates for |
| Section 7.2 Exploratory<br>Efficacy Analyses | CCI |
| Section 15.3.4 Extended<br>Loss to Follow-up or<br>Extended Time without an<br>Adequate Assessment | Clarified definitions specific to Arms A and B. |
| Section 15.4.2 Study<br>Population | Replaced "randomized" with "enrolled in study" |
| | <ul> <li>Added description of "post-interim [1]" report, and updated descriptions of<br/>Interim [2] and Interim [3] in Section 15.12.2.</li> </ul> |
| | <ul> <li>Made clarifying edits in titles/footnotes, programming notes, updates in<br/>delivery priority, and fixed typos in various displays to incorporate<br/>comments/decisions.</li> </ul> |
| | <ul> <li>Programming note to add "Relative Dose Intensity" to Table 1.042<br/>(Summary of Exposure)</li> </ul> |
| Section 15.12. Appendix | <ul> <li>Deleted tables and listings related to summarizing ORR based on<br/>unconfirmed responses in certain cases.</li> </ul> |
| 12: List of Data Displays | • Updated "Summary of Duration of Follow-up" (Tables 1.065/1.065), "Summary of Duration of Response" (Tables 2.009/2.010), "Summary of CCI (Tables 2.012/2.013), and "Summary of CCI (Tables 2.015/2.016) to be reported for both interim and SAC. |
| | <ul> <li>Added "Summary of Adverse Events" related to each specific study drug,<br/>as per ICH.</li> </ul> |
| | <ul> <li>Prioritized different displays with respect to being observed at interim and/or SAC</li> </ul> |
| Section 15.13 Appendix 13:<br>Example Mock Shells for<br>Data Displays | Made clarifying edits in title/footnote, added content, and fixed typos in various mock shells to incorporate comments from dry run reviews. |
| Statistical Analysis Plan RAP Amendment 2 [26-JUL-2022] | |
| Section 2 Summary of Key<br>Protocol Information | <ul> <li>Updated Summary of Key Protocol Information to be consistent with<br/>latest protocol amendment (Amendment 04)</li> </ul> |
| Section 2.1 Changes to the<br>Protocol Defined Statistical<br>Analysis Plan | Edited Table 1 to no longer include ccl and and ccl as they were both added to latest protocol amendment (Amendment 04). |
| Section 3.2 Primary and | Updated definition of Final Analysis to be consistent with latest protocol |

| RAP Section | Amendment Details |
|---|---|
| Final Analyses | amendment (Amendment 04) and add PACT language. |
| Section 6.5 Extent of Exposure | <ul> <li>Updated dose intensity and relative dose intensity (RDI) calculations with the following updates:</li> <li>Split lenalidomide calculations into 25 mg vs. 10 mg.</li> <li>No longer using "death date" as a potential end date.</li> <li>Separate RDI calculations into Cycle 1 and Post-Cycle 1.</li> </ul> |
| Section 7.1 Primary<br>Efficacy Analyses | Table 6: Add footnote to clarify how to handle Best Overall Response for subjects without adequate baseline data. |
| Section 7.2 Exploratory<br>Efficacy Analyses | CCI |
| Section 8 Safety Analyses | <ul> <li>Clarified the frequency and percentage of AEs (all grades) will be summarized and displayed in three ways: 1) in descending order of total incidence by PT only, 2) in descending order of total incidence by System Organ Classes (SOC) and PT, and 3) in descending order of total incidence by System Organ Classes (SOC) and PT and Maximum Grade.</li> <li>Added a section to describe Anti-Drug Antibody Analyses to be performed at final SAC.</li> </ul> |
| Section 15.5.2.1 Handling of Missing Data | Deleted statement about the storage of imputed dates. |
| Section 15.7.1 Pharmacokinetic / Pharmacodynamic Dataset Specification | Added wording to guide exposure-response analysis. |
| Section 15.11<br>Abbreviations &<br>Trademarks | Added relevant abbreviations |
| Section 15.12. Appendix 12: List of Data Displays | <ul> <li>Updated Deliveries</li> <li>Made clarifying edits in titles/footnotes, programming notes, updates in delivery priority, and fixed typos in various displays to incorporate comments/decisions.</li> </ul> |
| Statistical Analysis Plan RA | AP Amendment 3 [DD-MMM-2023] |
| Various sections | Edited grammatical errors and/or typos |
| Section 5.3.1 Examination of Subgroups | <ul> <li>Added/Edited subgroup analyses and clarified wording/categories on<br/>existing subgroups</li> </ul> |
| Section 6.2 Disposition of Participants | Edited displays being produced to understand the impact of COVID |
| Section 6.5 Extent of Exposure | Edited calculation of dose intensity and relative dose intensity of<br>Dexamethasone |
| Section 7.1.2 Summary<br>Measure | Edited wording on subgroup analyses |
| CI | |

| RAP Section | Amendment Details |
|---|---|
| Section 13.1 Compliance of PRO-CTCAE, OSDI, and EORTC QLQ-C30 | Corrected OSDI "summary" score to "total" score |
| Section 13.3.2 Ocular<br>Surface Disease Index | Edited summaries around OSDI score |
| Section 15.5.2.1 Handling of Missing and Partial Dates | Added wording under partial dates for Concomitant Medications/ Blood<br>Supportive Products |
| Section 15.12.2 | Added HDL RAPIDO deliveries |
| Section 15.12. Appendix 12: List of Data Displays | <ul> <li>Added/Edited displays, and made clarifying edits in titles/footnotes,<br/>programming notes, updates in delivery priority, and fixed typos in<br/>various displays to incorporate comments/decisions.</li> </ul> |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Overall Response Rate<br>(ORR) is defined as a<br>primary endpoint for Part 2<br>under the assessment of<br>clinical activity. | ORR will be calculated<br>for participants within<br>Part 1 and Part 2. | <ul> <li>Protocol states "Data from Part 1<br/>and Part 2 may be combined at<br/>interim, primary, and final analyses"<br/>which includes observing ORR for<br/>Parts 1 and 2.</li> </ul> |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | |
| Dose Escalation Determine safety, tolerability of belantamab mafodotin in combination with either Len/Dex (Arm A) or Bor/Dex (Arm B) to establish a recommended dose range and schedule to evaluate in Dose Expansion for participants with RRMM | Number (%) of participants with DLTs. Number (%) of participants with AEs, changes in clinical signs and laboratory parameters. |
| Dose Escalation and Expansion <sup>a</sup> Select the dose(s) and dosing schedule for further investigation based on safety and tolerability of belantamab mafodotin in combination with either Len/Dex (Arm A) or Bor/Dex (Arm B) for participants with RRMM | A comprehensive determination based on safety and SAE/AEs. |
| Dose Expansion To determine preliminary clinical activity of belantamab mafodotin in combination with either Len/Dex (Arm A) or Bor/Dex (Arm B) for participants with RRMM | A specific determination based on ORR defined as percentage (%) of participants achieving ≥PR as defined by the IMWG Uniform Response Criteria for MM [Kumar, 2016]. |
| Secondary Dose Escalation and Expansion | |
| To evaluate the pharmacokinetics profile of belantamab mafodotin when administered in combination with Len/Dex (Arm A) or Bor/Dex (Arm B) in participants with RRMM | Belantamab mafodotin PK parameters, as data permit |
| To evaluate the pharmacokinetics profile of lenalidomide when administered in combination with belantamab mafodotin and dexamethasone | Lenalidomide PK parameters, as data permit in Cycle 1 |
| To evaluate the pharmacokinetics profile of bortezomib when administered in combination with belantamab mafodotin and dexamethasone | Bortezomib PK parameters, as data permit in Cycle 1 |
| To assess anti-drug antibodies (ADAs) against belantamab mafodotin | Incidence and titers of ADAs against belantamab mafodotin pre-dose in Cycle 1 and selected subsequent cycles |
| To evaluate the effect and tolerability of belantamab mafodotin in combination with Len/Dex (Arm A) or Bor/Dex (Arm B) on symptomatic adverse events in participants with | Changes from baseline in symptoms and related impacts as measured by OSDI, NEI-VFQ-25 and PRO CTCAE |

| Objectives | Endpoints |
|---|---|
| RRMM | |
| To further characterize safety of belantamab mafodotin administered in combination with Len/Dex (Arm A) or Bor/Dex (Arm B) in participants with RRMM | Incidence of AEs, including SAEs and AEs of special interest (corneal events, thrombocytopenia and infusion related reactions). Ocular findings on ophthalmic exam |
| To evaluate the effect of belantamab mafodotin in combination with Len/Dex (Arm A) or Bor/Dex (Arm B) on health-related quality of life in participants with RRMM | Changes from baseline in health-related quality of life as measured by the EORTC QLQ-C30 and QLQ-MY20 |





Abbreviations: Len/Dex = Lenalidomide/Dexamethasone; Bor/Dex =
 Bortezomib/Dexamethasone; RRMM = Relapsed/Refractory Multiple Myeloma; DLT = Dose limiting toxicities; AE = Adverse Event; SAE = Serious Adverse Event; ORR = Overall
 Response Rate; PR = Partial Response; IMWG = International Myeloma Working Group; MM =
 Multiple myeloma; PK = Pharmacokinetic(s); OSDI = Ocular Surface Disease Index; NEI-VFQ 25 = National Eye Institute 25-item Visual Function Questionnaire; PRO CTCAE = Patient Reported Outcomes Version of the Common Term Criteria for Adverse Events; EORTC QLQ C30 = European Organization for Research and Treatment of Cancer Quality of Life
 Questionnaire 30-item Core module; QLQ-MY20 = European Organization for Research and

| Objectives | Endpoints |
|---|---|
| Treatment of Cancer Quality of Life Questionna | ire 20-item Multiple Myeloma module; ccl |
| ; VGPR = Very Good | Partial Response; BCMA = B-cell maturation |
| antigen; Cmax = Max | imum plasma concentration; AUC = Area under |
| the concentration time curve | |

a. Data from the both the Escalation and Expansion cohorts will be used to evaluate this composite endpoint.

# 2.3. Study Design

#### 2.3.1. Overall Design

This is a Phase I/II, open-label, dose escalation and expansion study to select the dose and dosing schedule of belantamab mafodotin when given in combination with Len/Dex (Arm A) on a 28-day cycle, or with Bor/Dex (Arm B) on a 21-day cycle, and to evaluate safety and clinical activity of the combination treatments in participants with RRMM. The study will consist of two parts.

**Part 1** is a dose escalation phase to evaluate the safety and tolerability of belantamab mafodotin in combination with two SoC regimens: Arm A – belantamab mafodotin with Len/Dex, and Arm B – belantamab mafodotin with Bor/Dex.

**Part 2** is a dose expansion phase to further evaluate the safety and clinical activity of belantamab mafodotin in combination with Len/Dex (Arm A) and Bor/Dex (Arm B).

#### 2.3.1.1. Arm A - Belantamab Mafodotin with Len/Dex



- Belantamab mafodotin (GSK2857916) SINGLE = full assigned dose of belantamab mafodotin administered on Day 1 of any 28-day cycle.
- b. Lenalidomide (25 mg on Days 1-21) + Dexamethasone (40 mg on Days 1, 8, 15, and 22) of any 28-day cycle.
- c. Belantamab mafodotin 2.5 mg/kg SPLIT= 1.25 mg/kg on Day 1 and 1.25 mg/kg on Day 8 of any 28-day cycle.
- d. \*Belantamab mafodotin 1.9 mg/kg STRETCH = belantamab mafodotin 1.9 mg/kg dose administered on Day 1 of alternate 28-day cycles i.e., Q8W (C1, C3, C5, C7 and so on)- this cohort may be evaluated if emerging data suggests that this schedule may further optimize the tolerability or offers an improved benefit/risk profile.

All participants will be operated under Amendment 03.

Note: Combination therapy continued until PD, death, intolerable toxicity, consent withdrawn. Cohorts followed up for and DE = Dose Escalation decision.

# Population: Adult participants with RRMM, who have undergone stem cell transplant (SCT), or are considered transplant ineligible, and who have been previously treated with at least 1 prior line of therapy, and who have documented evidence of disease progression during or after their most recent therapy. Objective: Part 1 is a dose escalation phase to evaluate the safety and tolerability of belantamab mafodotin in combination with Len/Dex. Part 2 is a dose expansion phase to further evaluate the safety and clinical activity of belantamab mafodotin in combination with Len/Dex.

#### Dosing

- **SINGLE** Dosing Schedule: belantamab mafodotin will be administered as a SINGLE full dose on Day 1 of each 28-day cycle.
- **SPLIT** Dosing Schedule: belantamab mafodotin will be split into two equal halves and each half dose will be administered on Day 1 and Day 8 of each 28-day cycle.
- STRETCH Dosing Schedule: A STRETCH dosing schedule for the 1.9 mg/kg dose level
  might be considered for Arm A if emerging data suggests that this schedule may further
  optimize the tolerability or offers an improved benefit/risk profile. In STRETCH schedule,
  belantamab mafodotin will be administered on Day 1 of alternate 28-day cycles with any 2
  consecutive planned belantamab mafodotin doses at least 56 (±3) days apart. The
  treatment cycle duration will remain at 28 days (4 weeks).
- Summary of Treatment Regimens and Schedules for Len/Dex are provided in Table 18 of the Protocol (Version: GSK Document Number TMF-14624358).

# Time & Events

Refer to Section 3 of Protocol – Schedule of Activities (Version: GSK Document Number TMF-14624358)

| Overview of St | udy Design and Key Features |
|---|---|
| Treatment Assignment | This is a non-randomized, double-arm, open label, two-part study |
| Interim<br>Analysis | Part 1: Dose Escalation No formal interim analysis is planned for Part 1. Data will be reviewed through data visualization tools to inform dose escalation decisions. The modified Toxicity Probability Interval (mTPI) design will be utilized to guide dose escalation/de-escalation decisions. mTPI is explained in Section 3.1.1.1. |
| | Part 2: Dose Expansion An interim analysis may be conducted when the last participant within each arm is followed for at least 1 cycle to evaluate safety, efficacy, and PK profiles at each dose level. Following the interim analysis, additional analyses may be performed to continue to evaluate safety, efficacy, and PK profiles at each dose level, prior to the primary and final analyses. If any dose level is not enrolled due to safety concerns, it will not be included in the interim or final analyses. Additionally, if enrollment is stopped within a dose group, data may be analyzed for participants within the dose group who take at least 1 dose of any study treatment. |
| | Continuous monitoring will be conducted for Part 2 starting from when 5 participants are dosed at each dose level within each arm. The observed number of participants permanently discontinuing study treatment within the first two cycles due to AE related to belantamab mafodotin will be compared against the safety stopping rule in Table 30 of the Protocol (Version: GSK Document Number TMF-14624358). Enrollment may stop if the safety stopping rule is met based on totality of safety data. For example, if 4 or more out of 5 participants permanently discontinued study treatment within the first 2 cycles due to AE related to belantamab mafodotin, enrollment may stop after review of all safety data; otherwise, enrollment will continue. |

#### 2.3.1.2. Arm B - Belantamab Mafodotin with Bor/Dex

#### Overview of Study Design and Key Features Arm B: Belantamab Mafodotin with Bortezomib/ Dexamethasone Part 1 Part 2 Belantamab Mafodotin 2.5 mg/kg SINGLE<sup>a</sup> 3.4 mg/kg SINGLEa + DE + Bor/Dexb [n ≤ 12] Bor/Dexb Belantamab Mafodotin 2.5 mg/kg SPLIT<sup>c</sup> + Bor/Dex<sup>b</sup> [n ≤ 12] Belantamab Mafodotir 2.5 mg/kg SINGLE<sup>a</sup> + Bor/Dex<sup>b</sup> Belantamab Mafodotin 3.4 mg/kg SINGLE<sup>a</sup> + Bor/Dex<sup>b</sup> [n ≤ 9] Belantamab Mafodotin 3.4 mg/kg SPLIT<sup>o</sup> + Bor/Dex<sup>b</sup> [n ≤ 12] Belantamab Mafodotin 2.5 mg/kg STRETCHe + Bor/Dexb [n ≤ 12#] Belantamab Mafodotin S/D STRETCHf + Bor/Dex<sup>b</sup> [n ≤ 12#] Belantamab Mafodotin 1.9 mg/kg SINGLE<sup>a</sup> + Bor/Dex<sup>b</sup> [n ≤ 12#] Belantamab Mafodotin 1.9 mg/kg STRETCHe + Bor/Dexb [n ≤ 12#] Belantamab mafodotin (GSK2857916) **SINGLE** = full assigned dose of belantamab mafodotin (1.9 mg/kg, 2.5 mg/kg, or 3.4 mg/kg) administered on Day 1 of any 21-day cycle. Bortezomib (1.3 mg/m<sup>2</sup> on Days 1, 4, 8, and 11) + Dexamethasone (20 mg on Days 1, 2, 4, 5, 8, 9, 11, and 12) of any 21-day cycle. Belantamab mafodotin 2.5 mg/kg SPLIT= 1.25 mg/kg on Day 1 and 1.25 mg/kg on Day 8 of any 21-day cycle. Belantamab mafodotin 3.4 mg/kg SPLIT= 1.7 mg/kg on Day 1 and 1.7 mg/kg on Day 8 of any 21-day cycle.

- e. Belantamab mafodotin **STRETCH**= belantamab mafodotin 1.9 mg/kg or 2.5 mg/kg dose administered on Day 1 of alternate 21-day cycles i.e., Q6W (C1, C3, C5, C7 and so on).
- f. Belantamab mafodotin **Step-Down (S/D) STRETCH** = belantamab mafodotin 2.5 mg/kg dose at C1D1 followed by 1.9 mg/kg step-down dose on Day 1 of alternate 21-day cycles C3 onwards (C3, C5, C7, and so on).

All participants will be operated under Amendment 03.

#New cohorts in Amendment 3.

Note: Combination therapy continued for up to 8 combination cycles; belantamab mafodotin further continued until PD, death, intolerable toxicity, consent withdrawn. Coborts followed up for walk and walk

#### death, intolerable toxicity, consent withdrawn. Cohorts followed up for and and DE=Dose Escalation decision; ; PD=Progressive Disease; CCI S/D=Stepdown. Design Population: Adult participants with RRMM, who have undergone stem cell transplant **Features** (SCT), or are considered transplant ineligible, and who have been previously treated with at least 1 prior line of therapy, and who have documented evidence of disease progression during or after their most recent therapy. Objective: Part 1 is a dose escalation phase to evaluate the safety and tolerability of belantamab mafodotin in combination with Bor/Dex. Part 2 is a dose expansion phase to further evaluate the safety and clinical activity of belantamab mafodotin in combination with Dosing **SINGLE** Dosing Schedule: belantamab mafodotin will be administered as a SINGLE full dose on Day 1 of each 21-day cycle. **SPLIT** Dosing Schedule: belantamab mafodotin will be split into two equal halves and each half dose will be administered on Day 1 and Day 8 of each 21-day cycle.

| Overview of St | udy Design and Key Features |
|---|---|
| | <ul> <li>STRETCH Dosing Schedule: belantamab mafodotin will be administered on Day 1 of alternate cycles with any two consecutive planned doses at least 42 (±3) days apart. The treatment cycle duration will remain at 21 days (3 weeks).</li> <li>Step-Down (S/D) STRETCH Dosing Schedule: belantamab mafodotin will be administered as a full 2.5 mg/kg dose on Day 1 of Cycle 1 followed by subsequent planned doses of 1.9 mg/kg S/D dose starting on Day 1 of alternate 21-day cycles (C3, C5, C7, and so on) with any two consecutive planned doses at least 42 (±3) days apart. The treatment cycle duration will remain at 21 days (3 weeks).</li> </ul> |
| | Summary of Treatment Regimens and Schedules for Bor/Dex are provided in Table 18 of the Protocol (Version: GSK Document Number TMF-14624358). |
| Time & Events | <ul> <li>Refer to Section 3 of Protocol – Schedule of Activities (Version: GSK Document Number<br/>TMF-14624358)</li> </ul> |
| Treatment Assignment | This is a non-randomized, double-arm, open label, two-part study |
| Interim<br>Analysis | Part 1: Dose Escalation No formal interim analysis is planned for Part 1. Data will be reviewed through data visualization tools to inform dose escalation decisions. The modified Toxicity Probability Interval (mTPI) design will be utilized to guide dose escalation/deescalation decisions. mTPI is explained in Section 3.1.1.1. |
| | Part 2: Dose Expansion An interim analysis may be conducted when the last participant within each arm is followed for at least 1 cycle to evaluate safety, efficacy, and PK profiles at each dose level. Following the interim analysis, additional analyses may be performed to continue to evaluate safety, efficacy, and PK profiles at each dose level, prior to the primary and final analyses. If any dose level is not enrolled due to safety concerns, it will not be included in the interim or final analyses. Additionally, if enrollment is stopped within a dose group, data may be analyzed for participants within the dose group who take at least 1 dose of any study treatment. |
| | Continuous monitoring will be conducted for Part 2 starting from when 5 participants are dosed at each dose level within each arm. The observed number of participants permanently discontinuing study treatment within the first two cycles due to AE related to belantamab mafodotin will be compared against the safety stopping rule in Table 30 of the Protocol (Version: GSK Document Number TMF-14624358). Enrollment may stop if the safety stopping rule is met based on totality of safety data. For example, if 4 or more out of 5 participants permanently discontinued study treatment within the first 2 cycles due to AE related to belantamab mafodotin, enrollment may stop after review of all safety data; otherwise, enrollment will continue. |

#### 2.4. Statistical Hypotheses / Statistical Analyses

#### 2.4.1. Arm A - Belantamab Mafodotin with Len/Dex

#### 2.4.1.1. Part 1 Dose Escalation

No formal statistical hypotheses are being tested in Part 1. Analysis of the data obtained from Part 1 will only utilize descriptive methods.

#### 2.4.1.2. Part 2 Dose Expansion

No formal statistical hypotheses are being tested in Part 2. Analysis of the data obtained from Part 2 will only utilize descriptive methods.

For Part 2, the number of participants who permanently discontinue study treatment due to AEs related to belantamab mafodotin within the first two cycles will be continuously monitored. For STRETCH dosing schedule, a cycle is a SoC cycle of 28 days. If the observed number of participants permanently discontinuing belantamab mafodotin is significantly higher than 12% (at 1-sided alpha of 0.01), then the combination treatment at that dose level or higher dose level will be considered to have unacceptable toxicity and the dose level as well as higher dosed levels will be closed.

#### 2.4.2. Arm B - Belantamab Mafodotin with Bor/Dex

#### 2.4.2.1. Part 1 Dose Escalation

No formal statistical hypotheses are being tested in Part 1. Analysis of the data obtained from Part 1 will only utilize descriptive methods.

#### 2.4.2.2. Part 2 Dose Expansion

No formal statistical hypotheses are being tested in Part 2. Analysis of the data obtained from Part 2 will only utilize descriptive methods.

For Part 2, the number of participants who permanently discontinued study treatment due to AEs related to belantamab mafodotin within the first two cycles will be continuously monitored starting from when 5 participants are dosed. For STRETCH dosing schedule, a cycle is a SoC cycle of 21 days. If the observed number of participants permanently discontinuing belantamab mafodotin is significantly higher than 12% (at 1-sided alpha of 0.01), then the combination treatment at that dose level or higher dose level will be considered to have unacceptable toxicity and the dose level as well as higher dose levels will be closed.

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

#### 3.1.1. Arm A – Belantamab Mafodotin with Len/Dex

#### 3.1.1.1. Part 1 Dose Escalation

During dose escalation, no formal interim analysis will be performed. Data will be reviewed through data visualization tool to inform dose escalation decisions. The mTPI design will be utilized to guide dose escalation/de-escalation decisions. More details of the dose escalation procedure are described below.

#### Description of the Modified Toxicity Probability Interval

The modified Toxicity Probability Interval (mTPI) design [Ji, 2010] will be used to guide dose escalation in Part 1 with a slight modification. Up to 2 dose levels of belantamab mafodotin (1.9 mg/kg [dose -1]; 2.5 mg/kg [dose 1]) and alternate dosing schedules are planned to be evaluated in combination with the fixed dose of the Len/Dex treatments. Based on emerging data under Protocol Amendment 1 from Arm A, the first dose investigated under Protocol Amendment 2 was 1.9 mg/kg (Dose Level -1). The design assumes the true underlying toxicity rate for maximum tolerated dose (MTD) of belantamab mafodotin falls within the range from 25% to 35% and centers at 30%. The rules for guiding dose escalations are provided in Figure 1. Columns provide the numbers of participants treated at the current dose level, and rows provide the corresponding numbers of participants experiencing toxicity. Cohorts will be recruited in blocks of three participants. Participants will be treated in a staggered approach with at least 1 day between each participant's first dose of belantamab mafodotin to minimize the risk of inadvertently exceeding the MTD in multiple participants.

In Part 1 up to 2 dose levels of belantamab mafodotin and up to 2 dosing schedules will be evaluated (Figure 1 and Table 2). Data from at least 3 DLT-evaluable participants are required before a decision is made to escalate to the next dose level. However, this is not required for enrollment of more participants at the same dose level in Part 2.

| | | | Number of | Participants t | reated at curr | ent dose | |
|----|---|---|-----------|----------------|----------------|----------|-----|
| S | | 1 | 2 | 3 | 4 | 5 | 6 |
| Ë | 0 | E | E | E | E | E | E |
| Ū. | 1 | D | S | S | S | S | E |
| Ö | 2 | | DU | D | S | S | S |
| pe | 3 | | | DU | DU | D | S |
| μn | 4 | | | | DU | DU | DU |
| Z | 5 | | | | | DU | DU |
| | 6 | | | | | | DII |

Figure 1 Dose-finding Criteria for the Modified Toxicity Probability Interval (mTPI) Dose-Finding Method

The spreadsheet was generated based on a beta/binomial model and precalculated before trial initiation. The letters in different colors are computed based on the decision rules under the mTPI method and represent different dose-finding actions. In addition to actions de-escalate the dose (D), stay at the same dose (S), and escalate the dose (E), the table includes action unacceptable toxicity (DU), which is defined as the execution of the dose-exclusion rule in mTPI. Excerpted from Ji, et al. [Ji, 2010].

The entries of Figure 1 are dose-finding decisions (i.e., E, S, and D) representing escalating the dose, staying at the same dose, and de-escalating the dose. In addition, decision DU means that the current dose level is unacceptable because of high toxicity; the current dose level and any higher dose level should be excluded from the trial.

For example, when 1 of 3 participants experiences toxicity, the decision can be located at row 1 and column 3, which is S- to stay at the current dose level. Consequently, the next cohort of participants will be treated at the same dose level currently being used. If zero of three participants experience toxicity, the decision is at row 0 and column 3, which is E- to escalate. Thus, the next cohort of participants will be treated at the next-higher dose level. If 3 of 3 participants experience toxicity, the decision is DU- to de-escalate to the next-lower dose level and exclude the current dose and any higher dose from the trial, because toxicity levels are unacceptable. In dose escalation (E)/de-escalation (D), no dose skipping is allowed.

Table 2 Dose Levels: Arm A, Part 1

| Treatment Group and Dose Level | Belantamab Mafodotin | Lenalidomide | Dexamethasone |
|---|---|---|---|
| Permissible Actions | Increase/Decrease | No changes | No changes |
| Dose Level -1<br>(de-escalation) | 1.9 mg/kg IV q28 days | 25 or 10 mg PO, QD on<br>Days 1 to 21 of each 28-<br>day cycle | 40 or 20 mg/week PO or IV on Days 1, 8, 15, and 22 of each 28-day cycle |
| Dose Level 1 | 2.5 mg/kg IV q28 days <sup>a</sup> | 25 or 10 mg PO, QD on<br>Days 1 to 21 of each 28-<br>day cycle | 40 or 20 mg/week PO or IV on Days 1, 8, 15, and 22 of each 28-day cycle |

IV = intravenous; PO = orally; QD = once daily; SC = subcutaneous

Alternate dosing schedule could be investigated such as 2.5 mg/kg SPLIT dosing schedule where belantamab mafodotin will be administered at 1.25 mg/kg each on Day 1 and Day 8

Any participant from Part 1 in Arm A who received at least 1 full dose of belantamab mafodotin and at least 75% of planned doses of Len/Dex by the end of Cycle 1 (Day 28 for Arm A) is considered DLT-evaluable. Participants in Part 1 who have received less than 1 full dose of belantamab mafodotin, or <75% of planned doses of Len/Dex, or who have been withdrawn from the study for reasons other than toxicity but prior to completion of DLT observation period will be replaced.

Part 1 starts with a cohort of 3 participants at a dose level of 1.9 mg/kg SINGLE. Safety data over the first cycle of treatment for each participant will be evaluated. Data from at least 3 DLT evaluable participants are required before a decision is made to escalate to the next dose level. The study will enroll participants in Part 1 will have staggered start times, but will run simultaneously as outlined below. If dose levels are open for both Part 1 and Part 2, priority for enrollment will be given to Part 1.

Rules for of mTPI dose escalation pertaining to Arm A only:

- If dose escalation decision is E, enrollment for Part 1 will be open at 2.5 mg/kg SINGLE and 2.5 mg/kg SPLIT. At the same time, Part 2 expansion could be opened to enroll additional participants at 1.9 mg/kg SINGLE.
- If dose escalation decision is S, three additional participants will be enrolled at 1.9 mg/kg SINGLE in Part 1 to achieve at least 6 DLT-evaluable participants at 1.9 mg/kg SINGLE. After review of data from the 6 participants:
  - o If dose escalation decision is E, 2.5 mg/kg SINGLE and 2.5 mg/kg SPLIT will be open for enrollment in Part 1. Part 2 expansion will not be open for the 1.9 mg/kg SINGLE dose level unless emerging data suggest 2.5 mg/kg SINGLE and 2.5 mg/kg SPLIT are not tolerable.
  - o If dose escalation decision is S, enrollment will not open for dose levels higher than 1.9 mg/kg SINGLE in Part 1. Part 2 expansion will be open to enroll additional participants at 1.9 mg/kg SINGLE.
  - o If dose escalation decision is D or DU, no more participants will be enrolled at 1.9 mg/kg SINGLE or higher dose levels in Part 1.

Once the 2.5 mg/kg SINGLE and 2.5 mg/kg SPLIT cohorts are open for enrollment in Part 1, a cohort of at least 3 participants will be enrolled for each dose. When Part 1 is filled, Part 2 expansion will open for enrollment at 2.5 mg/kg SINGLE and 2.5 mg/kg SPLIT. Data from at least 6 DLT-evaluable participants at 2.5 mg/kg SINGLE and 2.5 mg/kg SPLIT are not required for enrollment of additional participants in Part 2.

Operating characteristics of the dose escalation rules are shown in Table 3.

Table 3 Operating Characteristics of the Dose Escalation Rules for Arm A

| | Unde | erlying True Tox | lying True Toxicity Rate Average n. of participants dosed at each dosed level <sup>1</sup> | | | ed at each dose | Prob. of Selecting as MTD <sup>2</sup> | | |
|---|---|---|---|---|---|---|---|---|---|
| Scenario | 1.9 SINGLE | 2.5 SPLIT | 2.5 SINGLE | 1.9 SINGLE <sup>3</sup> | 2.5 SPLIT | 2.5 SINGLE | <1.9 | 1.9 SINGLE | 2.5 SINGLE /<br>2.5 SPLIT |
| 1 | 0.2 | 0.30 | 0.30 | 11 | 9 | 9 | 0.11 | 0.23 | 0.66 |
| 2 | 0.2 | 0.30 | 0.35 | 11 | 9 | 9 | 0.11 | 0.25 | 0.64 |
| 3 | 0.2 | 0.40 | 0.40 | 11 | 8 | 8 | 0.11 | 0.31 | 0.58 |
| 4 | 0.2 | 0.40 | 0.45 | 11 | 9 | 9 | 0.11 | 0.34 | 0.56 |
| 5 | 0.3 | 0.40 | 0.40 | 10 | 6 | 6 | 0.23 | 0.37 | 0.40 |
| 6 | 0.3 | 0.40 | 0.45 | 10 | 6 | 6 | 0.23 | 0.38 | 0.39 |
| 7 | 0.1 | 0.30 | 0.30 | 12 | 11 | 11 | 0.03 | 0.13 | 0.84 |
| 8 | 0.1 | 0.25 | 0.30 | 12 | 11 | 11 | 0.03 | 0.11 | 0.86 |
| 9 | 0.1 | 0.25 | 0.25 | 12 | 11 | 11 | 0.03 | 0.10 | 0.87 |
| 10 | 0.1 | 0.20 | 0.20 | 12 | 11 | 11 | 0.03 | 0.08 | 0.89 |
| 11 | 0.1 | 0.20 | 0.25 | 12 | 11 | 11 | 0.03 | 0.09 | 0.88 |

**Bold**: Dose too toxic/n of participants exposed to a toxic dose/prob. of selecting toxic dose as MTD *Italicized*: True MTD dose/prob. of selecting true MTD as MTD

<sup>1.</sup> Average n. of participants dosed at each dose level include n. of participants dosed in Part 2 assuming participants for each dose level in Part 2 are enrolled before dose escalation decision is made in Part 1, except for dose 1.9 mg/kg, for which Part 2 will not open for enrollment prior to dose escalation decision.

<sup>2.</sup> Based on participants enrolled in Part 1 and assume the underlying true MTD is 30%.

<sup>3.</sup> Number in this column represents maximum estimate where dose is escalated to 2.5 mg/kg but is de-escalated to 1.9 mg/kg based on Part 1 and Part 2 data from 2.5 mg/kg.

#### Dose Escalation Decisions

During Part 1, the decisions on dose escalation will be made based on the mTPI guidance, as well as the totality of the safety, and pharmacokinetics data as appropriate. The decisions will occur following review of all available data including participants data from Part 2 and joint discussion by the GSK medical monitor, participating investigators, and others as described in the Dose Escalation Plan.

The GSK study team, which includes but is not limited to, the GSK medical monitor, clinical scientist, safety physician, statistician, and clinical pharmacologist, will review critical safety data defined in the Dose Escalation Plan prior to making a recommendation for dose escalation. This includes review of all adverse events including non-DLT toxicities, laboratory assessments and other defined safety evaluations, as well as PK and/or PD data, when appropriate. The results from the mTPI method will be included in the decision for dose modification as described in Section 12.4.8 of the Protocol (Version: GSK Document TMF-14624358). Quality control of critical safety data will be described in the Dose Escalation Plan, which includes ongoing study monitoring visits, GSK review of the clinical database, and confirmation by participating investigators and/or delegate that the data are accurate and complete prior to making dose modification decisions.

The GSK medical monitor, in joint discussion with participating investigators, and others as described in the Dose Escalation Plan will be responsible for making dose escalation decisions. The dose-escalation decision and rationale for each cohort will be discussed with investigators during teleconference(s) and documented in writing, with copies maintained at each study site and in the study master file.

#### 3.1.1.2. Part 2 Dose Expansion

Once Part 2 expansion is open for the 2.5 mg/kg SINGLE and 2.5 mg/kg SPLIT dose levels, up to 9 participants will be enrolled at each dosing schedule, unless enrollment is stopped based on emerging data.

In addition, up to 12 more participants maybe potentially enrolled to evaluate an extended (STRETCH) dosing schedule for belantamab mafodotin at the 1.9 mg/kg dose level if emerging data suggests that this schedule may further optimize the tolerability or offers an improved benefit/risk profile.

For STRETCH Dosing Schedule, belantamab mafodotin will be administered FIRST (prior to Len/Dex) as a single dose on Day 1 of every alternate 28-day cycle (C1, C3, C5, C7 and so on) as a 30-60 min infusion, followed by 1 to 2 h rest period. If a planned dose of belantamab mafodotin was held/missed due to any reason, the next dose can be administered at Day 1 of the next planned 28-day cycle, as long as the interval between 2 consecutive doses is at least 56 (±3) days.

Safety data from all enrolled participants will be closely monitored while the study is ongoing. In addition, participants permanently discontinuing study treatment within the first two cycles due to AEs related to belantamab mafodotin will be continuously monitored starting from when 5 participants are dosed at each dose level following pre-

defined safety stopping rules (Section 12.4.8.1 of the Protocol –Version: GSK Document TMF-14624358). If safety concerns arise at a dose level, enrollment will stop for that dose level and higher dose level(s).

#### Safety Stopping Rule

Continuous monitoring will be conducted for Part 2 starting from when 5 participants are dosed at each dose level within each arm. The observed number of participants permanently discontinuing study treatment within the first two cycles due to AE related to belantamab mafodotin will be compared against the safety stopping rule in Table 4. Enrollment may stop if the safety stopping rule is met based on totality of safety data. For example, if 4 or more out of 5 participants permanently discontinued study treatment within the first 2 cycles due to AE related to belantamab mafodotin, enrollment may stop after review of all safety data; otherwise, enrollment will continue. Operating characteristics for the stopping rule are provided in Figure 2.

Table 4 Safety Stopping Rules for Part 2

| Number of dosed | Stop if number of | Observed Rate |
|-----------------|------------------------------|---------------|
| participants | participants discontinuing | |
| | study treatment within the | |
| | first two cycles due to AE | |
| | related to belantamab | |
| | mafodotin is larger or equal | |
| | to this number | |
| 5-8 | 4 | 0.5-0.8 |
| 9-12 | 5 | 0.42-0.56 |

Figure 2 Operating Characteristics of Safety Stopping Rule for Expansion Cohort



An interim analysis may be conducted when the last participant within each arm is followed for at least 1 cycle to evaluate safety, efficacy, and PK profiles at each dose level. Following the interim analysis, additional analyses may be performed to continue to evaluate safety, efficacy, and PK profiles at each dose level, prior to the primary and final analyses. If any dose level is not enrolled due to safety concerns, it will not be included in the interim or final analyses. Additionally, if enrollment is stopped within a dose group, data may be analyzed for participants within the dose group who take at least 1 dose of any study treatment.

#### 3.1.2. Arm B- Belantamab Mafodotin with Bor/Dex

#### 3.1.2.1. Part 1 Dose Escalation Phase

During dose escalation, no formal interim analysis will be performed. Data will be reviewed through the data visualization tool to inform dose escalation decisions. The mTPI design will be utilized to guide dose escalation/de-escalation decisions. More details of the dose escalation procedure are described below.

#### Description of the Modified Toxicity Probability Interval

An mTPI design will be implemented [Ji, 2010] to guide dose escalation in Part 1. Up to 3 dose levels of belantamab mafodotin (2.5 mg/kg [dose 1]; 3.4 mg/kg [dose +1]; 1.9 mg/kg [dose -1]), starting with 2.5 mg/kg, are planned to be evaluated in combination

with the fixed dose of Bor/Dex. Cohorts will be recruited in blocks of three participants. Participants will be entered in a staggered approach with at least 1 day between each participant's first dose of belantamab mafodotin to minimize the risk of inadvertently exceeding the maximum tolerated dose (MTD) in multiple participants. A maximum of 6 participants will be assigned to each dose (Table 5).

| Table 5 | Dose I | evels: | Δrm F | 3, Part 1 |
|---------|--------|-----------|-------|-----------|
| Iable J | DUSE | _cvci3. / | | J. Fait i |

| Treatment Group and Dose Level | Belantamab Mafodotin | Bortezomib | Dexamethasone |
|---|---|---|---|
| Permissible Actions | Increase/Decrease | No changes | No changes |
| Dose Level -1<br>(de-escalation) | 1.9 mg/kg IV q21 days | 1.3 mg/m² SC/IV on Days<br>1, 4, 8, and 11 of every<br>21-day cycle for a total<br>up to 8 cycles | 20 mg PO or IV on Days<br>1, 2, 4, 5, 8, 9, 11, and 12<br>of every 21-day cycle for<br>a total of up to 8 cycles. |
| Dose Level 1<br>Cohort | 2.5 mg/kg IV q21 days <sup>a</sup> | 1.3 mg/m² SC/IV on Days<br>1, 4, 8, and 11 of every<br>21-day cycle for a total<br>up to 8 cycles | 20 mg PO or IV on Days<br>1, 2, 4, 5, 8, 9, 11, and 12<br>of every 21-day cycle for<br>a total of up to 8 cycles. |
| Dose Level +1<br>Cohort | 3.4 mg/kg IV q21 days <sup>b</sup> | 1.3 mg/m² SC/IV on Days<br>1, 4, 8, and 11 of every<br>21-day cycle for a total<br>up to 8 cycles | 20 mg PO or IV on Days<br>1, 2, 4, 5, 8, 9, 11, and 12<br>of every 21-day cycle for<br>a total of up to 8 cycles. |

IV = intravenous; PO = orally; QD = once daily; SC = subcutaneous

Evaluation of the available safety data over the first cycle of treatment for each participant enrolled in that dose level is required from at least 3 participants before a decision is made to enroll additional participants at the same or the subsequent dose level. However, this is not required for enrollment of more participants at the same dose level in Part 2.

An additional dose level -1 of 1.9 mg/kg may be evaluated in case the starting dose of 2.5 mg/kg is considered not tolerated.

Rules for mTPI dose escalation pertaining to Arm B only:

- If 2.5 mg/kg is the current dose level and the decision is S, and if less than 6 participants have been evaluated for DLT and the planned maximum sample size is not reached, an additional cohort of 3 participants will be enrolled for DLT evaluation. If the dose escalation decision is S after this additional cohort, dose escalation is complete.
- If 2.5 mg/kg is the current dose level and the decision is U or DU, additional lower dose (e.g., 1.9 mg/kg) may be explored. If the dose of 1.9 mg/kg is not tolerated (i.e., results in excessive toxicity) the trial will be terminated early for lack of tolerability.

a. Alternate dosing schedule could be investigated such as SPLIT dosing schedule where belantamab mafodotin will be administered at 1.25 mg/kg each on Day 1 and Day 8

Alternate dosing schedule could be investigated such as SPLIT dosing schedule where belantamab mafodotin will be administered at 1.7 mg/kg each on Day 1 and Day 8

- If 3.4 mg/kg is the current dose level and the decision is E or S, and if less than 6 participants have been evaluated for DLT at the current dose, and the planned maximum sample size is not reached, an additional cohort of 3 participants will be evaluated for DLT at the current dose. If dose escalation is E or S after this additional cohort, dose escalation is complete.
- Otherwise, the dose escalation will continue until the planned maximum sample size (12 DLT-evaluable participants for each treatment) is reached. At the end of dose escalation, the rule proposed by Ji, et al. [Ji, 2010] used to guide the selection of the estimated MTD, from dose levels at which 3 or more participants have been evaluated for DLT.

During Part 1, the decisions on dose escalation will be made based on this guidance, as well as the totality of the safety, and pharmacokinetics data as appropriate.

The decisions will occur following review of these data and joint discussion by the GSK medical monitor, participating investigators, and others as described in the Dose Escalation Plan.

Any participant in Arm B who received at least 1 full dose of belantamab mafodotin and ≥75% of planned doses of Bor/Dex by the end of Cycle 1 (Day 21) will be evaluated for DLTs. Participants who have received less than 1 full dose of belantamab mafodotin, or <75% of planned doses of Bor/Dex, or who have been withdrawn from the study for reasons other than toxicity but prior to completion of DLT observation period will be replaced.

The dose escalation of belantamab mafodotin will not include doses higher than 3.4 mg/kg.

#### Dose Escalation Decisions

The GSK study team, which includes but is not limited to, the GSK medical monitor, clinical scientist, safety physician, statistician, and clinical pharmacologist, will review critical safety data defined in the Dose Escalation Plan prior to making a recommendation for dose escalation. This includes review of all adverse events including non-DLT toxicities, laboratory assessments and other defined safety evaluations, as well as PK and/or PD data, when appropriate. The results from the mTPI method will be included in the decision for dose modification. Quality control of critical safety data will be described in the Dose Escalation Plan, which includes ongoing study monitoring visits, GSK review of the clinical database, and confirmation by participating investigators and/or delegate that the data are accurate and complete prior to making dose modification decisions.

The GSK medical monitor, in joint discussion with participating investigators and GSK study team, will be responsible for making dose escalation decisions. The dose escalation decision and rationale for each cohort will be discussed with investigators during teleconference(s) and documented in writing, with copies maintained at each study site and in the study master file.

#### 3.1.2.2. Part 2 Dose Expansion Phase

In Part 2 enrollment will proceed in multiple expansion cohorts to further evaluate the safety profile and to evaluate the preliminary clinical activity of belantamab mafodotin in combination with Bor/Dex at 3 dose levels and 4 dosing schedules (2.5 mg/kg SPLIT, 2.5 mg/kg SINGLE, 3.4 mg/kg SPLIT, 3.4 mg/kg SINGLE, 2.5 mg/kg STRETCH, S/D STRETCH, 1.9 mg/kg SINGLE and 1.9 mg/kg STRETCH).

In Amendment 2, enrollment of each cohort was conducted by blocks of 3 participants each at 2.5 mg/kg SPLIT, 2.5 mg/kg SINGLE, 3.4 mg/kg SPLIT, and 3.4 mg/kg SINGLE with Bor/Dex for up to 12 participants each at 2.5 mg/kg SPLIT, 2.5 mg/kg SINGLE, 3.4 mg/kg SPLIT and up to 9 participants at 3.4 mg/kg SINGLE.

Similarly, in Amendment 3, enrollment of each cohort will be conducted by blocks of 3 participants each in 2.5 mg/kg STRETCH, S/D STRETCH, 1.9 mg/kg SINGLE and 1.9 mg/kg STRETCH, until approximately 12 participants are enrolled in each cohort.

For the SINGLE dosing schedule, belantamab mafodotin will be administered as a SINGLE full dose on Day 1 of each 21-day cycle. For example: A "3.4 mg/kg SINGLE" dosing schedule will administer a 3.4 mg/kg dose on Day 1 of each cycle. A 2.5 mg/kg SINGLE dosing schedule of belantamab mafodotin will administer a 2.5 mg/kg dose on Day 1 of each cycle. A 1.9 mg/kg SINGLE dosing schedule of belantamab mafodotin will administer a 1.9 mg/kg dose on Day 1 of each cycle

For the SPLIT dosing schedule, belantamab mafodotin will be split into two equal halves and each half dose will be administered on Day 1 and Day 8 of each 21-day cycle. For example: A "2.5 mg/kg SPLIT" dosing schedule will administer a 1.25 mg/kg dose on Day 1 and a 1.25 mg/kg dose on Day 8 of each cycle. A "3.4 mg/kg SPLIT" dosing schedule will administer a 1.7 mg/kg dose on Day 1 and a 1.7 mg/kg dose on Day 8 of each cycle.

For STRETCH Dosing Schedule, belantamab mafodotin will be administered FIRST (prior to Bor/Dex) as a single dose on Day 1 of every alternate 21-day cycle (C1, C3, C5, C7 and so on) as a 30-60 min infusion, followed by 1 to 2 h rest period. If a planned dose of belantamab mafodotin was held/missed due to any reason, the next dose can be administered at Day 1 of the next planned 21-day cycle, as long as the interval between 2 consecutive doses is at least 42 (±3) days.

For the S/D STRETCH schedule, belantamab mafodotin will be administered FIRST (prior to Bor/Dex) as a 2.5 mg/kg dose on Day 1 of Cycle 1, followed by 1.9 mg/kg S/D dose on Day 1 of all subsequent alternate 21-day cycles (C3, C5, C7 and so on), as a 30-60 min infusion, followed by 1 to 2 h rest period.

Safety data from all enrolled participants will be closely monitored while the study is ongoing. In addition, participants permanently discontinuing study treatment within the first two cycles due to AEs related to belantamab mafodotin will be continuously monitored starting from when 5 participants are dosed at each dose level following predefined safety stopping rules (Section 12.4.8.2 of the Protocol –Version: GSK Document

TMF-14624358). If safety concerns arise at a dose level, enrollment will stop for that dose level and higher dose level(s).

#### Safety Stopping Rule

Continuous monitoring will be conducted for Part 2 starting from when 5 participants are dosed at each dose level within each arm. The observed number of participants permanently discontinuing study treatment within the first two cycles due to AE related to belantamab mafodotin will be compared against the safety stopping rule in Table 4. Enrollment may stop if the safety stopping rule is met based on totality of safety data. For example, if 4 or more out of 5 participants permanently discontinued study treatment within the first 2 cycles due to AE related to belantamab mafodotin, enrollment may stop after review of all safety data; otherwise, enrollment will continue. Operating characteristics for the stopping rule are provided in Figure 2.

An interim analysis may be conducted when the last participant within each arm is followed for at least 1 cycle to evaluate safety, efficacy, and PK profiles at each dose level. Following the interim analysis, additional analyses may be performed to continue to evaluate safety, efficacy, and PK profiles at each dose level, prior to the primary and final analyses. If any dose level is not enrolled due to safety concerns, it will not be included in the interim or final analyses. Additionally, if enrollment is stopped within a dose group, data may be analyzed for participants within the dose group who take at least 1 dose of any study treatment.

#### 3.2. Final Analyses

Final analysis of the data captured in Part 1 and Part 2 for both Arm A and Arm B will be undertaken following 12 months post LSFD. Within each arm, data from the two parts may be combined for some analyses at the final analysis, as appropriate.

Following the final analysis, the study will move into the PACT phase and the clinical study database will be closed to new data. Participants who are receiving belantamab mafodotin monotherapy or in combination with Len/Dex (Arm A) or Bor/Dex (Arm B) may continue to receive belantamab mafodotin monotherapy or in combination with either Len/Dex (Arm A) or Bor/Dex (Arm B) if they are gaining clinical benefit as assessed by the investigator until they meet any criterion for permanent discontinuation of study intervention (see Section 9 and Section 10.2 of GSK Document Number TMF-14624358).

The end of study is defined when the last patient had their last visit (last subject last dose plus 70 days SAE reporting period). GSK retains the right to request additional information for any patient with ongoing AE(s)/SAE(s) ocular data at the end of the study. All participants will be monitored and receive follow-up care in accordance with standard local clinical practice.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Screened | All participants who sign the ICF to participate in the clinical trial. | Screen failure summary |
| All Treated | All participants who received at least one dose of study treatment. | Study Population,<br>Efficacy, Safety,<br>Patient Reported<br>Outcomes |
| Pharmacokinetic<br>(PK) | Participants in the All Treated population from whom at least one PK sample was obtained, analyzed, and was measurable. Separate PK populations will be defined for each drug (belantamab mafodotin, lenalidomide, and bortezomib). Lenalidomide PK population will be split between subjects on 25mg and 10mg of lenalidomide. | PK |
| Pharmacodynamic (PD) | Participants in the 'All Treated' population for whom a biomarker sample was obtained, was analysed and it was found measurable. | Biomarker |

Refer to Appendix 12 which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [Version 6.0, dated 14DEC2022].

- O Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations may also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Data Displays for Reporting [1] | | | |
|---|---|---|---|
| Description [2] | Data Display [2] | Order in TLF | Deliverable [3] |
| Arm A: GSK2857916 1.9 mg/kg<br>STRETCH + Len/Dex | GSK916 1.9mg/kg STRETCH +Rd | 1 | Interim 2, SAC |
| Arm A: GSK2857916 1.9 mg/kg<br>SINGLE + Len/Dex | GSK916 1.9mg/kg SINGLE +Rd | 2 | Interim 2, SAC |
| Arm A: GSK2857916 2.5 mg/kg<br>SPLIT + Len/Dex | GSK916 2.5mg/kg SPLIT +Rd | 3 | Interim 2, SAC |
| Arm A: GSK2857916 2.5 mg/kg<br>SINGLE + Len/Dex | GSK916 2.5mg/kg SINGLE +Rd | 4 | Interim 2, SAC |
| Arm B: GSK2857916 1.9 mg/kg<br>STRETCH + Bor/Dex | GSK916 1.9mg/kg STRETCH +Vd | 1 | Interim 3, SAC |
| Arm B: GSK2857916 1.9 mg/kg<br>SINGLE + Bor/Dex | GSK916 1.9mg/kg SINGLE +Vd | 2 | Interim 3, SAC |
| Arm B: GSK2857916 2.5 mg/kg<br>S/D STRETCH + Bor/Dex | GSK916 2.5mg/kg S/D STRETCH<br>+Vd | 3 | Interim 3, SAC |
| Arm B: GSK2857916 2.5 mg/kg<br>STRETCH + Bor/Dex | GSK916 2.5mg/kg STRETCH +Vd | 4 | Interim 3, SAC |
| Arm B: GSK2857916 2.5 mg/kg<br>SPLIT + Bor/Dex | GSK916 2.5mg/kg SPLIT +Vd | 5 | Interim 1, Interim 3,<br>SAC |
| Arm B: GSK2857916 2.5 mg/kg<br>SINGLE + Bor/Dex | GSK916 2.5mg/kg SINGLE +Vd | 6 | Interim 1, Interim 3,<br>SAC |
| Arm B: GSK2857916 3.4 mg/kg<br>SPLIT + Bor/Dex | GSK916 3.4mg/kg SPLIT +Vd | 7 | Interim 1, Interim 3,<br>SAC |
| Arm B: GSK2857916 3.4 mg/kg<br>SINGLE + Bor/Dex | GSK916 3.4mg/kg SINGLE +Vd | 8 | Interim 1, Interim 3,<br>SAC |

#### Notes:

<sup>[1]</sup> No randomization schedule is planned for this double-arm open label study

<sup>[2]</sup> Rd: Lenalidomide Plus Dexamethasone; Vd: Bortezomib Plus Dexamethasone

<sup>[3]</sup> SAC = Statistical Analysis Complete (final analysis); Specifics of Interim 1, Interim 2, Interim 3, and SAC deliverables are defined in Section 15.12.2.

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions), the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

For laboratory data, baseline will be the latest non-missing pre-dose value from central lab. If no central lab value is available, the latest non-missing pre-dose value from local lab will be used. If there are multiple assessments on the same day, the mean will be used as the baseline value.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Examination of Covariates, Other Strata and Subgroups

## 5.3.1. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- Subgroup analyses will be performed over all doses combined, within each Arm (Arms A and B), as well as within the 2.5 mg/kg SINGLE dose alone.
- If the percentage of participants is small within a particular subgroup, then the subgroup categories may be refined.

| Subgroup | Categories |
|---|---|
| Age Group (at screening) | 18 to <65, 65 to < 75, ≥ 75 |
| Sex | Male, Female |
| Race | White, Black, Other/Missing |
| ISS Staging at Screening | I vs II/III (do not include unknown stages) |
| Number of prior lines of therapy | 1 vs. 2/3 vs. 4+ and 1 vs. >1 |
| Myeloma Immunoglobulin | IgG, Non-IgG, Both |
| Cytogenetics Risk [1] | High, Other (non-high risk - all others) |
| ECOG Performance Status | 0-1, 2+ |
| Prior Bortezomib | No, Yes |
| Prior Daratumumab | No, Yes |
| Prior Lenalidomide | No, Yes |

#### NOTES:

<sup>[1]</sup> A participant is considered as high risk if the participant has any of the following cytogenetics: t(4;14), t(14;16), and 17p13del.
# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|-------------|----------------------------------------------------------------|
| Section15.1 | Appendix 1: Assessment Windows |
| Section15.2 | Appendix 2: Study Phases and Treatment Emergent Adverse Events |
| Section15.3 | Appendix 3: Data Display Standards & Handling Conventions |
| Section15.4 | Appendix 4: Derived and Transformed Data |
| Section15.5 | Appendix 5: Reporting Standards for Missing Data |
| Section15.6 | Appendix 6: Values of Potential Clinical Importance |

### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "All Treated" population, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, anti-cancer therapy, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12.

# 6.2. Disposition of Participants

A summary of subject status and reason for study withdrawal will be provided. This display will show the number and percentage of subjects who withdrew from the study, including primary reasons for study withdrawal. Reasons for study withdrawal will be presented in the order they are displayed in the eCRF.

A summary of study treatment status will be provided. This display will show the number and percentage of subjects who are ongoing or discontinued study treatment and a summary of the primary reasons for discontinuation of study treatment. Reasons for study treatment discontinuation will be presented in the order they are displayed in the eCRF. A listing of study treatment discontinuation will be generated. The listing will include last dose date and reasons for study treatment discontinuation.

To understand the impact of COVID-19, related analyses will include summaries of subject status, and subject disposition by relationship to COVID-19 pandemic. An additional summary of treatment status and reasons for discontinuation of belantamab mafodotin by relationship to COVID-19 pandemic will also be produced, and added to existing discontinuation displays.

# 6.3. Demographic and Baseline Characteristics

The demographic characteristics (e.g., age, race, ethnicity, sex, baseline height, baseline body weight and baseline BMI) will be summarized. Age, height, weight, and BMI will be summarized using the mean, standard deviation, minimum, median, and maximum. The count and percentage will be computed for sex and ethnicity.

Race and racial combinations may be summarized and listed.

Disease history and characteristics at screening will be summarized. Disease characteristics at screening will include stage, relapsed or refractory disease, extramedullary disease, lytic bone lesions, myeloma immunoglobulin, myeloma light chain, type of multiple myeloma, lines of therapy completed prior to screening, ECOG performance status, genetics, and high-risk cytogenetics. For lines of therapy completed prior to screening, groups will be displayed as no lines, 1 line, 2 lines, ..., 20 lines, more than 20 lines, and unknown. Lines of therapy completed prior to screening will also be

summarized with n, mean, standard deviation, median, min, and max. For ECOG performance status, groups will be displayed as 0, 1, 2, for both Arms A and B.

Substance use, including smoking history and alcohol use may be summarized.

Prior anti-cancer therapy will be coded using GSK Drug coding dictionary, then summarized by ingredient and listed.

# 6.4. Treatment Compliance

Summaries of study treatment exposure and dose modifications (e.g., number of dose reductions, number of dose delays) will further characterize compliance. These analyses are defined in Section 6.5 'Extent of Exposure'.

# 6.5. Extent of Exposure

Extent of exposure to belantamab mafodotin, lenalidomide, bortezomib, and dexamethasone will be summarized.

The start date of the overall study treatment is defined as the first dose date of belantamab mafodotin.

The overall duration of exposure to study treatment (defined in Section 15.4.2) will be calculated and summarized in weeks, using mean, median, standard deviation, minimum, and maximum.

Descriptive statistics of dose intensity will be summarized overall for belantamab mafodotin, lenalidomide, bortezomib, and dexamethasone separately. An additional table of dose intensity by expected duration of exposure may also be summarized. This "dose intensity by expected duration of exposure" summary will adjust for delayed cycles by using cumulative dose from the last non-missing visit, and an estimate of expected duration of exposure.

The dose intensity calculation is described below.

- For Arm A SINGLE/SPLIT belantamab mafodotin doses, as well as lenalidomide and dexamethasone: Dose intensity (units/4 weeks) = cumulative actual dose divided by duration of exposure in 4 weeks (duration of exposure in days / 28).
- For Arm A STRETCH belantamab mafodotin doses: Dose intensity (units/8 weeks) = cumulative actual dose divided by duration of exposure in 8 weeks (duration of exposure in days / 56).
- For Arm B SINGLE/SPLIT belantamab mafodotin doses, as well as bortezomib and dexamethasone: Dose intensity (units/3 weeks) = cumulative actual dose divided by duration of exposure in 3 weeks (duration of exposure in days / 21).

- For Arm B STRETCH belantamab mafodotin doses: Dose intensity (units/6 weeks) = cumulative actual dose divided by duration of exposure in 6 weeks (duration of exposure in days / 42).
- Duration of exposure in days used for the dose intensity calculation is defined as: end date of the cycle first dose date + 1 day. The end date of the cycle is defined as the cycle start date + 27 days (Arm A SINGLE/SPLIT belantamab mafodotin, Len, Dex), or + 55 days (Arm A STRETCH belantamab mafodotin), or + 20 days (Arm B SINGLE/SPLIT belantamab mafodotin, Bor, Dex), or + 41 days (Arm B STRETCH and S/D STRETCH belantamab mafodotin).

Note: Dose intensity units will depend on treatment being summarized (belantamab mafodotin, lenalidomide, bortezomib, dexamethasone). Specifics on treatment units can be found in Section 8 of study protocol (Version: GSK Document Number TMF-14624358). Also, dose intensity for lenalidomide will be split by subjects with a first dose of 25mg versus those with a first dose of 10mg.

Relative dose intensity (RDI) will also be summarized for belantamab mafodotin, lenalidomide, bortezomib, and dexamethasone separately. For belantamab mafodotin, RDI will be split, with a calculation for Dose 1 and a separate calculation post-Dose 1. Relative dose intensity is calculated as a percent and is defined as 100\*(mean overall dose intensity divided by planned dose intensity). Planned dose intensity for each treatment is calculated as:

- Belantamab Mafodotin = planned dose of 1.9 mg/kg, 2.5 mg/kg, or 3.4 mg/kg. For the 2.5 S/D STRETCH dose, 2.5 mg/kg will be used for RDI at Dose 1 and 1.9 mg/kg will be used for RDI post-Dose 1.
- Lenalidomide = 525 mg for subjects with a first dose of 25mg, and 210 mg for subjects with a first dose of 10 mg.
- Bortezomib =  $5.2 \text{ mg/m}^2$
- Dexamethasone = 160 mg for subjects with a first dose of 40mg (Arm A) or 20mg (Arm B), and 80mg for subjects with a first dose of 20mg (Arm A) or 10mg (Arm B). For Arm B, if a subject's first dose is ≥20mg, their first dose will be considered 20mg for planned dose, and a first dose <20mg will be considered 10mg for planned dose.

#### **Summaries of Dose Modifications:**

The summaries of dose modifications will be provided. All the dose reductions, infusion interruptions, and dose delays will be summarized or listed.

Dose reductions will be summarised by number of reductions and reasons for reductions. Dose delays will be summarised by number of delays, reasons for the delays, and delay duration (days). The number and percentage of the delays for intervals of 1-28, 29-56 and >56 days for participants in Arm A, and 1-21, 22-42 and >42 days for participants in Arm B, will be computed. Primary reasons for dose reductions and dose delays will also be summarized by visit.

Duration of delays is defined as period from the expected start date of dose to actual start date of current dose:

- Calculation for SINGLE dose: (actual start date of current dose expected start date of dose). Expected start date of dose = actual start date of previous dose + 28 (Arm A), and actual start date of previous dose + 21 (Arm B).
- Calculation for SPLIT dose:
  - O Day 1: (actual start date of current dose − (actual start date of previous dose + 21) (Arm A), and (actual start date of current dose − (actual start date of previous dose + 14) (Arm B). For Arm A the previous dose must be a day 8 − 28 and for Arm B the previous dose must be a day 8 − 21. If the previous dose is a day 1, then use the same calculation used for SINGLE dose.
  - Day 8: (actual start date of current dose (actual start date of previous dose + 7) (Arms A and B). For Arms A and B, the previous dose must be a day 1 7. If the previous dose is not a day 1, then use the same calculation used for SINGLE dose.
- Calculation for STRETCH dose: (actual start date of current dose expected start date of dose). Expected start date of dose = actual start date of previous dose + 56 (Arm A), and actual start date of previous dose + 42 (Arm B).

#### **Duration of Follow-up:**

Duration of Follow-Up will be summarized for all participants and is defined as the time from first dose to last contact or death. Duration of Follow-up will also be summarized for subjects with ongoing follow-up, that is, subjects within the collection follow-up period, with status alive or unknown.

#### 6.6. Concomitant Medications

Concomitant medications will be coded using GSK Drug coding dictionary, summarized, and listed. The summary of concomitant medications will show the number and percentage of subjects taking concomitant medications by Ingredient. Multi-ingredient products will be summarized by their separate ingredients rather than as a combination of ingredients. Anatomical Therapeutic Chemical (ATC) classification Level 1 (Body System) information will be included in the dataset created but will not appear on the listing or summary.

Concomitant medications will be summarized by base ingredient. Each participant is counted once within each ingredient . For example, if a participant takes Amoxycillin on two separate occasions, the participant is counted only once under the ingredient "Amoxycillin". Note: In order to be considered a concomitant medication, the concomitant medication must have been taken at some point during the on-treatment study phase.


207497

Blood products or blood supportive care products with onset date within the on-treatment study phase will be included in the summary tables. The frequency and percentage of subjects using blood products and blood supportive care products after the start of study medication will be provided. Supporting listings will also be provided.

# 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

#### 7.1.1. Endpoint/Variables

#### **BOR**

Best Overall Response (BOR) is defined as the best confirmed response (stringent Complete Response [sCR] > Complete Response [CR] > Very Good Partial Response [VGPR] > Partial Response [PR] > Minimal Response [MR] > Stable Disease [SD] > Progressive Disease [PD] > Not Evaluable [NE]) from treatment start date until disease progression or initiation of new anti-cancer therapy, whichever is earlier, as assessed by the investigator per IMWG (2016). Details on derivation of confirmed response are provided in Table 6.

#### ORR

Overall Response Rate (ORR), defined as the percentage of participants with a confirmed PR or better (i.e., PR, VGPR, CR, and sCR) as the BOR, per IMWG (2016).

ORR at final analysis will be analyzed based on the confirmed responses, which will be derived based on the algorithm specified in Table 6. ORR at interim analyses should also be analyzed based on confirmed responses if available.

# 7.1.1.1. Derivation of Confirmed Response

The derivation of confirmed response shall be based on the algorithm specified in Table 6. The date of the first of the two consecutive assessments will be used as the date of the confirmed response.

Table 6 Response confirmation algorithm

| # | Response at the First Time Point | Response at Subsequent Disease Assessment <sup>1</sup> | Confirmed Response at the First Time Point |
|---|---|---|---|
| 1 | sCR | sCR | sCR |
| 2 | sCR | CR | CR |
| 3 | CR | sCR/CR | 1 |
| 4 | sCR/CR | VGPR | VGPR |
| 5 | VGPR | sCR/CR/VGPR | ] |
| 6 | sCR/CR/VGPR | PR | PR |
| 7 | PR | sCR/CR/VGPR/PR | |
| 8 | sCR/CR/VGPR/PR | MR | MR |
| 9 | MR | sCR/CR/VGPR/PR/MR | |
| 10 | sCR/CR/VGPR/PR/MR | SD | SD |
| 11 | sCR/CR/VGPR/PR/MR | PD (any reason) OR No subsequent disease assessment: subject died or discontinued study or started new anti-cancer therapy before further adequate disease assessment | SD |
| 12 | PD (due to reasons other than imaging, i.e., plasmacytoma or bone lesion) | PD (any reason) including PD after initiation of new anticancer therapy OR No subsequent disease assessment: subject died due to PD before further adequate disease assessment (including death due to PD after initiation of new anti-cancer therapy) | PD |
| 13 | PD (due to reasons other than imaging, i.e., plasmacytoma or bone lesion) | SCR/CR/VGPR/PR/MR/SD OR No subsequent disease assessment: subject died due to reasons other than PD before further adequate disease assessment OR No subsequent disease assessment: subject discontinued study before further adequate disease assessment | NE |
| 14 | sCR/CR/VGPR/PR/MR/PD<br>(due to reasons other than<br>imaging, i.e., plasmacytoma | No subsequent disease assessment: subject has not died, discontinued from study | Unconfirmed sCR/CR/VGPR/PR/MR/PD |

| # | Response at the First Time Point | Response at Subsequent<br>Disease Assessment <sup>1</sup> | Confirmed Response at the First Time Point |
|---|---|---|---|
| | or bone lesion) | or (except for PD) started new<br>anti-cancer therapy; but as yet<br>has no further adequate | Will be categorized as NE for final ORR analysis. |
| | | disease assessments | For ORR analysis in IA, the unconfirmed response (PR or better) will be counted as responder. |
| 15 | SD | Any | SD |
| | | OR No subsequent disease assessment | |
| 16 | PD due to imaging (plasmacytoma or | Any | PD |
| | bone lesion) | OR No subsequent disease assessment | |
| 17 | NE or missing | Any | NE |
| | | OR<br>No subsequent disease<br>assessment | |

<sup>1.</sup>Subsequent disease assessment is defined as the next not missing or NE disease assessment following the first timepoint before (or on the same date of) start of new anti-cancer therapy except for confirmation of PD, for which PD or death due to PD after new anti-cancer therapy are considered for confirmation of PD. No minimal time interval is required for the subsequent disease assessment, but a different sample is required for confirmation.

#### Note:

- SD does not need to be confirmed.
- PD due to imaging (i.e., plasmacytoma or bone lesion) does not need to be confirmed.
- Where criteria are not mutually exclusive, take the first that applies.
- As per IMWG criteria (Kumar, 2016), "If patients do not have measurable disease at baseline, they can only be assessed for at least a complete response or progressive disease."

### 7.1.2. Summary Measure

#### ORR

The number and percentage of participants with the BOR in the following response categories will be summarized at interim and final analysis for each treatment arm: sCR, CR, VGPR, PR, overall response (sCR+CR+VGPR+PR), minimal response (MR), stable disease (SD), progressive disease (PD), and not evaluable (NE). The corresponding exact 95% CI for ORR will also be provided. Participants with unknown or missing responses will be treated as non-responders, i.e., these participants will be included in the denominator when calculating percentages of response.

For subgroup analysis, ORR will be presented using forest plot for categories defined in Section 5.3.1.

## 7.1.3. Population of Interest

The primary efficacy analyses will be based on the All Treated population for all analyses, unless otherwise specified.

### 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12 and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 2.2 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed.













### 8. SAFETY ANALYSES

The safety analyses will be based on the All Treated population, unless otherwise specified.

# 8.1. Adverse Events Analyses

Adverse events (AEs), Serious AEs (SAEs) and other significant AEs will be analyzed based on GSK Core Data Standards. AE displays showing information by preferred term and max grade will use treatment emergent AEs. All other AE displays will use ontreatment AEs. Details for treatment-emergent and on-treatment AEs are provided in Section 15.2.3. Dose-limiting toxicity (DLT) will also be summarized according to GSK Oncology Data Standards. The details of the planned displays are provided in Appendix 12.

Adverse events will be graded by the investigator according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03 [NCI, 2010]. Adverse events will be coded using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary) and grouped by system organ class (SOC). In addition, corneal findings will also be graded using the GSK scale for corneal events provided in Table 9.

An overview summary of AEs, including counts and percentages of subjects with any AE, AEs related to GSK2857916/study treatment, Grade 3&4 AEs, Grade 3&4 AEs related to GSK2857916/study treatment, AEs leading to permanent discontinuation of study treatment, AEs related to GSK2857916/study treatment and leading to permanent discontinuation of study treatment, AE leading to dose reductions, AEs leading to dose interruption/delay, AEs leading to Infusion stopped early and no completed, SAEs, SAEs related to GSK2857916/study treatment, fatal SAEs, and fatal SAEs related to GSK2857916/study treatment will be produced.

A summary of non-serious AEs that occurred in 5% of the subjects or above will be provided (no rounding for the percentage will be used in terms of 5% threshold, e.g., event with 4.9% incidence rate should not be included in this table). SOC and PT. will display the summary

The relationship between MedDRA PT, and Verbatim Text will be displayed.

A summary of number and percentage of subjects with any AEs by maximum grade will be produced. Adverse events will be sorted by Preferred term (PT) in descending order of total incidence. The summary will use the following algorithms for counting the subject:

- **Preferred term row:** Participants experiencing the same AE preferred term several times with different grades will only be counted once with the maximum grade.
- **Any event row:** Each participant with at least one adverse event will be counted only once at the maximum grade no matter how many events they have.

In addition, the frequency and percentage of AEs (all grades) will be summarized and displayed in three ways: 1) in descending order of total incidence by PT only, 2) in descending order of total incidence by System Organ Classes (SOC) and PT, and 3) in descending order of total incidence by System Organ Classes (SOC) and PT and Maximum Grade. In the SOC row, the number of subjects with multiple events under the same system organ class will be counted once.

A separate summary will be provided for study treatment-related AEs. A study treatment-related AE is defined as an AE for which the investigator classifies the relationship to study treatment as "Yes". A worst-case scenario approach will be taken to handle missing relatedness data, i.e., the summary table will include events with the relationship to study treatment as 'Yes' or missing. The summary table will be displayed in descending order of total incidence by PT and Maximum Grade.

A summary of the number of patients experiencing DLTs will be provided.

To understand the impact of COVID-19, the following displays will be provided:

• Number of subjects with suspected, probable, or confirmed for COVID-19 infection

Details on how to define when COVID-19 pandemic measures began are provided in Section 15.10.

# 8.2. Adverse Events of Special Interest Analyses

#### 8.2.1. Belantamab Mafodotin

Characteristics (e.g., number of occurrences, action taken, maximum grade, etc.) of the following AEs of special interest related to belantamab mafodotin will be summarized separately:

- Corneal events, Keratopathy events
- Thrombocytopenia
- Infusion related reactions

For thrombocytopenia and infusion-related reactions (IRR), in addition to events identified and collected in eCRF, a comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Other AESI will be identified based on list of terms of interests which will be produced in Integrated Coding Dictionary System by Clinical Dictionary Development & Management and provided to Statistics and Programming. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. The details of the planned displays are provided in Appendix 12.

For infusion related reactions, events would only be considered IRR if the event was reported on an infusion day after the start of infusion or within 24 hours following end of infusion, and led to a temporary interruption or prolongation of infusion time or treatment withdrawal.

The severity of all AESI will be graded utilizing the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) v.4.03 [NCI, 2010]. Severity of belantamab mafodotin treatment related corneal events will also be graded using the GSK scale for corneal events provided in Table 9 and should be used for evaluation of DLT. Additional guidance on grading visual acuity changes is provided in Section 15.3.5.

| Table 9 | Grading Scale <sup>a</sup> for Corneal Events Associated with Belantamab |
|---|---|
| | Mafodotin |

| Measure | Grade 1 per GSK | Grade 2 per GSK Scale | Grade 3 per GSK Scale | Grade 4 per GSK |
|---|---|---|---|---|
| | Scale | | | Scale |
| Ophthalmic | Mild superficial | Moderate punctate | Severe punctate | Corneal ulcer |
| exam findings | keratopathy | keratopathy | keratopathy | |
| | (change from | and/or | and/or | |
| | baseline) | Mild/patchy microcysts | Diffuse microcysts | |
| | | and/or | and/or | |
| | | Mild/patchy Epithelial or | Diffuse Epithelial or | |
| | | stromal edema | stromal edema | |
| | | and/or | and/or | |
| | | Sub-epithelial haze | Sub-epithelial haze | |
| | | (peripheral) | (central) | |
| | | and/or | and/or | |
| | | Active stromal opacity | Active stromal opacity | |
| | | (peripheral) | (central) | |
| Visual Acuity | Change of 1 line | Change of 2-3 lines from | Change of more than 3 | Worse than Vision |
| b, c | from baseline | baseline and not worse<br>than 20/200b | lines from baseline and not worse than 20/200b | 20/200b |
| | | (11d11 20/200° | WUISE (Hall ZU/ZUU | |

Note: Standardized guidance for grading ophthalmic findings associated with GSK2857916 is provided to sites in the eCRF and ophthalmology SRM information. Ophthalmic exam findings as described must be present in a participant to utilize the GSK grading scale.

- Grading is based on most severe finding. If eyes differ in severity, GSK grading scale should be based on the more severe eye.
- b. Change in visual acuity should be due to corneal events associated with GSK2857916. If change in vision is for reason other than corneal events, ophthalmic exam findings will drive event grading.
- c. See Section 15.3.5 for additional guidance on how to grade changes in visual acuity depending on baseline vision. If a participant has a baseline visual acuity of 20/200 or worse in an eye, ophthalmic exam findings will drive event grading

Summaries of the number and percentage of subjects with these events will be provided for each type of events separately by preferred term and maximum grade. The time of onset and duration of first occurrence for some events will be summarized using summary statistics mean, standard deviation, median, minimum value, and maximum. The number and percentage of subjects who have time of onset of first occurrence (1-28, 29-56, 57-84, >84 days for Arm A, and 1-21, 22-42, 43-63, >63 days for Arm B) will be reported. The number and percentage of subjects who have duration of first occurrence (1-28, 29-56, >56 days for Arm A, 1-21, 22-42, >42 days for Arm B) will be reported.

The summary of event characteristics will also be provided, including number of subjects with event, number of events, event characteristics (serious, study treatment related), number of events per subject (one, two, three or more), worst outcome (recovered/resolved, recovered/resolved with sequelae, recovering/resolving, not recovered/not resolved, fatal), and maximum grade. The percentage will be calculated in two ways, one with number of subjects with event as the denominator and the other with total number of subjects as the denominator, within each cohort and treatment group. The worst-case approach will be applied at subject level for the maximum grade, i.e., a subject will only be counted once as the worst case from all the events experienced by the subject. For action taken to an event, subject will be counted once under each action, e.g.,

if a subject has an event leading to both study treatment discontinuation and dose reduction, the subject will be counted once under both actions.

#### 8.2.1.1. Other Risks

Characteristics (e.g., number of occurrences, action taken, maximum grade, etc.) of the important other risk, neutropenia, will be summarized separately. The severity of neutropenia will be graded utilizing the NCI-CTCAE v.4.03 [NCI, 2010].

A comprehensive list of MedDRA preferred terms for neutropenia based on clinical review will be used to identify each type of event. Neutropenia will be identified based on list of terms of interests which will be produced in Integrated Coding Dictionary System by Clinical Dictionary Development & Management and provided to Statistics and Programming. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional risks; therefore, the list of terms to be used for each event and the specific events will be based on the safety review team (SRT) agreements in place at the time of reporting. The details of the planned displays are provided in Appendix 12.

Summaries of the number and percentage of subjects with these events will be provided for each type of events separately by preferred term and maximum grade.

The summary of event characteristics will also be provided and will be calculated similarly as the AESI for belantamab mafodotin as provided in Section 8.2.

# 8.2.2. Corneal events (GSK scale)

Following discussions with regulatory agencies, GSK developed a grading scale to capture both corneal examination findings and visual acuity changes in participants treated with belantamab mafodotin. This GSK scale differs from the CTCAE criteria for eye disorders which relies mainly on patient's symptoms and patient's ability to attend to 'activities of daily living' for grading of events. Details of derivation of this GSK scale based on corneal findings and visual acuity Ophthalmic Exam (collected from Ocular form) can be found in Table 33 and Table 34 of study protocol (Version: GSK Document Number TMF-14624358).

In addition to the listing, the following outputs will be provided for corneal events graded using the GSK scale:

- 1. Overview for corneal event (GSK scale)
- 2. Summary of Grade of GSK scale
  - a. Summary of Characteristics of Corneal Events (GSK scale) including the percentage of duration of exposure (see Section 15.4.2 for definition) that is having corneal events (GSK scale) with grade  $\geq 2$  and grade  $\geq 3$  respectively

- b. Summary of onset time and duration of the first occurrence of corneal event (GSK scale) of grade 2 or above
- 3. Summary of actions taken with study treatment (e.g., dose reduction/delay/study treatment withdrawn)
- 4. Summary of worst post-baseline corneal events (GSK scale)
- 5. Summary of Best Corrected Visual Acuity Test (BCVA) Scores (logMAR score) due to Corneal Event (GSK Scale)

Exposure-adjusted incidence rates for grade 3+ corneal events (GSK Scale) will be summarized. Exposure-adjusted rates (rate/100 PY) are defined as the number of participants with an occurrence of a grade 3+ corneal event (first occurrence in worse eye, max grade, GSK Scale), divided by the total exposure duration in years across all participants at risk within a dose group, multiplied by 100. Exposure duration in years for each participant is calculated as:

- For participants who do not experience a grade 3+ corneal event: (Duration of Exposure (as defined in Section 6.5)) / 365.25
- For participants that do experience a grade 3+ corneal event: (Date of first max grade 3+ corneal event in worse eye (GSK Scale) first dose date + 1) / 365.25

For recurring grade 3+ events, the first occurrence of the event will be reported.

Details of the planned displays are provided in Appendix 12.

### 8.2.3. Eye Disorder (CTCAE)

A summary of characteristics of blurred vision events (CTCAE) will be provided, including number of subjects with an event, total number of events, event characteristics (serious, related to GSK2857916, related to any study treatment), number of events per subject, worst outcome, maximum grade, and action taken.

#### 8.3. Deaths and Serious Adverse Events

All deaths will be summarised based on the number and percentage of participants. This summary will classify participants by time of death relative to the last dose of treatment (>30 days or  $\leq$ 30 days) and primary cause of death (disease under study, SAE possibly related to study treatment, or other).

All SAEs will be tabulated based on the number and percentage of subjects who experienced the event. Separate summaries will also be provided for study treatment-related SAEs. The summary tables will be displayed in descending order by PT. The summary of all SAEs will also be created by SOC and PT. In addition, a summary of cumulative incidence of SAE by number of doses received at first occurrence will be provided.

A study treatment-related SAE is defined as an SAE for which the investigator classifies the relationship to study treatment as "Yes". A worst-case scenario approach will be taken to handle missing data, i.e., the summary table will include events with the relationship to study treatment as 'Yes' or missing.

SAEs are included in the listing of all adverse events. Separate supportive listings with participant-level details will be generated for

Fatal SAEs

# 8.4. Adverse Events Leading to Discontinuation and Dose Modification

The following categories of AEs will be summarized separately in descending order of total incidence by PT and separate supportive listings will be generated with participant level details for those participants:

- AEs Leading to Permanent Discontinuation of Study Treatment
- AEs Leading to Dose Interruptions or Delays
- AEs Leadings to Dose Reductions

Additionally, dose modifications will be assessed separately for all AEs, corneal AEs, and non-corneal AEs.

# 8.5. Ocular findings from ophthalmic exam

As outlined in study protocol (Version: GSK Document Number TMF-14624358) Schedule of Activities, ophthalmic exams are scheduled at screening, during the study, and follow-up period for subjects in study. The ocular findings from ophthalmic exams will be analysed as described below.

- 1. Ocular findings for General study (Baseline to Last follow-up):
  - a. Summary of Best Corrected Visual Acuity Test (BCVA) Scores (logMAR score), and Summary of Best Corrected Visual Acuity Test (BCVA) Scores (logMAR score) due to Corneal Event (GSK Scale) includes summaries of BCVA (logMAR score) at baseline, EOT visit, and last follow-up visit as well as worst and most frequent category (definite worsen, possible worsen, and no change/improved) of change from baseline summarized by eye (R/L) and subject (better eye). Changes of logMAR score from baseline to end of treatment visit, last follow-up exam and maximum (worst) change from baseline will be summarized based on the following categories: no change/improved vision: a change from baseline <0.12; a possible worsened vision: a change from baseline >=0.12 to <0.3; a definite worsened vision: a change from baseline >=0.3.
  - b. Number (%) of Subjects with a Decline in Best Corrected Visual acuity (BCVA) to LP or NLP due to a Corneal Event Anytime Post-Baseline

- c. Summary of Worst Post-Baseline Best Corrected Visual Acuity (BCVA) Change in Snellen Results
- d. Shift in Corneal Epithelium Findings from Baseline to Worst Post-Baseline
- e. Summary of Findings for Punctate Keratopathy

The details of the planned displays are provided in Appendix 12.

## 8.6. Pregnancies

While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy for medical reasons will be recorded as an AE or SAE as described in the protocol. If participants and participants' partner become pregnant while on the study, the information will be included in the narratives and no separate table or listing will be produced.

# 8.7. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12. Summary of change from baseline by scheduled visits using mean, median, standard deviation, minimum and maximum will be provided.

Summaries of worst-case grade increase from baseline grade will be provided for all the lab tests that are gradable by CTCAE v4.03. These summaries will display the number and percentage of subjects with a maximum post-baseline grade increasing from their baseline grade. Any increase in grade from baseline will be summarized along with any increase to a maximum grade of 3 and any increase to a maximum grade of 4. Missing baseline grade will be assumed as grade 0. For laboratory tests that are graded for both low and high values, summaries will be done separately and labelled by direction, e.g., sodium will be summarized as hyponatremia and hypernatremia.

For lab tests that are not gradable by CTCAE v4.03, summaries of worst-case changes from baseline with respect to normal range will be generated. Decreases to low, changes to normal or no changes from baseline, and increases to high will be summarized for the worst-case post-baseline. If a participant has a decrease to low and an increase to high during the same time interval, then the participant is counted in both the "Decrease to Low" categories and the "Increase to High" categories.

Separate summary tables for haematology, and chemistry laboratory tests will be produced. Liver function laboratory tests will be included with chemical chemistry.

Detailed derivation of baseline assessment is specified in Section 5.2. Unless otherwise specified, the denominator in percentage calculation at each scheduled visit will be based on the number of subjects with non-missing value.

Unless otherwise specified, the denominator in percentage calculation at each scheduled visit will be based on the number of subjects with non-missing value.

# 8.8. Other Safety Analyses

#### 8.8.1. ECG

The analyses of non-laboratory safety test results including ECGs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12.

A summary of the number and percentage of subjects who had normal and abnormal (clinically significant and not clinically significant) ECG findings will be displayed by scheduled visits as well as for the worst-case post-baseline.

The QTc values based on Fridericia formula will be rounded to the integer and the values will be categorized into the following ranges: Grade 0 (<450), Grade 1 (450-480), Grade 2 (481-500), and Grade 3 (≥501). Summaries of grade increase will be provided for some analyses. These summaries will display the number and percentage of subjects with any grade increase.

The changes in QTc values will be categorized into the clinical concern ranges which are specific to changes in QTc: 31-60, and >60 msec, and >530msec. A summary of change in QTc value will display the number and percentage of subjects with a change within each range in the worst-case post-baseline only. Subjects with missing baseline values will be excluded from this summary.

The summaries of QTc will use the collected values based on Fridericia formula.

# 8.8.2. Anti-Drug Antibody Analyses

For each subject, the anti-GSK2857916 (drug) antibody results, titers, and neutralizing antibody assay results, and also ADC and total antibody concentration will be listed for each assessment time point. The frequency and percentage of subjects with positive and negative anti-drug antibody and neutralizing antibody assay results will be summarized for each assessment time and overall, for each subject by dose cohort. The conclusive results will be based on the total antibody concentration.

#### 8.8.3. Profile Plot

A profile plot for subjects within both Arms A and B will be produced. This plot will display Study Treatment Duration (Days) for each subject, along with an indication of each subject's actual dose over time, investigator assessed confirmed response, highlighting responders versus non-responders, and those ongoing on belantamab mafodotin study treatment (ongoing indicator at interims only).

## 9. PHARMACOKINETIC ANALYSES

Concentration-time data collected will be analyzed using standard non-compartmental methods; some parameters will be determined for all participants and cycles. The concentration-time data may be combined with data from other studies and will be analyzed in a population approach using nonlinear mixed effects modeling and may be provided in a separate report.

For all mean and median measures within tables or figures, means/medians will only be calculated if the number of evaluable samples is greater than or equal to 3. Similarly, standard deviation and coefficient of variation measures will only be calculated for samples greater than or equal to 3.

# 9.1. Drug Concentration Measures

Plasma concentrations of belantamab mafodotin, total mAb, and cys-mcMMAF will be summarized using descriptive statistics, graphically presented (where appropriate) and listed by treatment arm and dose group. All dose groups will be on each figure as appropriate (Refer to Appendix 3 (Section 15.3)).

Linear and semi-logarithmic individual concentration-time profiles and mean and median profiles (when appropriate) will be plotted for lenalidomide and bortezomib. Concentrations of bortezomib and lenalidomide will be listed for each participant and summarized (when appropriate) by planned time point.

#### 9.2. Derived Pharmacokinetic Parameters

# 9.2.1. Belantamab Mafodotin, Total mAb, and Cys-mcMMAF

Pharmacokinetic analyses of derived pharmacokinetic parameter values of belantamab mafodotin, total mAb, and/or cys-mcMMAF will be conducted based on the Pharmacokinetic (PK) Analysis Set, as data permit.

• The following pharmacokinetic parameters described in the table below will be determined separately for each analyte and dosing regimen, as data permit and as outlined in Table 10

Table 10 Derived Pharmacokinetic Parameters from NCA or Population PK analyses

| Parameter | Parameter Description |
|---|---|
| AUC(0-x) | Area under the concentration-time curve from time zero to time x (i.e., 168, 504, 672, 1008 hours) |
| AUC(0-τ) | Area under the concentration-time curve during the dosing interval |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data for each cycle. Cmax will not be derived when only predose and EOI samples were collected. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data for each cycle |
| Cτ, Ctrough | Trough concentration prior to the next dose for each cycle |
| C-EOI | Observed plasma concentration at the end of infusion |
| tlast | Time of last observed quantifiable concentration |

NOTES: Additional parameters may be included as required.

# Derived PK Parameters for Analytes and Dose Regimen for Arm A

| Analyte | Dosing Regimen | | |
|---|---|---|---|
| (Unit) | Single | Split | Stretch |
| Belantamab<br>mafodotin<br>(μg/mL)<br>AND<br>Total mAb<br>(μg/mL) | Cmax (C1D1)<br>Tmax (C1D1)<br>Tlast (C1D1)<br>AUC0-504h (C1D1)<br>AUC0-672h (C1D1) | Cmax (C1D1) Tmax (C1D1) Tlast (C1D1) AUC0-504h (C1D1) AUC0-672h (C1D1) Cmax (C1D8) Tmax (C1D8) | Cmax (C1D1) Tmax (C1D1) Tlast (C1D1) AUC0-504h AUC0-672h (C1D1) AUC0-1008h (C1D1) AUC0-1344 (C1D1) |
| cys-mcMMAF<br>(ng/mL) | Cmax (C1D1)<br>Tmax (C1D1)<br>Tlast (C1D1)<br>AUC0-168h (C1D1) | Cmax (C1D1) Tmax (C1D1) AUC0-168h (C1D1) AUC0-336h (C1D1) Tlast (C1D1) Cmax (C1D8) Tmax (C1D8) AUC0-168h (C1D8) | Cmax (C1D1)<br>Tmax (C1D1)<br>Tlast (C1D1)<br>AUC0-168h (C1D1) |

C1D1 is Cycle 1 Day 1 C1D8 is Cycle 1 Day 8

# Derived PK Parameters for Analytes and Dose Regimen for Arm B

| Analyta | Dosing Regimen | | |
|---|---|---|---|
| Analyte<br>(Unit) | Single | Split | Stretch and S/D<br>Stretch |
| Belantamab<br>mafodotin<br>(µg/mL)<br>AND<br>Total mAb<br>(µg/mL) | Cmax (C1D1)<br>Tmax (C1D1)<br>Tlast (C1D1)<br>AUC0-504h (C1D1) | Cmax (C1D1) Tmax (C1D1) Tlast (C1D1) AUC0-504h (C1D1) Cmax (C1D8) Tmax (C1D8) | Cmax (C1D1)<br>Tmax (C1D1)<br>Tlast (C1D1)<br>AUC0-504h (C1D1)<br>AUC0-1008h (C1D1) |
| cys-mcMMAF | Cmax (C1D1)<br>Tmax (C1D1) | Cmax (C1D1)<br>Tmax (C1D1) | Cmax (C1D1)<br>Tmax (C1D1) |

| (ng/mL) | Tlast (C1D1) | AUC0-168h (C1D1) | Tlast (C1D1) |
|---------|------------------|------------------|------------------|
| | AUC0-168h (C1D1) | AUC0-336h (C1D1) | AUC0-168h (C1D1) |
| | | Tlast (C1D1) | |
| | | Cmax (C1D8) | |
| | | Tmax (C1D8) | |
| | | AUC0-168h (C1D8) | |

C1D1 is Cycle 1 Day 1 C1D8 is Cycle 1 Day 8

- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin, version 6.3 or later, as data permit, or by population pharmacokinetic analysis (Section 11)
- The pharmacokinetic parameters C-EOI and Ctrough will be determined directly from the concentration-time dataset. Note: For the dosing occasions with only predose and end of infusion samples, the end of infusion sample will not be identified as Cmax. Ctrough will not be reported for cys-mcMMAF.
- All calculations of pharmacokinetic parameters will be based on actual sampling times.

#### 9.2.2. Lenalidomide and Bortezomib

Lenalidomide pharmacokinetics in the presence of belantamab mafodotin may be analyzed using standard non-compartmental methods, data permitting, according to the same methodology as described above, or analyzed using a published population pharmacokinetic model. Results of the population PK analysis may be provided in a separate report.

#### Lenalidomide PK parameters for Arm A

| Analyte | Dosing Regimen | | |
|---|---|---|---|
| (Unit) | Single | Split | Stretch |
| Bortezomib (ng/mL) | Cmax<br>Tmax<br>Tlast<br>AUC0-4<br>AUC0-24 | Cmax<br>Tmax<br>Tlast<br>AUC0-4<br>AUC0-24 | Cmax<br>Tmax<br>Tlast<br>AUC0-4<br>AUC0-24 |

Bortezomib pharmacokinetics (see table below) in the presence of belantamab mafodotin will be analyzed using standard non-compartmental methods, data permitting, according to the same methodology as described above.

# Bortezomib PK parameters for Arm A

| Analyte | Dosing Regimen | | | |
|---|---|---|---|---|
| (Unit) | Single | Single Split Stretch | | S/D Stretch |
| Bortezomib<br>(ng/mL) | Cmax<br>Tmax<br>Tlast<br>AUC0-last<br>AUC0-72h | Cmax<br>Tmax<br>Tlast<br>AUC0-last<br>AUC0-72h | Cmax<br>Tmax<br>Tlast<br>AUC0-last<br>AUC0-72h | Cmax<br>Tmax<br>Tlast<br>AUC0-last<br>AUC0-72h |

AUC0-last will be reported in the listings not in summary tables

# 9.3. Summary Measure

Parameters listed in Section 9.2 will be summarized.

# 9.4. Population of Interest

The pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

# 9.5. Statistical Analyses / Methods

Pharmacokinetic parameters will be listed and summarized descriptively (mean, standard deviation, median, minimum, maximum, geometric mean, and the standard deviation, CV%, and 95% CI of log-transformed parameters) by analyte, arm, dose group, and visit.

Details of the planned displays are provided in Appendix 12, based on GSK Standards and statistical principles.

# 10. PHARMACOKINETIC AND PHARMACODYNAMIC ANALYSES

# 10.1. Exposure-Response for Efficacy and Safety Endpoints

If deemed appropriate and if data permit, exposure-response relationships between belantamab mafodotin exposure (e.g., concentration, Cmax, or AUC) and clinical activity and/or toxicity (e.g., response, AESIs) may be explored using population methods. If data permit, the effects of covariates may be explored. Time to event endpoints will be analyzed using Kaplan-Meier plots and Cox proportional hazard models while probability of occurrence of event of interest will be evaluated using logistic regression.

These analyses will be performed using R (The R Foundation for Statistical Computing), NONMEM (ICON Solutions) with PsN (Perl Speaks NONMEM) or another software platform deemed appropriate. The analysis will be performed by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline using the currently supported versions of all software packages.

Results of this analysis may be provided in a separate report.

# 11. POPULATION PHARMACOKINETIC (POPPK) ANALYSIS

Plasma belantamab mafodotin, and/or cys-mcMMAF concentration-time data may be combined with data from other studies and analysed using a population pharmacokinetic approach. The objective of this analysis would be to derive individual pharmacokinetic parameter values.

Based on the individual *post hoc* parameters, derived pharmacokinetic parameter values (e.g., CL, Vss,  $t^{1/2}$ , AUC(0- $\tau$ )) will be generated on certain dosing occasions, data permitting (see Table 10). These values will be listed and summarized as described in Section 9.5.

The lenalidomide concentration-time data may also be analyzed following the above methodology, using a published population PK model for lenalidomide (Guglieri-Lopez, 2017).

Further details are provided in Section 15.8. The results of these analyses may be provided in a separate report.





### 13. PATIENT REPORTED OUTCOMES ANALYSES

All questionnaires will be collected electronically as Electronic Patient Reported Outcomes (ePRO). The EORTC QLQ-C30 (version 3.0), EORTC QLQ-MY20, and the PRO-CTCAE are three oncology-specific Health-Related Quality-of-Life (HRQoL) assessments that will be analysed in this study.

In addition, the impact of potential corneal event on function and health-related quality-of-life will be assessed with the use of two visual function questionnaires, the NEI-VFQ-25, and Ocular Surface Disease Index (OSDI).

The analyses for EORTC QLQ-C30, EORTC QLQ-MY20, PRO-CTCAE, NEI-VFQ-25, and OSDI will be based on the All Treated population, unless otherwise specified.

# 13.1. Compliance of PRO-CTCAE, OSDI, and EORTC QLQ-C30

A table to summarize the compliance of PRO-CTCAE, OSDI, and NEI-VFQ-25 and EORTC QLQ-C30 and EORTC-QLQ-MY20 by visit will be provided. The tables will include number of subjects remaining in study, number, and percentage of subjects with PRO-CTCAE score (based on first item), OSDI total score, NEI-VFQ-25 overall composite score, QLQ-C30 summary score, and QLQ-MY20 summary score. The percentage is calculated using number of subjects remaining in the study at given timepoint as denominator.

The frequency and proportion of missing data for each measure will be evaluated at each timepoint.

# 13.2. Patient Reported Outcome Version of the Common Term Criteria for Adverse Events (PRO-CTCAE)

The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in subjects on cancer clinical trials [Basch, 2014]. The PRO-CTCAE was designed to be used as a companion to the CTCAE, the standard lexicon for adverse event reporting in cancer trials. The PRO-CTCAE includes an item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE. PRO-CTCAE provides a systematic yet flexible tool for descriptive reporting of symptomatic treatment side effects in cancer clinical trials. In the present study, a subset of items selected from the PRO-CTCAE Version 1.0 Item library will be administered. The levels and related code values for PRO-CTCAE are shown below.

| | Levels and related code values | | | | |
|---|---|---|---|---|---|
| Response scale | 0 | 1 | 2 | 3 | 4 |
| Frequency | Never | Rarely | Occasionally | Frequently | Almost<br>Constantly |
| Severity | None | Mild | Moderate | Severe | Very severe |
| Interference | Not at all | A little bit | Somewhat | Quite a bit | Very much |
| Present/Absence | No | Yes | | | |

For each selected item from the library: proportion of PRO-CTCAE scores for attributes (frequency, severity and/or interference) will be presented with stacked bar charts by visit. Maximum PRO-CTCAE score at post-baseline for each item attribute will be summarized by counts and proportions. Proportion of patients with a maximum score of 3 or 4 for each item attribute (severe or very severe, frequently or almost constantly, quite a bit or very much) will also be reported. Proportions will be based on the number of patients with available data and subject with missing response will be excluded from analysis.

#### 13.3. Visual Function Questionnaires

## 13.3.1. National Eye Institute Function Questionnaire-25 (NEI-VFQ-25)

The NEI-VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question [Mangione, 2001]. The NEI-VFQ-25 generates the following vision-targeted sub-scales: global vision rating, difficulty with near vision activities; difficulty with distance vision activities; limitations in social functioning due to vision; role limitations due to vision; dependency on others due to vision; mental health symptoms due to vision; driving difficulties; limitations with peripheral vision, limitations with color vision; and ocular pain. Details of deriving domain scores and overall composite score can be found in Section 15.9.3.

For overall composite score and each of 11 sub-scale scores, the descriptive summary of the actual value and change from baseline by visit will be provided.

#### 13.3.2. Ocular Surface Disease Index

The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire designed to assess both the frequency of dry eye symptoms and their impact on vision-related functioning [Schiffman, 2000; Dougherty, 2011]. The OSDI has demonstrated good reliability, validity, sensitivity, and specificity, and can be used as a complement to other clinical and subjective measures of dry eye disease by providing a quantifiable assessment of dry eye symptom frequency and the impact of these symptoms on vision-related functioning.

For the OSDI, the total score will be calculated as well as scores for the three subscales (ocular symptom: item 1-3; visual related function: item 4-9; and environmental triggers: item 10-12).

The total OSDI score = ([sum of scores for all questions answered × 100]/[total number of questions answered ×4]). Subscale scores are computed similarly with only the questions from each subscale used to generate its own score. A score of 100 corresponds to complete disability (a response of "all of the time" to all questions answered), while a score of 0 corresponds to no disability (a response of "none of the time" to all questions answered). Therefore, decrease in score from baseline means improvement.

For total score and each of the three sub-scales, the descriptive summary of the actual value and change from baseline at selected time points will be provided. For the Vision-Related Functioning domain, the number and percentage of participants with post-baseline score worsening of  $\geq 12.5$  from baseline score will be summarized.

Plots of change from baseline (including baseline) and 95% confidence interval over time by visit, and at end of study treatment, last follow-up, and worst case post-baseline for total score will also be provided.

#### 13.4. Value Evidence and Outcome

# 13.4.1. European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core module (EORTC QLQ-C30)

The EORTC QLQ-C30 is a 30-item questionnaire containing both single- and multi-item measures [Aaronson, 1993]. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/QoL scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). Scores for each scale and single-item measure are averaged and transformed linearly to a score ranging from 0–100. Details of deriving domain scores (9 scales and 6 single items) and summary score can be found in Section 15.9.1.

- A high score for functional scales and for Global Health Status/QoL represent better functioning ability or Health-Related Qualify of Life (HRQoL), (higher score indicates improvement)
- whereas a high score for symptom scales and single items represents significant symptomatology [Proskorovsky, 2014]. (Lower score indicates improvement)

Descriptive summaries (mean, SD, median, min and max) of the actual value and change from baseline will be provided for EORTC QLQ-C30 domain scores. The number and percentage of participants with post-baseline score improved by  $\geq 10$  points, respectively from baseline score will be summarized. The number and percentage will be provided for each domain score.

Plots of change from baseline (including baseline) and 95% confidence interval over time by visit, and at end of study treatment, and worst case post-baseline for individual domains will also be provided.

# 13.4.2. European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 20-item Multiple Myeloma module (EORTC QLQ-MY20)

The EORTC QLQ-MY20 is a supplement to the QLQ-C30 instrument used in patients with multiple myeloma [Aaronson, 1993; Cocks, 2007]. The module comprises 20 questions that address four myeloma specific HRQoL domains: Disease Symptoms, Side Effects of Treatment, Future Perspective, and Body Image. Three of the four QLQ-MY20 domains are multi-item scales: Disease Symptoms (includes bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity); Side Effects of Treatment (includes drowsiness, thirst, feeling ill, dry mouth, hair loss, upset by hair loss, tingling hands or feet, restlessness/agitation, acid indigestion/heartburn, and burning or sore eyes); and Future Perspective (includes worry about death and health in the future, and thinking about illness). The Body Image scale is a single-item scale that addresses physical attractiveness. Details of deriving domain scores can be found in Section 15.9.2.

For each of four domain scores, the following summaries will be provided:

• The descriptive summary of the actual value and change from baseline by visit

Summary of the number (%) of patients with improvement in score  $\geq 10$  points by visit.

Plots of change from baseline (including baseline) and 95% confidence interval over time by visit, and at end of study treatment, and worst case post-baseline for disease domain will also be provided.

## 14. REFERENCES

Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Institute. 1993 Mar 3;85(5):365-76.

Basch E, Reeve BB, Mitchell SA, Clauser SB, Minasian LM, Dueck AC, et al. Development of the National Cancer Institute's patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE). J Natl Cancer Inst. 2014;106(9).

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics. 1982 Mar 1:29-41.

Cocks K, Cohen D, Wisløff F, Sezer O, Lee S, Hippe E, et al. An international field study of the reliability and validity of a disease-specific questionnaire module (the QLQMY20) in assessing the quality of life of patients with multiple myeloma. European Journal of Cancer. 2007 Jul 31;43(11):1670-8.

Dougherty BE, Nichols JJ, Nichols KK. Rasch analysis of the Ocular Surface Disease Index (OSDI). Invest Ophthalmol Vis Sci. 2011;52(12): 8630-8635.

Fayers et. al., The EORTC QLQ-C30 Scoring Manual (3rd Edition) 2001

GlaxoSmithKline Document Number TMF-14624358 Study ID207497. DREAMM-6: A Phase I/II, Open-label, Dose Escalation and Expansion Study to Evaluate Safety, Tolerability, and Clinical Activity of the Antibody-Drug Conjugate GSK2857916 Administered in Combination with Lenalidomide Plus Dexamethasone (Arm A), or Bortezomib Plus Dexamethasone (Arm B) in Participants with Relapsed / Refractory Multiple Myeloma – (DREAMM 6). Report Date 30-JUN-2022.

Guglieri-Lopez B, Perez-Pitarch A, Moes DJ, Porta-Oltra B, Climente-Martí M, Guchelaar HJ, et al. Population pharmacokinetics of lenalidomide in multiple myeloma patients. Cancer Chemother Pharmacol. 2017;79:189-200

Ji Y, Liu P, Li Y, Bekele BN. A modified toxicity probability interval method for dose-finding trials. Clin Trials. 2010;7:653-663.

Kumar S, et al. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. The Lancet Oncology. 2016;17: e328-e346.

Mangione CM, Lee PP, Gutierrez PR, Spritzer K, Berry S, Hays RD, et al. Development of the 25-item National Eye Institute Visual Function Questionnaire. Arch Ophthalmol. 2001;119(7):1050-8.

National Cancer Institute (NCI). CTCAE. National Cancer Institute (NCI), http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE 4.03; 2010. CTCAE Version 4.03.
Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44

Proskorovsky I., P. Lewis, C. D. Williams, K. Jordan, C. Kyriakou, J. Ishak, F. E. Davies. Mapping EORTC QLQ-C30 and QLQ-MY20 to EQ-5D in patients with multiple myeloma. Health Qual Life Outcomes. 2014 Mar 11; 12:35.

Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability, and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000;118(5):615-21.

### 15. APPENDICES

### 15.1. Appendix 1: Assessment Windows

No assessment windows will be applied.

## 15.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

### 15.2.1. Study Phases

Assessments and events will be classified according to the date/time of occurrence relative to date/time of first dose of study treatment.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 70 days |
| | For interim analyses when participants are still on treatment, Study Treatment Stop |
| | Date will be imputed following rules specified in Section 15.5.2.1. |
| Post-Treatment | Date > Study Treatment Stop Date + 70 days |

For assessment or event on the first dosing day, whether it is Pre-Treatment or On-Treatment should be based on time if available. If time is not available, the first dosing day (Day 1) is considered Pre-Treatment for ECOG, ECG, vital signs, liver events, lab tests, cardiac scan, and other safety domains, and On-Treatment for adverse events and concomitant medications.

Concomitant Medication and Blood and Blood Supportive Care Product start and end dates will be assigned to study time periods in relation to first dose of study treatment as defined below. The start date reference time variables and end date reference time flag variables will be added to the concomitant medications and blood and blood supportive products datasets, respectively.

- Start relative to treatment: Assign to 'BEFORE' if start date is prior to study treatment start date or if subject has not taken any study treatment or (start date is missing, and end date is before study treatment start date). Else assign to 'DURING' if the start date falls into the on-treatment period as defined above or if subject is ongoing (not all study treatment discontinuation records completed) or start date is missing. Else assign to 'AFTER' if start date is after the on-treatment period.
- End relative to treatment: Assign to 'BEFORE' if end date is prior to study treatment start date or if subject has not taken any study treatment. Else assign to 'DURING' if end date falls into the on-treatment period or if subject is ongoing (not all study treatment discontinuation records completed) or (end date is missing and start relative to treatment not 'AFTER'). Else assign to 'AFTER' if end date is after the on-treatment period or (end date is missing and start relative to treatment='AFTER').

Only on-treatment blood and blood supportive care products that start after the start of study treatment are included in the Blood Products and Blood Supportive Care Product summaries. Therefore, for summary tables, include blood and blood supportive care product records where start relative to treatment in ('DURING') and end relative to treatment in ('DURING','AFTER'). All data will be reported in listings.

Concomitant medication start relative to treatment and end relative to treatment flags are used to select data to include in the Concomitant Medication summaries as follows:

- Summary of Concomitant Medications: This summary will contain medications including those with start date prior to study treatment start date and continue (missing end date or end date after study treatment start date) on therapy. Note that any medications with start date and end date prior to study treatment start date will be excluded. In addition, any medication that was started during post-therapy will be excluded. Include concomitant medication records where start relative to treatment in ('BEFORE','DURING') and end relative to treatment in ('DURING','AFTER').
- Summary of Concomitant Medications with On-Therapy Onset: This summary will contain medications with start date after study treatment start date. In addition, any medication that was started during post-therapy (see above for definition of post-therapy) will be excluded. Include concomitant medication records where start relative to treatment in ('DURING') and end relative to treatment in ('DURING','AFTER').

### 15.2.2. Study Phases for Vital signs, ECG and Laboratory Values

| Study Phase | Definition |
|---------------|-----------------------------------|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date |

### 15.2.3. Treatment Emergent and On-treatment Flag for Adverse Events

Table 12 Treatment Emergent and On-treatment Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>Study Treatment Start Date ≤ AE Start Date ≤ min(Study Treatment Stop Date + 70 days, Start of Anti-Cancer Therapy)</li> <li>AE Start Date is missing</li> </ul> |
| On-treatment | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 70 days |

#### NOTES:

• Time of study treatment dosing and start time of AEs should be considered, if collected.

The "treatment emergent" definition of AEs will be used for all displays providing summaries by preferred term and maximum grade. All other AE displays will use the "on-treatment" definition.

# 15.3. Appendix 3: Data Display Standards & Handling Conventions

### 15.3.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : US1SALX00259 |
| HARP Compound | : arprod\gsk2859716\mid207497\ |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.1).</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for all tables. | |

### 15.3.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH or non-ICH listings
- Note: All displays (TLF) will use the term 'Subject' to reflect GSK Display Standards and CDISC SDTM/ADaM standards

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Reporting of data for PK related displays will be decided based on review of the data.
- Numeric data will be reported at the precision collected on the eCRF.
  - The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures, and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses, and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned assessments will be presented within the participant's listings.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
  - o For by planned time analysis, unscheduled visits will not be included.
  - o For worst-case analysis, unscheduled visits will be included.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### 15.3.3. Reporting Standards for Pharmacokinetic Data

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non- compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to SOP_314000: Non-Compartment Analysis of Clinical Pharmacokinetic Data [Note Concentration values will be imputed as per GUI_51487] |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| NONMEM/Pop PK<br>File | Not applicable. |
| NONMEM/PK/PD File | Not applicable. |
| Pharmacokinetic Para | meter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | The following PK parameters will be derived by the Programmer: Ctrough (predose) CEOI for each cycle, data permitting. Ctrough will not be derived for cys-mcMMAF. |
| Pharmacokinetic Para | meter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to [Standards for Handling NQ Impacted PK Parameters]. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |
| Untransformed PK parameter | tmax (TMAX), tlast (TLST) |

## 15.3.4. Extended Loss to Follow-up or Extended Time without an Adequate Assessment

For participants, if two or more scheduled disease assessments are missed and are then followed by an assessment of PD or death, will be censored at the last adequate assessment prior to PD or death. When the scheduled disease assessment is every 3 weeks, a window of 45 days (6 weeks + 3 day window) will be used to determine whether there was an extended time without adequate assessment. That is, if the time difference between PD/death and last adequate assessment is more than 45 days, then will be censored at the last adequate assessment prior to PD/death. When the scheduled disease assessment is every 4 weeks, a window of 59 days (8 weeks + 3 day window) will be used to determine whether there was an extended time without adequate assessment. That is, if the time difference between PD/death and last adequate assessment is more than 59 days, then will be censored at the last adequate assessment prior to PD/death.

In case there is no adequate assessment between first dose date and PD/death, and the time difference between PD/death and first dose date is more than 45 days (when disease assessment is every 3 weeks), or 59 days (when disease assessment is every 4 weeks), then will be censored at the first dose date.

# 15.3.5. Additional Guidance on Grading Based on Changes in Visual Acuity

| Baseline Vision (best corrected) | Grade 1<br>(Change of 1<br>line from<br>baseline) | Grade 2<br>(Change of 2-3 lines<br>from baseline and<br>not<br>worse than 20/200) | Grade 3 (Change of more than 3 lines from baseline and not worse than 20/200) | Grade 4<br>(Worse than 20/200) |
|---|---|---|---|---|
| 20/20 | 20/25 | 20/30 – 20/40 | 20/50 –20/200 | Worse than 20/200 |
| 20/25 | 20/30 | 20/40 – 20/50 | 20/60 –20/200 | Worse than 20/200 |
| 20/30 | 20/40 | 20/50 – 20/60 | 20/70 –20/200 | Worse than 20/200 |
| 20/40 | 20/50 | 20/60 – 20/70 | 20/80 –20/200 | Worse than 20/200 |
| 20/50 | 20/60 | 20/70 – 20/80 | 20/100 – 20/200 | Worse than 20/200 |
| 20/60 | 20/70 | 20/80 – 20/100 | 20/125 – 20/200 | Worse than 20/200 |
| 20/70 | 20/80 | 20/100 – 20/125 | 20/200 | Worse than 20/200 |
| 20/80 | 20/100 | 20/125 – 20/200 | N/A | Worse than 20/200 |
| 20/100 | 20/200 | 20/200 | N/A | Worse than 20/200 |

### 15.4. Appendix 4: Derived and Transformed Data

#### 15.4.1. General

### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables.

### Study Day for Safety

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Date ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### **Study Day for Efficacy**

- Calculated as the number of days from [First Dose Date/Randomization Date]:
  - Ref Date = Missing

- → Study Day = Missing
- Ref Date < [First Dose Date] → Study Day = Ref Date [First Dose Date/Randomization Date]</li>
- o Ref Date ≥ [First Dose Date] → Study Day = Ref Date [First Dose Date/Randomization Date] + 1

### **Change from Baseline**

- Change from Baseline = Post-Baseline Visit Value Baseline
- % Change from Baseline= 100 x (Post-Baseline Visit Value Baseline) / Baseline
- Maximum Increase/Decrease from Baseline = maximum (Increase/Decrease from Baseline)
- If either the Baseline or Post-Baseline Visit value is missing, Change from Baseline and % Change from Baseline is set to missing

### **Date of Response**

 For post-baseline disease assessments, the date of response (PR or better) is assigned to the latest date of disease assessments; for other response categories (MR, SD, NE, PD), the date of response is assigned to the earliest date of disease assessments.

### 15.4.2. Study Population

### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

- Arm A:
  - **SINGLE/SPLIT Doses:** Duration of Exposure = (Last Treatment Date+27) First Treatment Date + 1
  - STRETCH Doses: Duration of Exposure = (Last Treatment Date+55) First Treatment Date + 1
- o Arm B:
  - **SINGLE/SPLIT Doses:** Duration of Exposure = (Last Treatment Date+20) First Treatment Date + 1
  - STRETCH Doses: Duration of Exposure = (Last Treatment Date+41) First Treatment Date
     + 1
- The cumulative dose will be based on the formula:

### Cumulative Dose (mg/kg) = Sum of Dose at Each Dosing Interval

- Dose intensity will be calculated based on the formulas:
  - o Arm A:
    - SINGLE/SPLIT Doses: Dose intensity (mg/kg/4 week) = Cumulative Dose/((duration of exposure)/28)
    - STRETCH Doses: Dose intensity (mg/kg/8 week) = Cumulative Dose/((duration of exposure)/56)
  - o Arm B:
    - SINGLE / SPLIT Doses: Dose intensity (mg/kg/3 week) = Cumulative Dose/((duration of exposure)/21)
    - STRETCH Doses: Dose intensity (mg/kg/6 week) = Cumulative Dose/((duration of exposure)/42)

### 15.4.3. Safety

#### **Adverse Events**

### AEs of Special Interest (belantamab mafodotin)

- Corneal events
- Thrombocytopenia
- Infusion related reactions

#### **Duration of AE**

To report in months, divide the number of days by 30.4375; to report in weeks divide the number of days by 7; to report in years divide the number of days by 365.25.

- Calculated as the number of days from AE Start Date to AE Stop Date:
  - AE Start Date = Missing
- → Elapse Time = Missing
- AE Stop Date = Missing
- → Elapse Time = Missing

o Otherwise

→ Elapsed Time = AE Stop Date – AE Start Date + 1

### **ECHO/MUGA**

 Change from Baseline for cardiac data, e.g., Left Ventricular Ejection Fraction (LVEF), will be calculated based on the same modality (ECHO or MUGA) throughout the study for each participant. Post-baseline assessments with a different cardiac scan modality will not be used to calculate change from Baseline.

#### DLT

#### **DLT Evaluable**

A DLT evaluable participant is defined as any participant in Part 1 who received at least 1 full dose of GSK2857916 and ≥75% of the planned doses of the combination with Len/Dex (Arm A), or Bor/Dex (Arm B) in Cycle 1 will be evaluated for DLTs using NCI-CTCAE Version 4.03 [NCI, 2010]. Any participant who received at least 1 full dose of belantamab mafodotin and at least 75% of planned doses of the respective Arm SoC (Len/Dex – Arm A or Bor/Dex – Arm B) will also be considered DLT-evaluable. Participants that are not DLT-evaluable will be replaced.

### 15.4.4. Biomarker and/or Pharmacodynamic Data

### Pharmacodynamic biomarkers

### 15.5. Appendix 5: Reporting Standards for Missing Data

### 15.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>A participant will be considered to have completed the study if he or she received at<br/>least one dose of study treatment and has progressed or died before the end of the<br/>study, has not been lost to Follow-up, or has not withdrawn consent from study<br/>participation, or the study or a treatment arm has been terminated.</li> </ul> |
| | A participant will be considered to have withdrawn from the study if the participant has not died and is lost to Follow-up, or has withdrawn consent, or is no longer being followed at the investigator's discretion |
| | Documentation of the cause of death in the electronic case report form (eCRF) is required for all participants who die in the study regardless of the cause of death. |
| | Withdrawn participants for reasons other than toxicity, but prior to completion of DLT period will be replaced in the study. |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

### 15.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | <ul> <li>Any participants excluded from the summaries and/or statistical analyses will be<br/>documented along with the reason for exclusion in the clinical study report.</li> </ul> |

### 15.5.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in participant listing displays. However, where necessary, display macros may impute dates as temporary variables for sorting data in listings only. In addition, partial dates may be imputed for 'slotting' data to study phases (see Section 15.2.1) or for specific analysis purposes as outlined below.</li> <li>Imputed dates will not be used to derive study day, time to onset or duration (e.g., time to onset), or elapsed time variables (e.g., time since diagnosis). In addition, imputed dates are not used for deriving the last contact date in analysis dataset.</li> </ul> |
| Adverse Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.</li> <li>Partial dates for AE recorded in the CRF will be imputed using the following conventions:</li> <li>Missing start day</li> <li>If study treatment start date is missing (i.e., participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date, then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date, then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> </ul> </li> </ul> |
| | <ul> <li>Else set start date = 1st of month.</li> <li>Missing start day and month</li> <li>Else if study treatment start date is missing (i.e., participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date, then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date, then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> <li>Missing Last day of the month will be used.</li> </ul> |
| | Stop day Missing stop day and month Completely missing start/end date No imputation |
| Concomitant<br>Medications/<br>Blood Supportive<br>Products | <ul> <li>Completely missing start dates will not be imputed</li> <li>Partial start dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If day and month are missing:</li> <li>If treatment start date is missing (i.e., subject did not start study treatment), a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>If treatment start date is not missing</li> </ul> </li> </ul> |

| Element | Reporting Detail |
|---|---|
| | If year of start date = year of study treatment start date |
| | If stop date contains a full date which is earlier than the treatment start date, a '01' will be used for the day and 'Jan' will be used for the month. |
| | · else study treatment start date will be used |
| | <ul> <li>else a '01' will be used for the day and 'Jan' will be used for the<br/>month</li> </ul> |
| | <ul> <li>If medication was taken prior to study, a '01' will be used for the day and 'Jan' will be used for the month.</li> </ul> |
| | <ul> <li>If day is missing: <ul> <li>If treatment start date is missing (i.e., subject did not start study treatment), a '01' will be used for the day.</li> <li>If treatment start date is not missing</li> <li>If year and month of start date = year and month of study treatment start date</li> </ul> </li> </ul> |
| | <ul> <li>If stop date contains a full date which is earlier than the treatment start date, a '01' will be used for the day.</li> <li>else study treatment start date will be used</li> <li>else a '01' will be used for the day and 'Jan' will be used for the</li> </ul> |
| | month |
| | Completely missing end dates will not be imputed |
| | Partial end dates for any concomitant medications recorded in the CRF will be imputed using the following convention: # days and reports are recipied: |
| | <ul> <li>If day and month are missing</li> <li>Earliest of (Dec 31<sup>st</sup>, date of last contact) will be used</li> </ul> |
| | <ul> <li>If day is missing</li> <li>Earliest of (last day of the month, date of last contact) will be used</li> </ul> |
| New Anti-Cancer<br>Therapy/<br>Radiotherapy/<br>Surgical<br>Procedures for<br>Efficacy<br>Evaluation (e.g., | Start dates for follow-up anti-cancer therapy, radiotherapy (where applicable), and surgical procedures (where applicable) will be imputed in order to define event and censoring rules for the surgical procedures. Dates will only be imputed. |
| | when a month and year are available but the day is missing. The following rules will be used to impute the date when partial start dates are present on anti-cancer therapy, radiotherapy, and/or surgical procedures dataset[s]: |
| response rate, | Completely missing start dates will remain missing, with no imputation applied. |
| time to event) | Partial start dates will be imputed using the following convention: |
| | <ul> <li>If both month and day are missing, no imputation will be applied.</li> </ul> |
| | If only day is missing: |
| | <ul> <li>If the month of partial date is the same as the month of last dosing date,<br/>minimum of (last dosing date + 1, last day of the month) will be used for<br/>the day.</li> </ul> |
| | <ul> <li>If the month of partial date is the same as the month of last disease<br/>assessment and the last disease assessment is PD, minimum of (last<br/>date of disease assessment + 1, last day of the month) will be used for<br/>the day.</li> </ul> |
| | <ul> <li>If both conditions above are met, the later date will be used for the day.</li> <li>Otherwise, a '01' will be used for the day.</li> </ul> |

| Element | Reporting Detail Completely or partial missing end dates will remain missing, with no imputation applied; |
|---|---|
| Treatment end date | <ul> <li>Imputation of missing treatment end date will be applied to all applicable<br/>treatments following rules below and treatment end date is the latest treatment<br/>end date across all study treatments.</li> </ul> |
| | For daily oral treatment: |
| | <ul> <li>In general, completely missing end dates are not imputed, with the following exceptions for imputation of missing treatment end date at interim analyses.</li> <li>For imputation of missing exposure end date at an interim analysis when participants are still on treatment, the following conventions will be applied: If the missing end date is in the last exposure record, the earliest of: the date of the data cut-off, the date of withdrawal from the study, or the death date will be used</li> <li>If the missing end date is not in the last exposure record, treatment start date for the record will be used</li> <li>The imputed treatment end date will be used to calculate cumulative dose and duration of treatment as specified in Section 15.4.2.</li> </ul> |
| | For non-continual treatment: • If treatment end date is missing for a cycle, treatment start date for the cycle will be used. |

### 15.6. Appendix 6: Values of Potential Clinical Importance

To identify laboratory values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v [4.03]) will be used to assign grades for laboratory parameters including clinical chemistry, haematology, liver function tests, thyroid function tests, pancreatic enzyme tests, QTc (Bazett's or Fridericia's) values, vital signs (heart rate, blood pressure, temperature) and LVEF.

Reference ranges for all laboratory parameters collected throughout the study are provided by the central laboratory, or local laboratory if applicable. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data. Clinical laboratory test results outside of the reference range will be flagged in the listings.

### 15.7. Appendix 7: Pharmacokinetic / Pharmacodynamic Analyses

### 15.7.1. Pharmacokinetic / Pharmacodynamic Dataset Specification

If deemed appropriate and if data permit, exposure-response analyses may be conducted using population methods to explore the relationship between exposure measures of belantamab mafodotin (ADC and/or cys-mcMMAF) and clinical activity and/or toxicity endpoints (e.g., response, AESIs).If data permit, the effects of covariates may be explored.

Exposure-response analyses will use the same systems and data assembly process as described in Appendix 8.

The final popPK models for both ADC and cys-mcMMAF will be applied to generate the following *post hoc* exposure measures to be used in efficacy and safety exposure-response analyses: ADC maximum concentration (ADC Cmax), ADC trough concentration (ADC Ctau), ADC average concentration (ADC Cavg), cys-mcMMAF Cmax, and cys-mcMMAF Cavg.

Time to events endpoints will be analyzed using Kaplan-Meier plots and coxproportional hazard models while probability of occurrence of event of interest will be evaluated using logistic regression.

For each exposure-response analysis, univariate analysis will be performed first to identify the strongest individual associations of exposure and other relevant covariates to clinical endpoint using change in the objective function. Following the univariate analysis, covariate selection will be conducted using a stepwise forward inclusion and backward elimination method to determine the final multivariate model. Covariates would be retained in the model in a stepwise manner if their inclusion during forwarding addition decreased the objective function value (OFV) by  $\geq$ 6.64 (P<0.01) over the previous model, with the most significant covariate being retained at each stage. This iterative process will continue until all significant covariates are included, thus defining the full model. From the full model, the significance of each covariate will be tested individually by removing one by one until all non-significant covariates have been excluded. A covariate will be retained if, upon removal, the OFV increased by more than 10.83 points (P<0.001). The final model is defined as the model developed following the backward elimination step.

The results of these analyses may be provided in a separate report.

### 15.7.2. Pharmacokinetic / Pharmacodynamic Methodology

Details may be provided in a separate exposure-response analysis RAP

### 15.8. Appendix 8: Population Pharmacokinetic (PopPK) Analyses

Belantamab mafodotin, total mAb and/or cys-mcMMAF plasma concentration-time data will be analyzed by Pop PK methods using a non-linear mixed-effects modelling approach.

The key objective of this analysis is to:

• Predict individual pharmacokinetic parameter values for belantamab mafodotin, and/or cys-mcMMAF

### 15.8.1. Systems

The population PK analysis will be performed using NONMEM (ICON Solutions) and PsN (Perl Speaks NONMEM) or another software platform deemed appropriate. Graphical displays and data summary will be produced using R (The R Foundation for Statistical Computing). The analysis will be performed by, or under the direct auspices of, Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline using the currently supported versions of all software packages.

### 15.8.2. Data Assembly

Participant data will be collected in the electronic CRF and will be transmitted into a validated database by GSK data management. Derived/processed variables will be provided by or under the guidance of Clinical Programming. Plasma samples will be analyzed using approved analytical methodology. Data will be transferred electronically to data managers to be processed and stored in the GSK database. GSK or a designated third party will generate the NONMEM input dataset.

Previously generated belantamab mafodotin and/or cys-mcMMAF PK data may be merged with the PK data in order to provide a pooled NONMEM data set.

### 15.8.3. Model Development

The initial analysis will use the population pharmacokinetic model developed for Study BMA117159 and Study 205678; a more current population PK model may be used, if available.

Initially, empirical Bayes estimates will be derived applying the current PopPK model to the Study 207497 dataset with the MAXEVAL=0 option. If the corresponding model diagnostics indicate that this PopPK model is appropriate to represent the belantamab mafodotin, total mAb and/or cys-mcMMAF data from Study 207497 then individual PK parameter estimates will be based on the current PopPK parameters.

If the parameter set of the current PopPK model applied to the Study 207497 data set results in substantial bias or if a further exploration of the covariate effect in the Study 207497 population is deemed necessary, the parameters of the current PopPK model will be re-estimated for the Study 207497 PK data alone before generating the individual PK parameter estimates and/or for a pooled data set. Certain parameter values may be fixed

to the value in the current PopPK model if they cannot be estimated with sufficient precision within the Study 207497 PK population. Covariates not available for the Study 207497 PK population but present in the current PopPK model may be removed from the Study 207497 PopPK model. Lastly, a model refinement step, if needed, will include, but may not be limited to, a qualification and possible modification of the model's random effect structure.

### 15.8.4. Model Qualification

Any model development will be supported and the final model will be qualified using the following criteria where appropriate:

- Scientific plausibility of parameter estimates
- Goodness of fit plots
- Relative standard errors (RSE) of the parameter estimates
- Objective function value
- Distribution and shrinkage of random effects.
- Successful minimization and execution of covariance step
- Condition number (ratio of the largest and smallest eigenvalue of the covariance matrix
- Visual predictive check
- Bootstrap (if deemed necessary/feasible)

### 15.9. Appendix 9: Patient Reported Outcomes

### 15.9.1. EORTC QLQ-C30

The EORTC QLQ-C30 is a 30-item questionnaire containing both single- and multi-item measures [Aaronson, 1993]. These include five functional scales (Physical, Role, Cognitive, Emotional, and Social Functioning), three symptom scales (Fatigue, Pain, and Nausea/Vomiting), a Global Health Status/QoL scale, and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). The below image shows the details.

Table 1: Scoring the QLQ-C30 version 3.0

| | Scale | Number<br>of items | Item<br>range* | Version 3.0<br>Item numbers | Function scales |
|---|---|---|---|---|---|
| Global health status / QoL | | | | | |
| Global health status/QoL (revised) | QL2 | 2 | 6 | 29, 30 | |
| Functional scales | | | | | |
| Physical functioning (revised) <sup>†</sup> | PF2 | 5 | 3 | 1 to 5 | F |
| Role functioning (revised) <sup>†</sup> | RF2 | 2 | 3 | 6, 7 | F |
| Emotional functioning | EF | 4 | 3 | 21 to 24 | F |
| Cognitive functioning | CF | 2 | 3 | 20, 25 | F |
| Social functioning | SF | 2 | 3 | 26, 27 | F |
| Symptom scales / items | | | | | |
| Fatigue | FA | 3 | 3 | 10, 12, 18 | |
| Nausea and vomiting | NV | 2 | 3 | 14, 15 | |
| Pain | PA | 2 | 3 | 9, 19 | |
| Dyspnoea | DY | 1 | 3 | 8 | |
| Insomnia | SL | 1 | 3 | 11 | |
| Appetite loss | AP | 1 | 3 | 13 | |
| Constipation | CO | 1 | 3 | 16 | |
| Diarrhoea | DI | 1 | 3 | 17 | |
| Financial difficulties | FI | 1 | 3 | 28 | |

<sup>\*</sup> Item range is the difference between the possible maximum and the minimum response to individual items; most items take values from 1 to 4, giving range = 3.

Scores for each scale and single-item measure are averaged and transformed linearly to a score ranging from 0–100. (See below image for details). A high score for functional scales and for Global Health Status/QoL represent better functioning ability or HRQoL, whereas a high score for symptom scales and single items represents significant symptomatology [Proskorovsky, 2014].

<sup>† (</sup>revised) scales are those that have been changed since version 1.0, and their short names are indicated in this manual by a suffix "2" – for example, PF2.

### **Technical Summary**

In practical terms, if items  $I_1$ ,  $I_2$ , ...  $I_n$  are included in a scale, the procedure is as follows:

#### Raw score

Calculate the raw score

$$RawScore = RS = (I_1 + I_2 + ... + I_n)/n$$

### Linear transformation

Apply the linear transformation to 0-100 to obtain the score S,

Functional scales: 
$$S = \left\{1 - \frac{(RS - 1)}{range}\right\} \times 100$$

Symptom scales / items:  $S = \{(RS-1)/range\} \times 100$ Global health status / QoL:  $S = \{(RS-1)/range\} \times 100$ 

Range is the difference between the maximum possible value of RS and the minimum possible value. The QLQ-C30 has been designed so that all items in any scale take the same range of values. Therefore, the range of RS equals the range of the item values. Most items are scored 1 to 4, giving range = 3. The exceptions are the items contributing to the global health status / QoL, which are 7-point questions with range = 6, and the initial yes/no items on the earlier versions of the QLQ-C30 which have range = 1.

### Scoring of the QLQ-C30 Summary Score

The EORTC QLQ-C30 Summary Score is calculated from the mean of 13 of the 15 QLQ-C30 scales (the Global Quality of Life scale and the Financial Impact scale are not included). Prior to calculating the mean, the symptom scales need to be reversed to obtain a uniform direction of all scales. The summary score should only be calculated if all of the required 13 scale scores are available.

QLQ-C30 Summary Score = [Physical Functioning+ Role Functioning+ Social Functioning+ Emotional Functioning+ Cognitive Functioning+ (100- Fatigue)+ (100- Pain)+ (100-Nausea\_Vomiting)+ (100-Dyspnoea)+ (100-Sleeping Disturbances)+ (100-Appetite Loss)+ (100-Constipation)+ (100-Diarrhoea)]/13.

### Handling of missing items

Single-item measures: if the item is missing, the score S will be set to missing.

Scales requiring multiple items: if at least half of the items from the scale are available, the score S will be calculated based on available items. If more than half of the items from the scale are missing, the score S will be set to missing (Fayers, 2001).

Minimal Important Difference (MID): In a sample of patients who received chemotherapy for either breast cancer or small-cell lung cancer (n=246, n=80 respectively), the mean change in EORTC QLQ-C30 score between baseline and follow-

up was about 5 to 10 points on a 0-100 scale for patients who indicated "a little" change on the Subjective Significance Questionnaire (SSQ), either for better or for worse (Osoba, 1998).

### 15.9.2. EORTC QLQ-MY20

The EORTC QLQ-MY20 is a supplement to the QLQ-C30 instrument used in patients with multiple myeloma [Aaronson, 1993; Cocks, 2007]. The module comprises 20 questions that address four myeloma specific HRQoL domains: Disease Symptoms, Side Effects of Treatment, Future Perspective, and Body Image. Three of the four QLQ-MY20 domains are multi-item scales: Disease Symptoms (includes bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity); Side Effects of Treatment (includes drowsiness, thirst, feeling ill, dry mouth, hair loss, upset by hair loss, tingling hands or feet, restlessness/agitation, acid indigestion/heartburn, and burning or sore eyes); and Future Perspective (includes worry about death and health in the future, and thinking about illness). The Body Image scale is a single-item scale that addresses physical attractiveness. (See below image for details).

### Scoring

| | Scale<br>name | Number<br>of items | Item<br>range | QLQ-MY20<br>item numbers |
|---|---|---|---|---|
| Functional scales / items | | | | |
| Future perspective | MYFP | 3 | 3 | 18 - 20 |
| Body image | MYBI | 1 | 3 | 17 |
| Symptom scales | | | | |
| Disease symptoms | MYDS | 6 | 3 | 1 – 6 |
| Side effects of treatment | MYSE | 10 | 3 | 7 – 16 |

#### Remarks

Question 12 is considered scored "not at all" if question 11 is scored "not al all".

As with the QLQ-C30, QLQ-MY20 domain scores are also averaged and transformed linearly to a score ranging from 0–100 (see below for details).

### 1) Raw score

For each multi-item scale, calculate the average of the corresponding items.

$$Raw\ Score = RS = \{(I_1 + I_2 + ... + I_n)/n\}$$

For the single-item measure, the score of the concerning item corresponds to the raw score.

### 2) Linear Transformation

To obtain the Score S, standardize the raw score to a 0 - 100 range following the appropriate transformation:

Symptom scales:  $S = \{(RS-1)/range\} \times 100$ 

Functional scales:  $S = \{1 - (RS - 1)/range\} \times 100$ 

A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes [Proskorovsky, 2014].

Missing items can be handled similarly to EORTC QLQ-C30 as described in Section 15.9.1.

#### 15.9.3. NEI-VFQ-25

The NEI-VFQ-25 consists of a base set of 25 vision-targeted questions representing 11vision-related constructs, plus an additional single-item general health rating question [Mangione, 2001]. The NEIVFQ-25 generates the following 11 vision-targeted subscales: global vision rating, difficulty with near vision activities; difficulty with distance vision activities; limitations in social functioning due to vision; role limitations due to vision; dependency on others due to vision; mental health symptoms due to vision; driving difficulties; limitations with peripheral vision, limitations with color vision; and corneal pain.

The following two tables (from the NEI-VFQ-25 User Manuals) provide the details of converting the original response category to the recoded values, and items of which recoded values need to be averaged to generate the VFQ-25 sub-scales. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Hence scores represent the average for all items in the sub-scale that the respondent answered. Sub-scales with at least one item answered can be used to generate a sub-scale score. To calculate an overall composite score for the VFQ-25, simply average the 11 vision-targeted sub-scale scores.

Table 2. Scoring Key: Recoding of Items

| Item Numbers | Change original response category (a) | To recoded value of: |
|---|---|---|
| 1,3,4,15c(b) | 1 | 100 |
| | | 75 |
| | 2 3 | 50 |
| | 4 | 25 |
| | 5 | 0 |
| 2 | 1 | 100 |
| | 2 | 80 |
| | 3 | 60 |
| | 4 | 40 |
| | 5 | 20 |
| | 6 | 0 |
| 5,6,7,8,9,10,11,12,13,14,16,16a | 1 | 100 |
| A3,A4,A5,A6,A7,A8,A9(c) | 2 | 75 |
| | 2 3 | 50 |
| | 4 | 25 |
| | 5 | 0 |
| | 6 | * |
| 17,18,19,20,21,22,23,24,25, | 1 | 0 |
| A11a,A11b,A12,A13 | 2 | 25 |
| | 3 | 50 |
| | 4 | 75 |
| | 5 | 100 |
| A1,A2 | 0 | 0 |
| | to | to |
| | 10 | 100 |

<sup>(</sup>a) Precoded response choices as printed in the questionnaire.

If 15b=2, then 15c should be recoded to missing.

If 15b=3, then 15c should be recoded to missing.

<sup>(</sup>b) Item 15c has four-response levels, but is expanded to a five-levels using item 15b. Note: If 15b=1, then 15c should be recoded to "0"

<sup>&</sup>quot;A" before the item number indicates that this item is an optional item from the Appendix. If optional items are used, the NEI-VFQ developers encourage users to use all items for a given sub-scale. This will greatly enhance the comparability of sub-scale scores across studies.

<sup>\*</sup> Response choice "6" indicates that the person does not perform the activity because of non-vision related problems. If this choice is selected, the item is coded as "missing."

Table 3. Step 2: Averaging of Items to Generate VFQ-25 Sub-Scales

| Scale | Number of items | Items to be averaged (after recoding per Table 2) |
|---|---|---|
| General Health | 1 | 1 |
| General Vision | 1 | 2 |
| Ocular Pain | 2 | 4, 19 |
| Near Activities | 3 | 5, 6, 7 |
| Distance Activities | 3 | 8, 9, 14 |
| Vision Specific: | | |
| Social Functioning | 2 | 11, 13 |
| Mental Health | 4 | 3, 21, 22, 25 |
| Role Difficulties | 2 | 17, 18 |
| Dependency | 3 | 20, 23, 24 |
| Driving | 3 | 15c, 16, 16a |
| Color Vision | 1 | 12 |
| Peripheral Vision | 1 | 10 |

### 15.10. Appendix 10: COVID-19 Impact

Government or health authority enforced measures to slow the spread of COVID-19 infection (such as lockdowns, social distancing, and travel restrictions) may have impacted recruitment, study treatment administration, study assessment schedule and subject retention.

To understand the impact of the pandemic measures implemented at a country level, alerts set by the GSK country Issue Management Team (IMT) were used to determine when pandemic measures began. The alert levels for a country are based on multiple factors including government or health authority guidance advice, disease spread, and business/public life impact. The alert levels are escalated and de-escalated over time and the scale used for the recording of alerts is standardised: green (low impact), yellow (low to moderate impact), orange (moderate to high impact), red (high impact), and black (high impact with severe disruption). Date of when pandemic measures began was defined based on the IMT alert levels and used in analyses.

### 15.11. Appendix 11: Abbreviations & Trademarks

### 15.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADA | Anti-Drug Antibodies |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| A&R | Analysis and Reporting |
| BM | Bone Marrow |
| BMI | Body mass index |
| BOR | Best Overall Response |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CR | Complete Response |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| ECHO | Echocardiogram |
| eCRF | Electronic Case Record Form |
| eGFR | Estimated glomerular filtration rate |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| FTIH | First Time in Human Trial |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IMWG | International Myeloma Working Group |
| IB | Investigational Brochure |
| IP | Investigational Product |
| irAE | Immune-related Adverse Event |
| iSRC | Internal Safety Review Committee |
| ISS | International Staging System |
| LVEF | Left ventricular ejection fraction |
| MedDRA | Medical Dictionary for Regulatory Affairs |
| MR | Minimal Response |
| CCI | |
| MTD | Maximum Tolerated Dose |
| mTPI | modified Toxicity Probability Interval |

| Abbreviation | Description |
|---|---|
| MUGA | Multigated acquisition scan |
| NE | Not Evaluable |
| NCI | National Cancer Institute |
| NCI-CTCAE | National Cancer Institute Common Toxicity Criteria for Adverse Events |
| ORR | Overall Response Rate |
| PACT | Post analysis continued treatment |
| PD | Progressive Disease |
| PO | Per os (oral) |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RP2D | Recommended Phase 2 Dose |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| sCR | stringent Complete Response |
| SD | Stable Disease |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Classes |
| SOP | Standard Operation Procedure |
| SRM | Study Reference Manual |
| SRT | Safety Review Team |
| TA | Therapeutic Area |
| TLF | Tables, Listings, & Figures |
| VGPR | Very Good Partial Response |

### 15.11.2. Trademarks

| Tra | demarks of the GlaxoSmithKline<br>Group of Companies |
|-----|------------------------------------------------------|
| ADV | ATR |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Chiron RIBA |
| SAS |
| WinNonlin |

### 15.12. Appendix 12: List of Data Displays

### 15.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|----------------------------------|------------------|----------------|
| Study Population | 1.001 to 1.xxx | None |
| Efficacy | 2.001 to 2.xxx | 2.xxx to 2.xxx |
| Safety | 3.001 to 3.xxx | 3.xxx to 3.xxx |
| Pharmacokinetic | 4.001 to 4.xxx | 4.xxx to 4.xxx |
| Pharmacodynamic and/or Biomarker | None | 5.xxx to 5.xxx |
| Patient Reported Outcome | 6.001 to 6.xxx | None |
| Section | Listings | |
| ICH Listings | 1.001 to 1.xxx | |
| Other Listings | 30.001 to 30.xxx | |

### 15.12.2. Deliverables

| Delivery [Priority] [1] | Description |
|---|---|
| IA [1] | Interim Analysis 1 for Arm B cohorts from Protocol Amendment 1 and 2 |
| Post-Interim [1] | Re-run of cohorts from Interim [1] – select displays |
| IA [2] | Interim Analysis 2 for Arm A – all cohorts |
| IA [3] | Interim Analysis 3 for Arm B – all cohorts |
| HDL [1] | Headline Results for Final Analysis (may be completed) |
| SAC [X] | Statistical Analysis Complete for Final Analysis |
| AAC [X] | All Analysis Complete for Final Analysis |
| RAPIDO DV at | Listings that will not be reported within HDL, SAC, nor AAC, but listing |
| <delivery></delivery> | configurations will be created to view within RAPIDO DV. |

### NOTES:

<sup>1.</sup> Indicates priority (i.e., order) in which displays will be generated for the reporting effort

### 15.12.3. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Subject Disposition | | | | |

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.001 | All Treated | ES8 | Summary of Subject Status and Reason for Study Withdrawal (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3, FDAAA, EudraCT Add the following categories under Subject Status – Ongoing: On study treatment, In follow-up – Alive, In follow-up – Unknown. Footnote for "On Study Treatment": Any study treatment component Footnote for "In follow-up - Alive": Subjects that are alive at last contact and within the follow-up period. Footnote for "In follow-up – Unknown": Subjects whose status is unknown at last contact within the contact within the contact within the contact within the contact within the contact may have only one primary reason for withdrawal. Footnote for "Study Terminated By Sponsor": is indicative of subjects continuing into PACT. At SAC, add "Related to COVID-19" as subcategories for applicable study withdrawal categories. | IA [2], HDL<br>[1], SAC [1] |

| S | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| N | lo. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1 | .002 | All Treated | ES8 | Summary of Subject Status and Reason for Study Withdrawal (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA<br>[3], HDL [1],<br>SAC [1] |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 1.003 | All Treated | SD4 | Summary of Treatment Status and Reasons for Discontinuation of GSK2857916 (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 Add footnotes: For "discontinued" under Treatment status: [1] Includes subjects who have discontinued treatment or died prior to End of Treatment Visit. For "Primary reason ": [2] Subjects may have only one primary reason for discontinuation. [3] Subjects who died prior to End of Treatment Visit may not have a reason recorded. Footnote for "'Study Terminated By Sponsor'": 'Study Terminated By Sponsor'" is indicative of subjects continuing into PACT. Add this note starting at SAC for Arm A: "Note: 'Protocol-Specified Withdrawal Criterion Met' indicates discontinuation of study treatment for abnormal liver tests." At SAC, add "Related to COVID-19" as subcategories for applicable study withdrawal categories. | IA [2], SAC<br>[1] |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.004 | All Treated | SD4 | Summary of Treatment Status and Reasons for Discontinuation of GSK2857916 (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above Add this note starting at IA [3] for Arm B: "Note: 'Protocol-Specified Withdrawal Criterion Met' indicates discontinuation of study treatment for abnormal liver tests." | IA [1], IA<br>[3], SAC [1] |
| 1.005 | All Treated | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Lenalidomide (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | IA [2], SAC<br>[1] |
| 1.006 | All Treated | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Bortezomib (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above, except for different wording for footnote related to "Protocol-Specified Withdrawal Criterion Met": 'Protocol-Specified Withdrawal Criterion Met' indicates completion of protocol-specified treatment of Bortezomib | IA [1], IA<br>[3], SAC [1] |
| 1.007 | All Treated | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Dexamethasone (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | IA [2], SAC<br>[1] |
| 1.008 | All Treated | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Dexamethasone (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above, except for different wording for footnote related to "Protocol-Specified Withdrawal Criterion Met": 'Protocol-Specified Withdrawal Criterion Met' indicates completion of protocol-specified treatment of Dexamethasone | IA [1], IA<br>[3], SAC [1] |
| 1.009 | All<br>Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC [1] |
| 1.010 | All Treated | NS1 | Summary of Number of Subjects by Country and Site ID (Arm A – GSK2857916 + Len/Dex (Rd) | EudraCT/Clinical Operations. | SAC [1] |

| Study | Study Population Tables | | | | | |
|---|---|---|---|---|---|--|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | |
| 1.011 | All Treated | NS1 | Summary of Number of Subjects by Country and Site ID (Arm B – GSK2857916 + Bor/Dex (Vd)) | EudraCT/Clinical Operations. | SAC [1] | |
| Protoc | ol Deviation | | | | | |
| 1.012 | All Treated | DV1 | Summary of Important Protocol Deviations (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] | |
| 1.013 | All Treated | DV1 | Summary of Important Protocol Deviations (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | IA [3], SAC<br>[1] | |
| 1.014 | All Treated | IE1 | Summary of Inclusion/Exclusion Criteria Deviations (Arm A – GSK2857916 + Len/Dex (Rd)) | | SAC [1] | |
| 1.015 | All Treated | IE1 | Summary of Inclusion/Exclusion Criteria Deviations (Arm B – GSK2857916 + Bor/Dex (Vd)) | | SAC [1] | |
| 1.016 | All Treated | PAN4 | Summary of Visits impacted by COVID-19 Pandemic (Arm A – GSK2857916 + Len/Dex (Rd)) | | SAC [1] | |
| 1.017 | All Treated | PAN4 | Summary of Visits impacted by COVID-19 Pandemic (Arm B – GSK2857916 + Bor/Dex (Vd)) | | SAC [1] | |
| Demog | graphic and B | aseline Cha | racteristics | | | |
| 1.018 | All Treated | DM1 | Summary of Demographic Characteristics (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3, FDAAA, EudraCT | IA [2], SAC<br>[1] | |
| 1.019 | All Treated | DM1 | Summary of Demographic Characteristics (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3, FDAAA, EudraCT | IA [1], IA<br>[3], SAC [1] | |
| 1.020 | All Treated | DM11 | Summary of Age Ranges (Arm A – GSK2857916 + Len/Dex (Rd)) | EudraCT | SAC [1] | |
| 1.021 | All Treated | DM11 | Summary of Age Ranges (Arm B – GSK2857916 + Bor/Dex (Vd)) | EudraCT | SAC [1] | |
| 1.022 | All Treated | DM5 | Summary of Race and Racial Combinations (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3, FDA, FDAAA, EudraCT | SAC [1] | |
| Study | Study Population Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | |
| 1.023 | All Treated | DM5 | Summary of Race and Racial Combinations (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3, FDA, FDAAA, EudraCT | SAC [1] | | | |
| Diseas | Disease Characteristics | | | | | | | |

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.024 | All Treated | DC2 | Summary of Disease Characteristics at Screening (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 if collected Summarize Stage, Relapsed or refractory disease, Does the subject have Extramedullary Disease, Myeloma immunoglobulin, Does the subject have light chain myeloma, Type of multiple myeloma, Lines of therapy completed prior to screening, Lytic Bone Lesions, ECOG performance status. Include genetic characteristics, if collected For Lines of therapy completed prior to screening, display using summary statistics (n, mean, standard deviation, median, min, max). For ECOG performance status, include groups as 0, 1, 2 Add a "missing" category to Genetics for any subject missing genetics information at screening For High Risk Cytogenetics, use the following groups: High-Risk (positive), Other (non-high risk, negative, not evaluable, not done). | IA [2], HDL<br>[1], SAC [1] |

| Study | Population Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.025 | All Treated | DC2 | Summary of Disease Characteristics at Screening (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA<br>[3], HDL [1],<br>SAC [1] |
| Prior a | nd Concomita | ant Medicat | ons | | • |
| 1.026 | All Treated | MH1 | Summary of Current Medical Conditions (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 1.027 | All Treated | MH1 | Summary of Current Medical Conditions (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| 1.028 | All Treated | MH1 | Summary of Past Medical Conditions (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 1.029 | All Treated | MH1 | Summary of Past Medical Conditions (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| 1.030 | All Treated | CM8 | Summary of Concomitant Medications (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 include 'medications taken on-<br>treatment (including those started prior to<br>treatment), and "Medications that started on<br>treatment' Column 1 by "Ingredient-Route" | SAC [1] |
| 1.031 | All Treated | CM8 | Summary of Concomitant Medications (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | SAC [1] |
| Prior A | Anti-Cancer Th | nerapy | | | |
| 1.032 | All Treated | AC2 | Summary of Prior Anti-Cancer Therapy by Drug Class of Agents (Arm A – GSK2857916 + Len/Dex (Rd)) | See Table 1.0200 in Study 205678 (primary_01). Add footnote: Note: Subjects may be included in more than one category. | IA [2], SAC<br>[1] |
| 1.033 | All Treated | AC2 | Summary of Prior Anti-Cancer Therapy by Drug Class of Agents (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA<br>[3], SAC [1] |

## CONFIDENTIAL

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expos | Exposure and Treatment Compliance | | | | |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 1.034 | All Treated | OEX1 | Summary of Exposure to GSK2857916 (Arm A – GSK2857916 + Len/Dex (Rd)) | *Include "Time on Study Treatment (weeks)"; "Dose Intensity (mg/kg/4 weeks)"; n, Mean, SD, Median, Min, Max; Relative Dose Intensity (%). *See definition of Dose Intensity in Section 6.5 *Label Dose Intensity as (mg/kg/interval), with a footnote for interval to state "interval is 4 weeks for SINGLE and SPLIT dosing and 8 weeks for STRETCH dosing." Footnotes: [1] The time on study treatment does not exclude dose interruptions. [2] Interval is 4 weeks for SINGLE and SPLIT dosing, and 8 weeks for STRETCH and S/D STRETCH dosing. [3] dose intensity, date of discontinuation is the date of last dose. [4] Relative dose intensity (Dose 1) is calculated as a percent and is defined as 100*(mean overall Dose Intensity for Dose 1 divided by planned dose intensity (post-Dose 1) is calculated as a percent and is defined as 100*(mean overall Dose Intensity post Dose 1 divided by planned dose intensity post Dose 1 divided by planned dose intensity post Dose 1 divided by planned dose intensity post Dose 1). | IA [2], SAC<br>[1] |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| | | | | *Include "Time on Study Treatment (weeks)"; "Dose Intensity (mg/kg/4 weeks)"; n, Mean, SD, Median, Min, Max; Relative Dose Intensity (%) | |
| | | | | *For S/D Stretch dose, DI and RDI calculations for post-C1D1 only. | |
| | | | | *See definition of Dose Intensity in Section 6.5 | |
| | | | | *Label Dose Intensity as (mg/kg/interval),<br>with a footnote for interval to state "interval is<br>3 weeks for SINGLE and SPLIT doses and 6<br>weeks for STRETCH and S/D STRECH<br>doses." | |
| 1.035 | All Treated | OEX1 | Summary of Exposure to GSK2857916 (Arm B – GSK2857916 + Bor/Dex (Vd)) | Footnotes: [1] The time on study treatment does not exclude dose interruptions. [2] Interval is 3 weeks for SINGLE and SPLIT dosing, and 6 weeks for STRETCH and S/D STRETCH dosing. [3] For dose intensity, date of discontinuation is the date of last dose. [4] Relative dose intensity (Dose 1) is calculated as a percent and is defined as 100*(mean overall Dose Intensity for Dose 1 divided by planned dose intensity for Dose | IA [1], Post-<br>Interim [1],<br>IA [3], SAC<br>[1] |
| | | | 113 | 1). [5] Relative dose intensity (post-Dose 1) is calculated as a percent and is defined as 100*(mean overall Dose Intensity post Dose 1 divided by planned dose intensity post Dose 1). Note: ID 801 (GSK916 2.5mg/kg SPLIT + Vd cohort) was dosed with 2.5 mg/kg of GSK2857916 on Day 1 and 8. | |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 1.036 | All Treated | OEX1 | Summary of Exposure to Lenalidomide (Arm A – GSK2857916 + Len/Dex (Rd)) | Within the table, separate out the calculation to create dose intensity for subjects who's first dose was 25mg, vs. those whose first dose was 10mg. Therefore, we will have 2 DI calculations (first dose 25mg and first dose 10mg). We will still have 1 Relative DI calculation At SAC add: Time on Study Treatment (weeks) [1] Dose Intensity (mg/4 weeks) – 10mg [2] Dose Intensity (mg/4 weeks) – 25mg [2] Relative Dose Intensity [3] Footnotes: [1] The time on study treatment does not exclude dose interruptions. [2] For dose intensity, date of discontinuation is the date of last dose. [3] Relative dose intensity is calculated as a percent and is defined as 100*(mean overall Dose Intensity divided by planned dose intensity). Note: Lenalidomide is administered as 25mg/day in subjects with eGFR >=60 mL/min/1.73 m^2. The dose of lenalidomide is reduced to 10mg/day in subjects with eGFR of 40-60 mL/min/1.73 m^2. | IA [2], SAC<br>[1] |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.037 | All Treated | OEX1 | Summary of Exposure to Bortezomib (Arm B – GSK2857916 + Bor/Dex (Vd)) | Add: Time on Study Treatment (weeks) [1] Dose Intensity (mg/m2/3 weeks) [2] Relative Dose Intensity [3] Footnotes: [1] The time on study treatment does not exclude dose interruptions. [2] For dose intensity, date of discontinuation is the date of last dose. [3] Relative dose intensity is calculated as a percent and is defined as 100*(mean overall Dose Intensity divided by planned dose intensity). | IA [1], IA<br>[3], SAC [1] |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | <u> </u> | | Within the table, separate out the calculation to create dose intensity for subjects who's first dose was 20mg, vs. those whose first dose was 40mg. Therefore, we will have 2 DI calculations (first dose 20mg and first dose 40mg). We will still have 1 Relative DI calculation Add: Time on Study Treatment (weeks) [1] Dose Intensity (mg/4 weeks) – 20mg [2] | |
| 1.038 | All Treated | OEX1 | Summary of Exposure to Dexamethasone (Arm A – GSK2857916 + Len/Dex (Rd)) | Dose Intensity (mg/4 weeks)— 40mg [2] Relative Dose Intensity [3] Footnotes: [1] The time on study treatment does not | SAC [1] |
| | exclude dose interruptions. [2] For dose intensity, date of disconting is the date of last dose. [3] Relative dose intensity is calculate | [2] For dose intensity, date of discontinuation | | | |
| | | | | 100*(mean overall Dose Intensity divided by planned dose intensity). | |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| | | | | Within the table, separate out the calculation to create dose intensity for subjects who's first dose was 10mg, vs. those whose first dose was 20mg. Therefore, we will have 2 DI calculations (first dose 20mg and first dose 40mg). We will still have 1 Relative DI calculation | |
| 1.039 | All Treated | OEX1 | Summary of Exposure to Dexamethasone (Arm B – GSK2857916 + Bor/Dex | Time on Study Treatment (weeks) [1] Dose Intensity (mg/3 weeks) – 10mg [2] Dose Intensity (mg/3 weeks) – 20mg [2] | SAC [1] |
| 1.000 | All Treated | Footnotes: [1] The time on study treatment does not exclude dose interruptions. [2] For dose intensity, date of discontinual is the date of last dose. [3] Relative dose intensity is calculated a percent and is defined as | (Vd)) | [1] The time on study treatment does not | ONO [1] |
| | | | [2] For dose intensity, date of discontinuation is the date of last dose. | | |
| | | | | percent and is defined as | |
| | | | | 100*(mean overall Dose Intensity divided by planned dose intensity). | |

| Study | Population Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.040 | All Treated | ODMOD1 | Summary of Dose Reductions of GSK2857916 (Arm A – GSK2857916 + Len/Dex (Rd)) | *Replace "Planned Time" with "Visit" for "Number of Subjects with Dose Reduction by Planned Time." *Add footnotes: For Arm A, each cycle is 4 weeks (28 days) No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE | IA [2], SAC<br>[1] |
| 1.041 | All Treated | ODMOD1 | Summary of Dose Reductions of GSK2857916 (Arm B – GSK2857916 + Bor/Dex (Vd)) | *Replace "Planned Time" with "Visit" for "Number of Subjects with Dose Reduction by Planned Time." *Add footnotes: For Arm B, each cycle is 3 weeks (21 days) No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE, and 2.5 mg/kg S/D STRETCH | IA [1], IA<br>[3], SAC [1] |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.042 | All Treated | ODMOD3 | Summary of Dose Delays of GSK2857916 (Arm A – GSK2857916 + Len/Dex (Rd)) | *Replace "Planned Time" with "Visit" for "Number of Subjects with Dose Delays by Planned Time." Under "Delay Duration (days)" use the following groups: 1-28, 29-56, >56 *Add a footnote: "For Arm A, each cycle is 4 weeks (28 days)" *Add the following note in the footnotes: Note: From the Exposure eCRF, dose delays are defined when a dose modification has been indicated as "Delay". For the "Adverse Event" category under "Primary Reason", these events correspond to the GSK2857916 Exposure eCRF where primary reason has been recorded as Adverse Event. | IA [2], SAC<br>[1] |

| Study | Population Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.043 | All Treated | ODMOD3 | Summary of Dose Delays of GSK2857916 (Arm B – GSK2857916 + Bor/Dex (Vd)) | *Replace "Planned Time" with "Visit" for "Number of Subjects with Dose Delays by Planned Time." Under "Delay Duration (days)" use the following groups: 1-21, 22-42, >42 *Add a footnote: "For Arm B, each cycle is 3 weeks (21 days)" *Add the following note in the footnotes: Note: From the Exposure eCRF, dose delays are defined when a dose modification has been indicated as "Delay". For the "Adverse Event" category under "Primary Reason", these events correspond to the GSK2857916 Exposure eCRF where primary reason has been recorded as Adverse Event. | IA [1], IA<br>[3], SAC [1] |
| 1.044 | All Treated | ODMOD5 | Summary of Primary Reason for Dose Reductions of GSK2857916 by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | *Changed "planned time" columns to "visit" *Add footnotes: For Arm A, each cycle is 4 weeks (28 days) No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE | IA [2], SAC<br>[1] |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.045 | All Treated | OEX6 | Summary of Dose Intensity of GSK2857916 by Expected Duration of Exposure (Arm A – GSK2857916 + Len/Dex (Rd)) | *This display was created for IA [1] and Post Interim [1] only. After Post-Interim [1], this display was removed, hence the renumbering of displays. This is a summary of dose intensity by a patient's actual or expected duration of exposure for Arm A (Q4W). *Add footnotes: [1] Dose intensity is the cumulative actual dose divided by duration of exposure (or expected duration of exposure) in mg/kg/4weeks. Note: For Arm A, expected duration of exposure is every 4 weeks (28 days). | IA [1], Post<br>Interim [1] |
| 1.045 | All Treated | ODMOD5 | Summary of Primary Reason for Dose Reductions of GSK2857916 by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | *Changed "planned time" columns to "visit" *Add footnotes: For Arm B, each cycle is 3 weeks (21 days) No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE, and 2.5 mg/kg S/D STRETCH | IA [1], IA<br>[3], SAC [1] |

| IDSL / | | Study Population Tables | |
|---|---|---|---|
| n Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ODMOD6 | Summary of Primary Reason for Dose Delays of GSK2857916 by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | *Changed "planned time" columns to "visit" *Add a footnote: "For Arm A, each cycle is 4 weeks (28 days)" *Add the following note in the footnotes: Note: From the Exposure eCRF, dose delays are defined when a dose modification has been indicated as "Delay". For the "Adverse Event" category under "Primary Reason", these events correspond to the GSK2857916 Exposure eCRF where primary reason has been recorded as Adverse Event. | IA [2], SAC<br>[1] |
| ODMOD6 | Summary of Primary Reason for Dose Delays of GSK2857916 by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above, except for the following footnote: *Add a footnote: "For Arm B, each cycle is 3 weeks (21 days)" | IA [1], IA<br>[3], SAC [1] |
| | ODMOD6 | ODMOD6 Summary of Primary Reason for Dose Delays of GSK2857916 by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) ODMOD6 Summary of Primary Reason for Dose Delays of GSK2857916 by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | ODMOD6 Summary of Primary Reason for Dose Delays of GSK2857916 by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) ODMOD6 Summary of Primary Reason for Dose Delays of GSK2857916 by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) ODMOD6 Summary of Primary Reason for Dose Delays of GSK2857916 by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) Summary of Primary Reason for Dose Delays of GSK2857916 by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) *Changed "planned time" columns to "visit" *Add a footnote: "For Arm A, each cycle is 4 weeks (28 days)" *Add a footnote: "For Arm B, each cycle is 3 weeks (21 days)" |

| Study | Population Ta | ables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.048 | All Treated | FAC2 | Summary of Duration of Follow-Up (Arm A – GSK2857916 + Len/Dex (Rd)) | Add a Total column at SAC [1] Footnotes: [1] Duration of Follow-Up is defined as the time from first dose to last contact or death. [2] Subjects with ongoing Follow-Up are those within the column Follow-Up period, with status Alive or Unknown For SAC, do not report subjects with ongoing follow-up, as participants are moving into PACT. | IA [2], SAC<br>[1] |
| 1.049 | All Treated | FAC2 | Summary of Duration of Follow-Up (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above Add a Total column at IA [3] and SAC [1] | IA [3], SAC<br>[1] |
| Blood | and Blood Su | pportive Ca | are Products | | 1 |
| 1.050 | All Treated | BP1A | Summary of Blood Products (Arm A – GSK2857916 + Len/Dex (Rd)) | | SAC [1] |
| 1.051 | All Treated | BP1A | Summary of Blood Products (Arm B – GSK2857916 + Bor/Dex (Vd)) | | SAC [1] |
| 1.052 | All Treated | BP1C | Summary of Blood Supportive Care Products (Arm A – GSK2857916 + Len/Dex (Rd)) | | SAC [1] |
| 1.053 | All Treated | BP1C | Summary of Blood Supportive Care Products (Arm B – GSK2857916 + Bor/Dex (Vd)) | | SAC [1] |
| Substa | ance Use | | | | |
| 1.054 | All Treated | SU1 | Summary of Substance Use (Arm A – GSK2857916 + Len/Dex (Rd)) | | SAC [1] |
| 1.055 | All Treated | SU1 | Summary of Substance Use (Arm B – GSK2857916 + Bor/Dex (Vd)) | | SAC [1] |

## 15.12.4. Efficacy Tables

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Respons | ses | | | | |
| 2.001 | All Treated | RE1a | Summary of Investigator-Assessed Best Response with confirmation (IMWG criteria) (Arm A – GSK2857916 + Len/Dex (Rd)) | Best Response: Stringent Complete Response (sCR), Complete response (CR), Very Good Partial Response (VGPR), Partial Response (PR), Minimal Response (MR), Stable Disease (SD), Progressive Disease (PD), Not Evaluable (NE). *Display each of the summaries below in this order: CCI (sCR+CR+VGPR+PR+MR) Overall Response Rate: (sCR+CR+VGPR+PR) CCI (sCR+CR+VGPR+PR) CCI (sCR+CR) Footnote: The 95% Confidence Interval is based on Exact method. | IA [2], HDL [1],<br>SAC [1] |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.002 | All Treated | RE1a | Summary of Investigator-Assessed Best Response with confirmation (IMWG criteria) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | Post-Interim [1],<br>IA [1], IA [3],<br>HDL [1], SAC<br>[1] |
| Time-to- | Event | | | | |
| 2.003 | All Treated | TTE1a | Summary of CCI Based on Investigator-Assessed Response (Arm A – GSK2857916 + Len/Dex (Rd)) | Among responders only Add footnote: | SAC [1] |
| 2.004 | All Treated | TTE1a | Summary of CCI Based on Investigator-Assessed Response (Arm B – GSK2857916 + Bor/Dex (Vd)) | | IA [3], SAC [1] |
| | | | Summary of CCI Based on Investigator- | Among responders only Add footnote: | |
| 2.005 | All Treated | TTE1a | Assessed Response (Arm A – GSK2857916 + Len/Dex (Rd)) | CCI | SAC [1] |
| 2.006 | All Treated | TTE1a | Summary of CCI Based on Investigator-Assessed Response (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | SAC [1] |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.007 | All Treated | TTE1a | Summary of | Among responders only Add footnote: is documented per IMWG; or death due to PD occurs among participants who achieve an overall response, i.e., confirmed PR or better. Include the estimated probability at Month 4 at interim and Month 6, 9, 12, and 18 at final analysis. | IA [2], HDL [1],<br>SAC [1] |
| 2.008 | All Treated | TTE1a | Summary of CCI Based on Investigator-Assessed Response (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [3], HDL [1],<br>SAC [1] |
| 2.009 | All Treated | TTE1a | Summary of CCI Based on Investigator-Assessed Response (Arm A – GSK2857916 + Len/Dex (Rd)) | Include the estimated probability at Month 4 at interim and Month 6, 9, 12, and 18 at final analysis. Footnotes: [1] Confidence Intervals estimated using the Brookmeyer Crowley method. Note column is defined as the time from first dose until the earliest date of confirmed disease progression (PD) per IMWG, or death due to any cause. | IA [2], HDL [1],<br>SAC [1] |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.010 | All Treated | TTE1a | Summary of CCI Based on Investigator-Assessed Response (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [3], HDL [1],<br>SAC [1] |
| 2.011 | All Treated | TTE1a | Summary of CCI Based on Investigator-Assessed Response (Arm A – GSK2857916 + Len/Dex (Rd)) | Footnotes: [1] Confidence Intervals estimated using the Brookmeyer Crowley method. Note: CO per IMWG, or death due to PD. | SAC [1] |
| 2.012 | All Treated | TTE1a | Summary of CCI Based on Investigator-Assessed Response (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | SAC [1] |
| 2.013 | All Treated | TTE1a | Summary of CCI (Arm A – GSK2857916 + Len/Dex (Rd)) | Include the estimated probability at Month 4 at interim and Month 6, 9, 12, and 18 at final analysis. Footnotes: [1] Confidence Intervals estimated using the Brookmeyer Crowley method. Note: pc: | IA [2], SAC [1] |
| 2.014 | All Treated | TTE1a | Summary of CQ (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [3], SAC [1] |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| | | | | See Table 2.4 in Study 207503 (internal_02). | |
| | | | | For each dose group (Inv-Assessed only): | |
| | | | | Coll and 95% Confidence Interval for sCR/CR and sCR/CR/VGPR groups. | |
| | | | | Add small n for "Data Available" to reflect number of subjects with any data. | |

## 15.12.5. Efficacy Figures

| Efficacy: Fi | gures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Response | | | | | |
| 2.017 | All Treated | Programming<br>note | Forest Plot - Overall Response Rate (ORR) Based on Investigator-Assessed-Assessed Response (Arm A – GSK2857916 + Len/Dex (Rd)) | Similar to Figure 2.0020 in Study 205678 (primary_01). See Section 5.3.1 for the subgroups to be included. Create one Forest Plot for all doses combined, and then a second Forest Plot for the 2.5 mg/kg SINGLE dose only. | SAC [1] |
| 2.018 | All Treated | Programming note | Forest Plot - Overall Response Rate (ORR) Based on Investigator-Assessed Response (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | SAC [1] |
| Time-to-Ev | ent | | | | |
| 2.019 | All Treated | TTE10 | Graph of Kaplan Meier Curves of CCI<br>Based on Investigator-Assessed Response (Arm A –<br>GSK2857916 + Len/Dex (Rd)) | Labels: X-axis: Time since CCI (Months) Y-axis: Proportion Alive and | SAC [1] |
| 2.020 | All Treated | TTE10 | Graph of Kaplan Meier Curves of CCI<br>Based on Investigator-Assessed Response (Arm B –<br>GSK2857916 + Bor/Dex (Vd)) | Labels: X-axis: Time since CCI (Months) Y-axis: Proportion Alive and | SAC [1] |

| Efficacy: Fi | gures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.021 | All Treated | TTE10 | Graph of Kaplan Meier Curves of COL<br>Based on Investigator-Assessed Response (Arm A –<br>GSK2857916 + Len/Dex (Rd)) | Labels: X-axis: Time since Treatment Start Date (Months) Y-axis: Proportion Alive and | SAC [1] |
| 2.022 | All Treated | TTE10 | Graph of Kaplan Meier Curves of CCI Based on Investigator-Assessed Response (Arm B – GSK2857916 + Bor/Dex (Vd)) | Labels: X-axis: Time since Treatment Start Date (Months) Y-axis: Proportion Alive and | SAC [1] |
| 2.023 | All Treated | TTE10 | Graph of Kaplan Meier Curves of Colonia Based on Investigator-Assessed Response (Arm A – GSK2857916 + Len/Dex (Rd)) | Labels: X-axis: Time since Treatment Start Date (Months) Y-axis: Proportion Alive and | SAC [1] |
| 2.024 | All Treated | TTE10 | Graph of Kaplan Meier Curves of Colonia Based on Investigator-Assessed Response (Arm B – GSK2857916 + Bor/Dex (Vd)) | Labels: X-axis: Time since Treatment Start Date (Months) Y-axis: Proportion Alive and | SAC [1] |
| 2.025 | All Treated | TTE10 | Graph of Kaplan Meier Curves of CCI Arm A – GSK2857916 + Len/Dex (Rd)) | Labels: X-axis: Time since Treatment Start Date (Months) Y-axis: | SAC [1] |

| Efficacy: Fig | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.026 | All Treated | TTE10 | Graph of Kaplan Meier Curves of CCI (Arm B – GSK2857916 + Bor/Dex (Vd)) | Labels: X-axis: Time since Treatment Start Date (Months) Y-axis: | SAC [1] |

## 15.12.6. Safety Tables

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| Adverse I | Events (AEs) | | | | |
| | | | | See mock in Section 15.13 with categories and footnotes to include. In shell, for rows that state "Lenalidomide/Bortezomib" – use "Lenalidomide" for Arm A. | |
| 3.001 | All Treated | AE13 | Adverse Event Overview (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], HDL [1], SAC [1] |
| | | | | Add footnote: No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE | |
| | | | | See mock in Section 15.13 with categories and footnotes to include. In shell, for rows that state "Lenalidomide/Bortezomib" – use "Bortezomib" for Arm B. | |
| 3.002 | All Treated | AE13 | Adverse Event Overview (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [1], IA [3], HDL<br>[1],SAC [1] |
| | | | | Add footnote: No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE, and 2.5 mg/kg S/D STRETCH | |
| 3.003 | All Treated | OAE07 | Summary of Adverse Events by Preferred Term and Maximum Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 Add summary over all cohorts | IA [2], HDL [1], SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.004 | All Treated | OAE07 | Summary of Adverse Events by Preferred Term and Maximum Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 Add summary over all cohorts | IA [1], IA [3], HDL [1],<br>SAC [1] |
| 3.005 | All Treated | OAE07 | Summary of Adverse Events Related to GSK2857916 by Preferred Term and Maximum Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | Add footnote: 'Related to GSK2857916 includes responses of 'Yes' only, to the following question: 'Is there a reasonable possibility that the AE may have been caused by the study treatment?' for GSK2857916 Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [2], SAC [1] |
| 3.006 | All Treated | OAE07 | Summary of Adverse Events Related to GSK2857916 by Preferred Term and Maximum Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |
| 3.007 | All Treated | OAE07 | Summary of Adverse Events Related to Lenalidomide by Preferred Term and Maximum Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | 'Related to Lenalidomide includes responses of 'Yes' only, to the following question: 'Is there a reasonable possibility that the AE may have been caused by the study treatment?' for Lenalidomide Use definition of treatment emergent AEs as seen in Section 15.2.3 | SAC [1] |
| 3.008 | All Treated | OAE07 | Summary of Adverse Events Related to Bortezomib by Preferred Term and Maximum Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | 'Related to Bortezomib includes responses of 'Yes' only, to the following question: 'Is there a reasonable possibility that the AE may have been caused by the study treatment?' for Bortezomib Use definition of treatment emergent AEs as seen in Section 15.2.3 | SAC [1] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.009 | All Treated | OAE07 | Summary of Adverse Events Related to Dexamethasone by Preferred Term and Maximum Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | 'Related to Dexamethasone includes responses of 'Yes' only, to the following question: 'Is there a reasonable possibility that the AE may have been caused by the study treatment?' for Dexamethasone Use definition of treatment emergent AEs as | SAC [1] |
| | | | Company of Advance Frants Deleted to | seen in Section 15.2.3 | |
| 3.010 | All Treated | OAE07 | Summary of Adverse Events Related to Dexamethasone by Preferred Term and Maximum Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | SAC [1] |
| 3.011 | All Treated | OAE07 | Summary of Adverse Events Related to Study<br>Treatment by Preferred Term and Maximum Grade<br>(Arm A – GSK2857916 + Len/Dex (Rd)) | 'Related to Study Treatment' includes responses of 'Yes' and missing responses to the following question: 'Is there a reasonable possibility that the AE may have been caused by the study treatment?' Use definition of treatment emergent AEs as seen in Section 15.2.3 Include a footnote: AEs related to at least one component of study treatment are included. | IA [2], SAC [1] |
| 3.012 | All Treated | OAE07 | Summary of Adverse Events Related to Study<br>Treatment by Preferred Term and Maximum Grade<br>(Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |
| 3.013 | All Treated | AE3 | Summary of Adverse Events of Maximum Grade 3 or Higher by Preferred Term (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [2], SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.014 | All Treated | AE3 | Summary of Adverse Events of Maximum Grade 3 or Higher by Preferred Term (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [1], IA [3],<br>SAC [1] |
| 3.015 | All Treated | AE1 | Summary of All Adverse Events by System Organ<br>Class and Preferred Term (Arm A – GSK2857916 +<br>Len/Dex (Rd)) | ICH E3 Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], SAC [1] |
| 3.016 | All Treated | AE1 | Summary of All Adverse Events by System Organ<br>Class and Preferred Term (Arm B – GSK2857916 +<br>Bor/Dex (Vd)) | ICH E3 Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [1], IA [3],<br>SAC [1] |
| 3.017 | All Treated | AE3 | Summary of Common (>=5%) Adverse Events by Preferred Term (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.018 | All Treated | AE3 | Summary of Common (>=5%) Adverse Events by Preferred Term (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.019 | All Treated | AE15 | Summary of Common (>=5%) Non-serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) (Arm A –<br>GSK2857916 + Len/Dex (Rd)) | FDAAA, EudraCT Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.020 | All Treated | AE15 | Summary of Common (>=5%) Non-serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) (Arm B –<br>GSK2857916 + Bor/Dex (Vd)) | FDAAA, EudraCT Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.021 | All Treated | AE3 | Summary of Common (>=5%) Grade 3+ Adverse<br>Events by Preferred Term (Arm A – GSK2857916 +<br>Len/Dex (Rd)) | ICH E3 Use definition of on-treatment AEs as seen in Section15.2.3 | SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.022 | All Treated | AE3 | Summary of Common (>=5%) Grade 3+ Adverse<br>Events by Preferred Term (Arm B – GSK2857916 +<br>Bor/Dex (Vd)) | ICH E3 Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.023 | All Treated | AE3 | Summary of Common (>=5%) Drug-Related Grade 3+Adverse Events by Preferred Term (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 *Drug-Related = GSK2857916, Len, and/or Dex Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.024 | All Treated | AE3 | Summary of Common (>=5%) Drug-Related Grade 3+<br>Adverse Events by Preferred Term (Arm B –<br>GSK2857916 + Bor/Dex (Vd)) | ICH E3 *Drug-Related = GSK2857916, BOR, and/or Dex Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.025 | All Treated | PAN1A | Number of subjects with suspected, probable or confirmed for COVID-19 infection (Arm A – GSK2857916 + Len/Dex (Rd)) | | SAC [1] |
| 3.026 | All Treated | PAN1A | Number of subjects with suspected, probable, or confirmed for COVID-19 infection (Arm B – GSK2857916 + Bor/Dex (Vd)) | | SAC [1] |
| Serious a | nd Other Signi | ficant Adverse Eve | ents | | |
| 3.027 | All Treated | AE3 | Summary of Serious Adverse Events (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of on-treatment AEs as seen in Section 15.2.3. Sort in descending order of total incidence. | IA [2], SAC [1] |
| 3.028 | All Treated | AE3 | Summary of Serious Adverse Events (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of on-treatment AEs as seen in Section 15.2.3. Sort in descending order of total incidence. | IA [1], IA [3],<br>SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.029 | All Treated | OAE07 | Summary of Serious Adverse Events Related to GSK2857916 by Preferred Term and Maximum Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | Add footnote: 'Related to GSK2857916 includes responses of 'Yes' only, to the following question: 'Is there a reasonable possibility that the SAE may have been caused by the study treatment?' for GSK2857916 Use definition of treatment emergent AEs as seen in Section 15.2.3 Add summary over all cohorts | IA [2], SAC [1] |
| 3.030 | All Treated | OAE07 | Summary of Serious Adverse Events Related to GSK2857916 by Preferred Term and Maximum Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [3], SAC [1] |
| 3.031 | All Treated | AE3 | Summary of AEs Leading to Permanent Discontinuation of Study Treatment by Preferred Term (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], SAC [1] |
| 3.032 | All Treated | AE3 | Summary of AEs Leading to Permanent Discontinuation of Study Treatment by Preferred Term (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [1], IA [3],<br>SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.033 | All Treated | AE3 | Summary of Adverse Events Leading to Dose<br>Reductions/Interruptions/Delays (Arm A –<br>GSK2857916 + Len/Dex (Rd)) | *Add the following notes in the footnotes: Note: This summary includes responses of "Dose reduced", "Dose interrupted/delayed", and "Infusion stopped early and not completed", to the following question: "Were any action(s) taken with GSK2857916 (also Lenalidomide and Dexamethasone) as a result of the AE?" from the AE eCRF. No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], SAC [1] |
| 3.034 | All Treated | AE3 | Summary of Adverse Events Leading to Dose<br>Reductions/Interruptions/Delays (Arm B –<br>GSK2857916 + Bor/Dex (Vd)) | *Add the following notes in the footnotes: Note: This summary includes responses of "Dose reduced", "Dose interrupted/delayed", and "Infusion stopped early and not completed", to the following question: "Were any action(s) taken with GSK2857916 (also Bortezomib and Dexamethasone) as a result of the AE?" from the AE eCRF. No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE, and 2.5 mg/kg S/D STRETCH Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [1], IA [3],<br>SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| Adverse E | Events of Spec | ial Interest | | | |
| 3.035 | All Treated | ESI1 | Summary of Characteristics of Corneal Events<br>(Overall GSK scale) (Arm A – GSK2857916 + Len/Dex<br>(Rd)) | See mock in Section 15.13 with categories and footnotes to include. | IA [2], HDL [1], SAC [1] |
| | | | | Same as above | |
| 3.036 | All Treated | ESI1 | Summary of Characteristics of Corneal Events<br>(Overall GSK scale) (Arm B – GSK2857916 + Bor/Dex<br>(Vd)) | Also, add a footnote: For IDs 2, 3, 6 (Arm B 2.5 mg/kg SINGLE), total number of adverse events may be overreported due to a site related unfixable non-standard logging of ongoing events. | IA [1], Post-Interim [1],<br>IA [3], HDL [1],<br>SAC [1] |
| 3.037 | All Treated | AE13_GSK | Corneal Event Overview (Overall GSK Scale) (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock in Section 15.13 with categories and footnotes to include Add footnote: No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE | IA [2], SAC [1] |
| 3.038 | All Treated | AE13_GSK | Corneal Event Overview (Overall GSK Scale) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], Post-Interim [1],<br>IA [3],<br>SAC [1] |
| 3.039 | All Treated | ESI2b | Summary of Onset and Duration of the First<br>Occurrence of Corneal Events (Overall GSK Scale) of<br>Grade 2 or Above (Arm A – GSK2857916 + Len/Dex<br>(Rd)) | Time of onset: 1-28, 29-56, 57-84, >84.<br>Duration: 1-28, 29-56, >56. Mean, SD,<br>Median, Min, Max | IA [2], SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.040 | All Treated | ESI2b | Summary of Onset and Duration of the First<br>Occurrence of Corneal Events (Overall GSK Scale) of<br>Grade 2 or Above (Arm B – GSK2857916 + Bor/Dex<br>(Vd)) | Same as above, except for Time of Onset and Duration groups: Time of onset: 1-21, 22-42, 43-63, >63. Duration: 1-21, 22-42, >42. Mean, SD, Median, Min, Max | IA [1], Post-Interim [1],<br>IA [3],<br>SAC [1] |
| 3.041 | All Treated | SAFE_T2a | Summary of Corneal Events (Overall GSK Scale)<br>Leading to Action Taken with GSK2857916 (Arm A –<br>GSK2857916 + Len/Dex (Rd)) | | IA [2], SAC [1] |
| 3.042 | All Treated | SAFE_T2a | Summary of Corneal Events (Overall GSK Scale)<br>Leading to Action Taken with GSK2857916 (Arm B –<br>GSK2857916 + Bor/Dex (Vd)) | | IA [1], IA [3],<br>SAC [1] |
| 3.043 | All Treated | Programming<br>Note | Summary of Worst Post-Baseline Corneal Events (GSK Scale) (Arm A – GSK2857916 + Len/Dex (Rd)) | See Section 15.13 for mock | IA [2], SAC [1] |
| 3.044 | All Treated | Programming<br>Note | Summary of Worst Post-Baseline Corneal Events (GSK Scale) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |
| 3.045 | All Treated | Mock-up<br>SAFE_T3 | Shift in Grade of Corneal Events (Overall GSK Scale) from Baseline to Week 13 (Arm A – GSK2857916 + Len/Dex (Rd)) | See Section 15.13 for mock | IA [2] |
| 3.046 | All Treated | Mock-up<br>SAFE_T3 | Shift in Grade of Corneal Events (Overall GSK Scale) from Baseline to Week 10 (Arm B – GSK2857916 + Bor/Dex (Vd)) | See Section 15.13 for mock | IA [3] |
| 3.047 | All Treated | Mock-up<br>SAFE_T3 | Shift in Grade of Corneal Events (Overall GSK Scale) from Baseline to End of Treatment (Arm A – GSK2857916 + Len/Dex (Rd)) | See Section 15.13 for mock | SAC [1] |
| 3.048 | All Treated | Mock-up<br>SAFE_T3 | Shift in Grade of Corneal Events (Overall GSK Scale) from Baseline to End of Treatment (Arm B – GSK2857916 + Bor/Dex (Vd)) | See Section 15.13 for mock | SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.049 | All Treated | AE17A | Summary of Exposure Adjusted Incidence Rates of Grade 3+ Corneal Events (Overall GSK Scale) (Arm A – GSK2857916 + Len/Dex (Rd)) | Only provide exposure adjusted rates for grade 3+ corneal events (using definition in Section 8.2.2). No subgroups needed. Only ANY EVENT. Delete the "Total PY" column. Only keep footnote [1] See Section 15.13 for mock Only create for IA2 if time allows | IA [2], SAC [1] |
| 3.050 | All Treated | AE17A | Summary of Exposure Adjusted Incidence Rates of<br>Grade 3+ Corneal Events (Overall GSK Scale) (Arm B<br>– GSK2857916 + Bor/Dex (Vd)) | Only provide exposure adjusted rates for grade 3+ corneal events (using definition in Section 8.2.2). No subgroups needed. Only ANY EVENT. Delete the "Total PY" column. Only keep footnote [1] See Section 15.13 for mock | IA [3], SAC [1] |
| 3.051 | All Treated | ESI1 | Summary of Characteristics of Corneal Events (CTCAE) (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock in Section 15.13 with categories and footnotes to include. Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], SAC [1] |
| 3.052 | All Treated | ESI1 | Summary of Characteristics of Corneal Events (CTCAE) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.053 | All Treated | AE13 | Corneal Event Overview (CTCAE) (Arm A – GSK2857916 + Len/Dex (Rd)) | - See mock in Section 15.13 with categories and footnotes to include. In shell, for rows that state "Lenalidomide/Bortezomib" – use "Lenalidomide" for Arm A. - For all categories use "corneal" AEs and "corneal "events" Use definition of on-treatment AEs as seen in Section 15.2.3 Add footnote: No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE | SAC [1] |
| 3.054 | All Treated | AE13 | Corneal Event Overview (CTCAE) (Arm B – GSK2857916 + Bor/Dex (Vd)) | - See mock in Section 15.13 with categories and footnotes to include. In shell, for rows that state "Lenalidomide/Bortezomib" – use "Bortezomib" for Arm B. - For all categories use "corneal" AEs and "corneal "events" Use definition of on-treatment AEs as seen in Section 15.2.3 Add footnote: No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE, and 2.5 mg/kg S/D STRETCH | IA [3], SAC [1] |

| Safety: Ta | Safety: Tables | | | | | | |
|---|---|---|---|---|---|--|--|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] | | |
| 3.055 | All Treated | OAE07 | Summary of Corneal Events (CTCAE) by Preferred<br>Term and Maximum Grade (Arm A – GSK2857916 +<br>Len/Dex (Rd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [2], SAC [1] | | |
| 3.056 | All Treated | OAE07 | Summary of Corneal Events (CTCAE) by Preferred<br>Term and Maximum Grade (Arm B – GSK2857916 +<br>Bor/Dex (Vd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [1], IA [3],<br>SAC [1] | | |
| 3.057 | All Treated | AE6 | Summary of Cumulative Incidence of Corneal Events (CTCAE) by Preferred Term and Number of Doses Received at First Occurrence (Arm A – GSK2857916 + Len/Dex (Rd)) | Only PT. The number of doses received at first occurrence will be <= 1, <= 2, <= 4, <= 6, <= 8, <= 10, and Any Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], SAC [1] | | |
| 3.058 | All Treated | AE6 | Summary of Cumulative Incidence of Corneal Events (CTCAE) by Preferred Term and Number of Doses Received at First Occurrence (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] | | |
| 3.059 | All Treated | ESI1 | Summary of Characteristics of Keratopathy Events (CTCAE) (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock in Section 15.13 with categories and footnotes to include. Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], SAC [1] | | |
| 3.060 | All Treated | ESI1 | Summary of Characteristics of Keratopathy Events (CTCAE) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above Also, add a footnote: For IDs 2, 3, 6 (Arm B 2.5 mg/kg SINGLE), total number of adverse events may be overreported due to a site related unfixable non-standard logging of ongoing events. | IA [1], IA [3],<br>SAC [1] | | |
| Safety: Ta | Safety: Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] | | | |
| 3.061 | All Treated | ESI1 | Summary of Characteristics of Blurred Vision Events (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock in Section 15.13 with categories and footnotes to include. Additional Footnote: Note: Blurred Vision events as collected in the AE eCRF, including MedDRA terms based on clinical review. Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], SAC [1] | | | |
| 3.062 | All Treated | ESI1 | Summary of Characteristics of Blurred Vision Events (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above Also, add a footnote: For IDs 2, 3, 6, total number of adverse events may be overreported due to a site related unfixable non-standard logging of ongoing events | IA [3], SAC [1] | | | |
| 3.063 | All Treated | ESI1 | Summary of Characteristics of Thrombocytopenia<br>(Arm A – GSK2857916 + Len/Dex (Rd)) | See mock in Section 15.13 with categories and footnotes to include. Use definition of on-treatment AEs as seen in Section 15.2.3 Add an additional footnote: Note: Thrombocytopenia events as collected in the AE eCRF, including MedDRA terms based on clinical review. | IA [2], SAC [1] | | | |
| 3.064 | All Treated | ESI1 | Summary of Characteristics of Thrombocytopenia (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] | | | |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.065 | All Treated | OAE07 | Summary of Thrombocytopenia by Preferred Term and Maximum Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [2], SAC [1] |
| 3.066 | All Treated | OAE07 | Summary of Thrombocytopenia by Preferred Term and Maximum Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [1], IA [3],<br>SAC [1] |
| 3.067 | All Treated | ESI2b | Summary of Onset and Duration of the First<br>Occurrence of Thrombocytopenia (Arm A –<br>GSK2857916 + Len/Dex (Rd)) | Time of onset: 1-28, 29-56, 57-84, >84. Duration: 1-28, 29-56, >56. Mean, SD, Median, Min, Max Use definition of on-treatment AEs as seen in Section 15.2.3 Footnotes: [1] Not Evaluable means the event outcome was 'NOT RECOVERED/NOT RESOLVED' or 'RECOVERING/RESOLVING' with no end date. Note: Time of onset assessed only for those subjects experiencing Thrombocytopenia. Note: Thrombocytopenia events as collected in the AE eCRF, including MedDRA terms based on clinical review. | IA [2], SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.068 | All Treated | ESI2b | Summary of Onset and Duration of the First<br>Occurrence of Thrombocytopenia (Arm B –<br>GSK2857916 + Bor/Dex (Vd)) | Time of onset: 1-21, 22-42, 43-63, >63. Duration: 1-21, 22-42, >42. Mean, SD, Median, Min, Max Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [1], IA [3],<br>SAC [1] |
| 3.069 | All Treated | AE6 | Summary of Cumulative Incidence of Thrombocytopenia by Preferred Term and Number of Doses Received at First Occurrence (Arm A – GSK2857916 + Len/Dex (Rd)) | Only PT. The number of doses received at first occurrence will be <= 1, <= 2, <= 4, <= 6, <= 8, <= 10, and Any Use definition of on-treatment AEs as seen in Section 15.2.3 Footnote: Note: Thrombocytopenia events as collected in the AE eCRF, including MedDRA terms based on clinical review. | SAC [1] |
| 3.070 | All Treated | AE6 | Summary of Cumulative Incidence of Thrombocytopenia by Preferred Term and Number of Doses Received at First Occurrence (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.071 | All Treated | SAFE_T11 | Summary of Thrombocytopenia and Bleeding Event (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of on-treatment AEs as seen in Section 15.2.3 Footnotes: [1] Lab data where Toxicity='Platelet count decreased' and Standard Toxicity Grade=3 or 4. [2] On-treatment Bleeding events include: Haemorrhage events as collected in the AE eCRF, including MedDRA terms based on clinical review; as well as Thrombocytopenia events as collected in the AE eCRF with 'Was there bleeding associated with the thrombocytopenia?'=Y, with Maximum Grade 2 or above. [3] Concomitant events are those from statement [1] and statement [2] that occur on the same day or within +/- 3 days and the event is on-treatment. | IA [2], SAC [1] |
| 3.072 | All Treated | SAFE_T11 | Summary of Thrombocytopenia and Bleeding Event (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.073 | All Treated | ESI1 | Summary of Characteristics of Infusion-Related Reactions (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock in Section 15.13 with categories and footnotes to include. Use definition of on-treatment AEs as seen in Section 15.2.3 Additional Footnote: Note: IRR events as collected in the AE eCRF, including MedDRA terms based on clinical review. | IA [2], SAC [1] |
| 3.074 | All Treated | ESI1 | Summary of Characteristics of Infusion-Related Reactions (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |
| 3.075 | All Treated | OAE07 | Summary of Infusion-Related Reactions by Preferred Term and Maximum Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [2], SAC [1] |
| 3.076 | All Treated | OAE07 | Summary of Infusion-Related Reactions by Preferred Term and Maximum Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [1], IA [3],<br>SAC [1] |
| 3.077 | All Treated | ESI1 | Summary of Characteristics of Neutropenia (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock in Section 15.13 with categories and footnotes to include. Use definition of on-treatment AEs as seen in Section 15.2.3 Additional Footnote: Note: Neutropenia events as collected in the AE eCRF, including MedDRA terms based on clinical review. | IA [2], SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.078 | All Treated | ESI1 | Summary of Characteristics of Neutropenia (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1],<br>SAC [1] |
| 3.079 | All Treated | OAE07 | Summary of Neutropenia by Preferred Term and Maximum Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | SAC [1] |
| 3.080 | All Treated | OAE07 | Summary of Neutropenia by Preferred Term and Maximum Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of treatment emergent AEs as seen in Section 15.2.3 | IA [1],<br>SAC [1] |
| 3.081 | All Treated | AE6 | Summary of Cumulative Incidence of Neutropenia by Preferred Term and Number of Doses Received at First Occurrence (Arm A – GSK2857916 + Len/Dex (Rd)) | Only PT. The number of doses received at first occurrence will be <= 1, <= 2, <= 4, <= 6, <= 8, <= 10, and Any Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.082 | All Treated | AE6 | Summary of Cumulative Incidence of Neutropenia by Preferred Term and Number of Doses Received at First Occurrence (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1],<br>SAC [1] |
| 3.083 | All Treated | SAFE_T11a | Summary of Neutropenia and Infection Event (Arm A – GSK2857916 + Len/Dex (Rd)) | Use definition of on-treatment AEs as seen in Section 15.2.3 | SAC [1] |
| 3.084 | All Treated | SAFE_T11a | Summary of Neutropenia and Infection Event (Arm B – GSK2857916 + Bor/Dex (Vd)) | Use definition of on-treatment AEs as seen in Section 15.2.3 | IA [1],<br>SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.085 | All Treated | ESI1 | Summary of Characteristics of Haematological Toxicity (Arm A – GSK2857916 + Len/Dex (Rd)) | *See mock shell in Section 15.13 for specifications Use definition of on-treatment AEs as seen in Section 15.2.3 Additional Footnote: Note: Haematological Toxicity events, identified using MedDRA terms based on clinical review. | IA [2], SAC [1] |
| 3.086 | All Treated | ESI1 | Summary of Characteristics of Haematological Toxicity (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above Also, add a footnote: For IDs 2, 3, 6, total number of adverse events may be overreported due to a site related unfixable non-standard logging of ongoing events. | IA [1], IA [3],<br>SAC [1] |
| Deaths | 1 | | | , - | |
| 3.087 | All Treated | DTH1a | Summary of Deaths (Arm A – GSK2857916 + Len/Dex (Rd)) | IDSL Include Subject Status, Primary Cause of Death, and Time to Death from Last Dose | IA [2], HDL [1], SAC [1] |
| 3.088 | All Treated | DTH1a | Summary of Deaths (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3], HDL [1],<br>SAC [1] |
| Laborator | Laboratory: Chemistry | | | | |
| 3.089 | All Treated | LB1 | Summary of Chemistry Changes from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3. | SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.090 | All Treated | LB1 | Summary of Chemistry Changes from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3. | SAC [1] |
| 3.091 | All Treated | OLB9B | Summary of Worst Case Chemistry Grade Changes from Baseline Grade (Arm A – GSK2857916 + Len/Dex (Rd)) | | SAC [1] |
| 3.092 | All Treated | OLB9B | Summary of Worst Case Chemistry Grade Changes from Baseline Grade (Arm B – GSK2857916 + Bor/Dex (Vd)) | | SAC [1] |
| 3.093 | All Treated | OLB11B | Summary of Worst Case Chemistry Changes from Baseline with Respect to the Normal Range (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | IA [2], SAC [1] |
| 3.094 | All Treated | OLB11B | Summary of Worst Case Chemistry Changes from Baseline with Respect to the Normal Range (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | IA [1], IA [3],<br>SAC [1] |
| Laborato | y: Haematoloզ | Jy | | | |
| 3.095 | All Treated | LB1 | Summary of Haematology Changes from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 3.096 | All Treated | LB1 | Summary of Haematology Changes from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| 3.097 | All Treated | OLB9B | Summary of Worst Case Haematology Grade<br>Changes from Baseline Grade (Arm A – GSK2857916<br>+ Len/Dex (Rd)) | | SAC [1] |
| 3.098 | All Treated | OLB9B | Summary of Worst Case Haematology Grade<br>Changes from Baseline Grade (Arm B – GSK2857916<br>+ Bor/Dex (Vd)) | | SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.099 | All Treated | OLB11B | Summary of Worst Case Haematology Changes from Baseline with Respect to the Normal Range (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | IA [2], SAC [1] |
| 3.100 | All Treated | OLB11B | Summary of Worst Case Haematology Changes from Baseline with Respect to the Normal Range (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | IA [1], IA [3],<br>SAC [1] |
| Laborator | y: Urinalysis | | | | |
| 3.101 | All Treated | LB1 | Summary of Urine Concentration Changes from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 3.102 | All Treated | LB1 | Summary of Urine Concentration Changes from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| 3.103 | All Treated | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 3.104 | All Treated | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| Laborator | y: Hepatobilia | ry (Liver) | | | |
| 3.105 | All Treated | LIVER1 | Summary of Liver Monitoring/Stopping Event<br>Reporting (Arm A – GSK2857916 + Len/Dex (Rd)) | IDSL | SAC [1] |
| 3.106 | All Treated | LIVER1 | Summary of Liver Monitoring/Stopping Event<br>Reporting (Arm B – GSK2857916 + Bor/Dex (Vd)) | IDSL | SAC [1] |
| 3.107 | All Treated | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities (Arm A – GSK2857916 + Len/Dex (Rd)) | IDSL | SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.108 | All Treated | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities (Arm B – GSK2857916 + Bor/Dex (Vd)) | IDSL | SAC [1] |
| ECG | | | | | |
| 3.109 | All Treated | OECG2B | Summary of Worst-case Amount of Increase from Baseline Value in Fridericia's QTc (Arm A – GSK2857916 + Len/Dex (Rd)) | Use same definition of "worst-case" as study 159 in Table 3.0392 (primary_02). Add categories as seen in Section 8.8 No "Planned Time" column is necessary. Add footnote to the "category" column: [2] Counts within categories may not add up to counts within 'n'. | IA [2], SAC [1] |
| 3.110 | All Treated | OECG2B | Summary of Worst-case Amount of Increase from Baseline Value in Fridericia's QTc (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |
| Vital Sign | s | | | | |
| 3.111 | All Treated | VS1 | Summary of Change from Baseline in Vital Signs (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 Add footnote: Note: 'BASELINE' visit displays actual Vital Signs at Baseline. Any post-baseline visit displays change from baseline in Vital Signs." | SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.112 | All Treated | VS1 | Summary of Change from Baseline in Vital Signs (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 Add footnote: Note: 'BASELINE' visit displays actual Vital Signs at Baseline. Any post-baseline visit displays change from baseline in Vital Signs." | SAC [1] |
| Dose Limi | iting Toxicity ( | DLT) | | | |
| 3.113 | All Treated | AE19 | Summary of Dose-Limiting Toxicities during the Determinative Period (Arm A – Part 1) | ICH E3 | SAC [1] |
| 3.114 | All Treated | DL1 | Summary of Dose-Limiting Toxicities during the Determinative Period (Arm B – Part 1) | ICH E3 | IA [1], IA [3],<br>SAC [1] |
| Ocular fin | dings for Gene | eral study (Baselin | e to Last follow-up) | | |
| 3.115 | All Treated | Programming<br>note | Summary of Best Corrected Visual Acuity Test (BCVA)<br>Scores (logMAR score) (Arm A – GSK2857916 +<br>Len/Dex (Rd)) | Use Table 3.0501 from BMA117159 (primary_01) study as template. Following "worst change from baseline', add summary for 'Most frequent Visual Acuity Change, and pick the worst category if there is tie. Under column 'Eye', in addition to Right/Left add 'Better' (better of two eye). Definition of 3 categories of change are same as in BMA117159 (primary_01). See Section 15.13 for mock and footnotes. | IA [2], SAC [1] |
| 3.116 | All Treated | Programming note | Summary of Best Corrected Visual Acuity Test (BCVA)<br>Scores (logMAR score) (Arm B – GSK2857916 +<br>Bor/Dex (Vd)) | Same as above | IA [1], Post-Interim [1],<br>IA [3],<br>SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.117 | All Treated | Programming<br>note | Summary of Best Corrected Visual Acuity Test (BCVA) Scores (logMAR score) due to Corneal Event (Arm A – GSK2857916 + Len/Dex (Rd)) | [1] Use Table 3.0501 from BMA117159 (primary_01) study as template. Following "worst change from baseline', add summary for 'Most frequent Visual Acuity Change, and pick the worst category if there is tie. Under column 'Eye', in addition to Right/Left add 'Better' (better of two eye). Definition of 3 categories of change are same as in BMA117159 (primary_01). Only include those visits with BCVA due to corneal event flag='Y'. See Section 15.13 for mock. | IA [2], SAC [1] |
| 3.118 | All Treated | Programming note | Summary of Best Corrected Visual Acuity Test (BCVA)<br>Scores (logMAR score) due to Corneal Event (Arm B –<br>GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |
| 3.119 | All Treated | Mock-up<br>SAFE_T8 | Number (%) of Subjects with a Decline in Best<br>Corrected Visual acuity (BCVA) to LP or NLP due to a<br>Corneal Event Anytime Post-Baseline (Arm A –<br>GSK2857916 + Len/Dex (Rd)) | Eye (R/L) and subject (either eye) Add footnote: 'n' denotes subjects who have any post-Baseline Best Corrected Visual acuity (BCVA) score, where the Visual Acuity is due to corneal findings. Categories displayed are only counting where 'Light Perception' or 'No Light Perception' was selected on the Non-Snellen Acuity item on the Visual Acuity (Best Corrected) eCRF, therefore may not add up to 'n'. | IA [2], SAC [1] |
| 3.120 | All Treated | Mock-up<br>SAFE_T8 | Number (%) of Subjects with a Decline in Best<br>Corrected Visual acuity (BCVA) to LP or NLP due to a<br>Corneal Event Anytime Post-Baseline (Arm B –<br>GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], Post-Interim [1],<br>IA [3],<br>SAC [1] |

| Safety: Ta | ables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.121 | All Treated | BCVACHANGE | Summary of Worst Post-Baseline Best Corrected Visual Acuity (BCVA) Change in Snellen Results (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock figure in Section 15.13 Groups for "Number of Lines Change from Baseline" (Better Eye, Worse Eye): Improved BCVA <= 2 Lines decline >= 3 Lines decline Add footnotes as seen in the mock figure. | IA [2], HDL [1], SAC [1] |
| 3.122 | All Treated | BCVACHANGE | Summary of Worst Post-Baseline Best Corrected Visual Acuity (BCVA) Change in Snellen Results (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [3], HDL [1], SAC [1] |
| 3.123 | All Treated | BCVACHANGE | Summary of Worst Post-Baseline Best Corrected Visual Acuity (BCVA) due to Corneal Event Change in Snellen Results (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock figure in Section 15.13 Groups for "Number of Lines Change from Baseline" (Better Eye, Worse Eye): Improved BCVA <= 2 Lines decline >= 3 Lines decline Add footnotes as seen in the mock figure. | IA [3], SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.124 | All Treated | BCVACHANGE | Summary of Worst Post-Baseline Best Corrected Visual Acuity (BCVA) due to Corneal Event Change in Snellen Results (Arm B – GSK2857916 + Bor/Dex (Vd)) | See mock figure in Section 15.13 Groups for "Number of Lines Change from Baseline" (Better Eye, Worse Eye): Improved BCVA <= 2 Lines decline >= 3 Lines decline Add footnotes as seen in the mock figure. | IA [3], SAC [1] |
| 3.125 | All Treated | Mock-up<br>SAFE_T9 | Shift in Corneal Epithelium Findings from Baseline to Worst Post-Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | By eye (R/L) and subject (worse eye). See<br>Section 8.5 Ocular findings from ophthalmic<br>exam for details. | IA [2], SAC [1] |
| 3.126 | All Treated | Mock-up<br>SAFE_T9 | Shift in Corneal Epithelium Findings from Baseline to Worst Post-Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | By eye (R/L) and subject (worse eye). See<br>Section 8.5 Ocular findings from ophthalmic<br>exam for details. | IA [1], Post-Interim [1],<br>IA [3],<br>SAC [1] |
| 3.127 | All Treated | Mock-up<br>SAFE_T14 | By eye (R/L) and subject (worse eye). See Section 8.5 Ocular findings from ophthalmic exam for details. Mock-up Summary of Findings for Punctate Keratopathy (Arm A | | IA [2], SAC [1] |
| 3.128 | All Treated | Mock-up<br>SAFE_T14 | Summary of Findings for Punctate Keratopathy (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], Post-Interim [1],<br>IA [3], SAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| Anti-Drug | nti-Drug Antibody | | | | |
| | | | | Use Table 3.0940 from Study 207495 (primary_01) study as template | |
| 3.129 | All Treated | IMM1 | Summary of Anti-GSK2857916 Antibody Results by Planned Time and Treatment (Arm A – GSK2857916 + Len/Dex (Rd)) | Table will be produced by each visit and present data as shown in the mock-shell. | AAC [1] |
| | | | | Do not include Conclusive and Inconclusive rows. And only keep Titer data if there are positive results. | |
| | | | | Use Table 3.0940 from Study 207495 (primary_01) study as template | |
| 3.130 | All Treated | All Treated IMM1 Planned Time and Treatment (Arm B – GSK2857916 present data + Bor/Dex (Vd)) Do not include rows. And or | Table will be produced by each visit and present data as shown in the mock-shell. | AAC [1] | |
| | | | | Do not include Conclusive and Inconclusive rows. And only keep Titer data if there are positive results. | |
| 3.131 | All Treated | | Summary of Neutralizing Anti-GSK2857916 Antibody<br>Results by Planned Time and Treatment (Arm A – | Use Table 3.0950 from Study 207495 (primary_01) study as template | AAC [1] |
| | | | GSK2857916 + Len/Dex (Rd)) | Table will be produced by each visit and present data as shown in the mock-shell. | |
| 3.132 | All Treated | IMM2 | Summary of Neutralizing Anti-GSK2857916 Antibody Results by Planned Time and Treatment (Arm B – | Use Table 3.0950 from Study 207495 (primary_01) study as template | AAC [1] |
| | | | GSK2857916 + Bor/Dex (Vd)) | Table will be produced by each visit and present data as shown in the mock-shell. | |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.133 | All Treated | IMM4 | GSK2857916 Immunogenicity Incidence and<br>Summary (Arm A – GSK2857916 + Len/Dex (Rd)) | Use Table 3.0955 from Study 207495 (primary_01) study as template Produce Transient and Persistent Rows if possible. Use definitions in the Immunogenicity Display Standard Text Document. | AAC [1] |
| 3.134 | All Treated | IMM4 | GSK2857916 Immunogenicity Incidence and Summary (Arm B – GSK2857916 + Bor/Dex (Vd)) Produce Transient and Persistent Rows if possible. Use definitions in the Immunogenicity Display Standard Text Document. | | AAC [1] |

| Safety: Ta | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | itle Programming Notes | | Deliverable [Priority] |
| Additiona | Tables | | | | |
| 3.137 | All Treated | AE13 | Adverse Event Overview for Non-Corneal Events (Arm A – GSK2857916 + Len/Dex (Rd)) | This table will be produced for all AEs that are not categorized as corneal events. See mock in Section 15.3 with categories and footnotes to include. In shell, for rows that state "Lenalidomide/Bortezomib" – use "Lenalidomide" for Arm A. Use definition of on-treatment AEs as seen in Section 15.2.3 Add footnote: No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE | SAC [1] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 3.138 | All Treated | AE13 | Adverse Event Overview for Non-Corneal Events (Arm B – GSK2857916 + Bor/Dex (Vd)) | This table will be produced for all AEs that are not categorized as corneal events. See mock in Section 15.13with categories and footnotes to include. In shell, for rows that state "Lenalidomide/Bortezomib" – use "Bortezomib" for Arm B. Use definition of on-treatment AEs as seen in Section 15.2.3 Add footnote: No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE, and 2.5 mg/kg S/D STRETCH | SAC [1] |

# 15.12.7. Safety Figures

| Safety | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |

| Safety | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Profile | Plot | | | | |
| 3.135 | All Treated | Programming<br>Note | Profile Plot for Subjects (Arm A – GSK2857916 + Len/Dex (Rd)) | See similar Figure 3.0031 from BCMA Study 205678 (primary_01). Make the max x-axis value equal to the max study treatment duration (days) for all subjects. Create for IA [2] if time allows | IA [2], SAC [1] |
| 3.136 | All Treated | Programming<br>Note | Profile Plot for Subjects (Arm B – GSK2857916 + Bor/Dex (Vd)) | See similar Figure 3.0031 from BCMA Study 205678 (primary_01). Make the max x-axis value equal to the max study treatment duration (days) for all subjects. Create for IA [3] if time allows | IA [1], IA [3],<br>SAC [1] |

## 15.12.8. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Paramet | ter | | | | |
| 4.001 | PK GSK2857916 | PK06 | Summary of Derived GSK2857916 (ADC) PK Parameters (Arm A – GSK2857916 + Len/Dex (Rd)) | PK06 with both transformed and untransformed values. Only display means, median, SD, and CVb if n ≥ 3, and only display visits up to Week 13 Day 8 for CEOI/CTROUGH Any concentration pk parameters for ADC/Tab will be reported at ug/mL and for cys-mcMMAF in ng/mL. For Ctrough, add the following footnote: "Ctrough for a dosing profile, represents the concentration prior to the next dose." For tlast, add the following footnote: "The dose reference for Tlast is the time since most recent dose" | AAC [1] |
| 4.002 | PK GSK2857916 | PK06 | Summary of Derived GSK2857916 (ADC) PK Parameters (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>AAC [1] |

| Pharmacok | kinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.003 | PK GSK2857916 | PK06 | Summary of Derived GSK2857916 (Total Antibody) PK Parameters (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | AAC [1] |
| 4.004 | PK GSK2857916 | PK06 | Summary of Derived GSK2857916 (Total Antibody) PK Parameters (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>AAC [1] |
| 4.005 | PK GSK2857916 | PK06 | Summary of Derived cys-mcMMAF PK Parameter (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | AAC [1] |
| 4.006 | PK GSK2857916 | PK06 | Summary of Derived cys-mcMMAF PK Parameter (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>AAC [1] |
| 4.007 | PK Lenalidomide<br>25mg | PK06 | Summary of Derived Lenalidomide 25mg PK Parameter (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | IA [2], AAC [1] |
| 4.008 | PK Lenalidomide<br>10mg | PK06 | Summary of Derived Lenalidomide 10mg PK Parameter (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | IA [2], AAC [1] |
| 4.009 | PK Bortezomib | PK06 | Summary of Derived Bortezomib PK Parameter (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above. Also, summarize by route (IV vs. SC) | IA [3], AAC [1] |
| 4.010 | PK GSK2857916 | PK13 | Listing of Derived GSK2857916 (ADC) PK Parameters (Untransformed) (Arm A – GSK2857916 + Len/Dex (Rd)) | Produce Listing by Treatment Add a column for "Actual Dose" and "Dose Number" to the listing. "Dose Number" column only applicable for ADC, Tab, cysmcMMAF. | AAC [1] |
| 4.011 | PK GSK2857916 | PK13 | Listing of Derived GSK2857916 (ADC) PK Parameters (Untransformed) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>AAC [1] |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4.012 | PK GSK2857916 | PK13 | Listing of Derived GSK2857916 (Total Antibody) PK Parameters (Untransformed) (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | AAC [1] |
| 4.013 | PK GSK2857916 | PK13 | Listing of Derived GSK2857916 (Total Antibody) PK Parameters (Untransformed) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3]<br>AAC [1] |
| 4.014 | PK GSK2857916 | PK13 | Listing of Derived cys-mcMMAF PK Parameters (Untransformed) (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | AAC [1] |
| 4.015 | PK GSK2857916 | PK13 | Listing of Derived cys-mcMMAF PK Parameters (Untransformed) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3]<br>AAC [1] |
| 4.016 | PK Lenalidomide<br>25mg | PK13 | Listing of Derived Lenalidomide 25mg PK Parameters (Untransformed) (Arm A – GSK2857916 + Len/Dex (Rd)) | Produce Listing by Treatment Dose Number column not applicable | IA [2], AAC [ |
| 4.017 | PK Lenalidomide<br>10mg | PK13 | Listing of Derived Lenalidomide 10mg PK Parameters (Untransformed) (Arm A – GSK2857916 + Len/Dex (Rd)) | Produce Listing by Treatment Dose Number column not applicable | IA [2], AAC |
| 4.018 | PK Bortezomib | PK13 | Listing of Derived Bortezomib PK Parameters (Untransformed) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Produce Listing by Treatment Also, add in column for Route (IV vs. SC Dose Number column not applicable | IA [3], AAC |

| Pharmacol | kinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.019 | PK GSK2857916 | PK01 | Summary of Plasma GSK2857916 (ADC) PK Concentration-<br>Time Data (Arm A – GSK2857916 + Len/Dex (Rd)) | By cohort Only display mean, median, and SD if n ≥ 3 | AAC [1] |
| 4.020 | PK GSK2857916 | PK01 | Summary of Plasma GSK2857916 (ADC) PK Concentration-<br>Time Data (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [3], AAC [1] |
| 4.021 | PK GSK2857916 | PK01 | Summary of Plasma GSK2857916 (Total Antibody) PK<br>Concentration-Time Data (Arm A – GSK2857916 + Len/Dex<br>(Rd)) | Same as above | AAC [1] |
| 4.022 | PK GSK2857916 | PK01 | Summary of Plasma GSK2857916 (Total Antibody) PK<br>Concentration-Time Data (Arm B – GSK2857916 + Bor/Dex<br>(Vd)) | Same as above | IA [3], AAC [1] |
| 4.023 | PK GSK2857916 | PK01 | Summary of Plasma cys-mcMMAF PK Concentration-Time Data (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | AAC [1] |
| 4.024 | PK GSK2857916 | PK01 | Summary of Plasma cys-mcMMAF PK Concentration-Time Data (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [3], AAC [1] |
| 4.025 | PK Lenalidomide<br>25mg | PK01 | Summary of Lenalidomide 25mg PK Concentration-Time Data (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | AAC [1] |
| 4.026 | PK Lenalidomide<br>10mg | PK01 | Summary of Lenalidomide 10mg PK Concentration-Time Data (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above | AAC [1] |
| 4.027 | PK Bortezomib | PK01 | Summary of Bortezomib PK Concentration-Time Data (Arm A – GSK2857916 + Len/Dex (Rd)) | Same as above<br>Also, summarize by route (IV vs.<br>SC) | IA [3], AAC [1] |

# 15.12.9. Pharmacokinetic Figures

| Pharmacoki | netic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Concentration | on | • | | | |
| 4.028 | PK<br>GSK2857916 | PK16 | Individual Plasma GSK2857916 (ADC) Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxx" | AAC [1] |
| 4.029 | PK<br>GSK2857916 | PK16 | Individual Plasma GSK2857916 (ADC) Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxx" | IA [1], IA [3],<br>AAC [1] |
| 4.030 | PK<br>GSK2857916 | PK16 | Individual Plasma cys-mcMMAF Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxx" | AAC [1] |
| 4.031 | PK<br>GSK2857916 | PK16 | Individual Plasma cys-mcMMAF Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxx" | IA [1], IA [3],<br>AAC [1] |
| 4.032 | PK<br>GSK2857916 | PK16 | Individual Plasma Total Antibody Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxx" | AAC [1] |
| 4.033 | PK<br>GSK2857916 | PK16 | Individual Plasma Total Antibody Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxx" | IA [3], AAC [1] |

| Pharmacoki | netic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.034 | PK Lenalidomide<br>25mg | PK16 | Individual Plasma Lenalidomide 25mg Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxxx" | IA [2], AAC [1] |
| 4.035 | PK Lenalidomide 10mg Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxx" | | IA [2], AAC [1] | | |
| 4.036 | PK Bortezomib | PK16 | Individual Plasma Bortezomib Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | In second title, add "Treatment" to include cohort for each subject: "Treatment = x.x mg/kg, Subject = xxxxxxx", also add route of administration (IV or SC) | IA [3], AAC [1] |
| 4.037 | PK<br>GSK2857916 | PK17 | Mean Plasma GSK2857916 (ADC) Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | AAC [1] |
| 4.038 | PK<br>GSK2857916 | PK17 | Mean Plasma GSK2857916 (ADC) Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Overlay mean lines for all doses on the same plot Only display mean line for treatment Groups with N≥3 | IA [1],<br>AAC [1] |
| 4.039 | PK<br>GSK2857916 | PK17 | Mean Plasma GSK2857916 (cys-mcMMAF) Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | AAC [1] |

| Pharmacoki | netic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.040 | PK<br>GSK2857916 | PK17 | Mean Plasma GSK2857916 (cys-mcMMAF) Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | IA [1],<br>AAC [1] |
| 4.041 | PK<br>GSK2857916 | PK17 | Mean Plasma GSK2857916 (Total Antibody) Concentration-<br>Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 +<br>Len/Dex (Rd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | AAC [1] |
| 4.042 | PK<br>GSK2857916 | PK17 | Mean Plasma GSK2857916 (Total Antibody) Concentration-<br>Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 +<br>Bor/Dex (Vd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | AAC [1] |
| 4.043 | PK<br>GSK2857916 | PK18 | Median Plasma GSK2857916 (ADC) Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | Overlay median lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | AAC [1] |
| 4.044 | PK<br>GSK2857916 | PK18 | Median Plasma GSK2857916 (ADC) Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Overlay median lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | IA [1], IA [3],<br>AAC [1] |
| 4.045 | PK<br>GSK2857916 | PK18 | Median Plasma GSK2857916 (cys-mcMMAF) Concentration-<br>Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 +<br>Len/Dex (Rd)) | Overlay median lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | AAC [1] |
| 4.046 | PK<br>GSK2857916 | PK18 | Median Plasma GSK2857916 (cys-mcMMAF) Concentration-<br>Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 +<br>Bor/Dex (Vd)) | Overlay median lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | IA [1], IA [3]<br>AAC [1] |

| Pharmacoki | netic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.047 | PK<br>GSK2857916 | PK18 | Median Plasma GSK2857916 (Total Antibody) Concentration-<br>Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 +<br>Len/Dex (Rd)) | Overlay median lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | AAC [1] |
| 4.048 | PK<br>GSK2857916 | PK18 | Median Plasma GSK2857916 (Total Antibody) Concentration-<br>Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 +<br>Bor/Dex (Vd)) | Overlay median lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | IA [3], AAC [1] |
| 4.049 | PK Lenalidomide<br>25mg | PK18 | Mean Plasma Lenalidomide 25mg Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | IA [2], AAC [1] |
| 4.050 | PK Lenalidomide<br>10mg | PK18 | Mean Plasma Lenalidomide 10mg Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | IA [2], AAC [1] |
| 4.051 | PK Lenalidomide<br>25mg | PK18 | Median Plasma Lenalidomide 25mg Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | IA [2], AAC [1] |
| 4.052 | PK Lenalidomide<br>10mg | PK18 | Median Plasma Lenalidomide 10mg Concentration-Time Plots (Linear and Semi-Log) (Arm A – GSK2857916 + Len/Dex (Rd)) | Overlay mean lines for all doses on<br>the same plot<br>Only display mean line for treatment<br>Groups with N≥3 | IA [2], AAC [1] |

| Pharmacoki | harmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.053 | PK Bortezomib | PK17 | Mean Plasma Bortezomib Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Overlay mean lines for all doses on the same plot Only display mean line for treatment Groups with N≥3 Add footnotes: Note: IV=Intravenous, SC=Subcutaneous. Note: LLQ= 0.1 ng/mL. Note: The initial bioanalytical method had a LLQ of 0.5 ng/mL. This method was updated with a LLQ of 0.1 ng/mL. Samples with <llq are="" concentration="" groups="" initial="" less="" method="" method.="" n="2" not="" note:="" or="" presented.<="" reanalyzed="" td="" the="" treatment="" updated="" were="" with=""><td>IA [3], AAC [1]</td></llq> | IA [3], AAC [1] |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4.054 | PK Bortezomib | PK18 | Median Plasma Bortezomib Concentration-Time Plots (Linear and Semi-Log) (Arm B – GSK2857916 + Bor/Dex (Vd)) | Overlay median lines for all doses on the same plot Only display mean line for treatment Groups with N≥3 Add footnotes: Note: IV=Intravenous, SC=Subcutaneous. Note: LLQ= 0.1 ng/mL. Note: The initial bioanalytical method had a LLQ of 0.5 ng/mL. This method was updated with a LLQ of 0.1 ng/mL. Samples with <llq are="" concentration="" groups="" initial="" less="" method="" method.="" n="2" not="" note:="" or="" presented.<="" reanalyzed="" td="" the="" treatment="" updated="" were="" with=""><td>IA [3], AAC [1]</td></llq> | IA [3], AAC [1] |
| Cmax Plots | | | | | |
| 4.055 | PK<br>GSK2857916 | Mock-up<br>PK_1 | Individual and Mean Cmax by Dose/Schedule and Day for Cycle 1 – ADC (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock figure in Section 15.13 | AAC [1] |
| 4.056 | PK<br>GSK2857916 | Mock-up<br>PK_1 | Individual and Mean Cmax by Dose/Schedule and Day for Cycle 1 – ADC (Arm B – GSK2857916 + Bor/Dex (Vd)) | See mock figure in Section 15.13 | IA [1], IA [3],<br>AAC [1] |
| 4.057 | PK<br>GSK2857916 | Mock-up<br>PK_1 | Individual and Mean Cmax by Dose/Schedule and Day for Cycle 1 – cys-mcMMAF (Arm A – GSK2857916 + Len/Dex (Rd)) | See mock figure in Section 15.13 | AAC [1] |
| 4.058 | PK<br>GSK2857916 | Mock-up<br>PK_1 | Individual and Mean Cmax by Dose/Schedule and Day for Cycle 1 – cys-mcMMAF (Arm B – GSK2857916 + Bor/Dex (Vd)) | See mock figure in Section 15.13 | IA [1], IA [3],<br>AAC [1] |

| Pharmacoki | harmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.059 | PK<br>GSK2857916 | Mock-up<br>PK_1 | See mod | See mock figure in Section 15.13 | AAC [1] |
| 4.060 | PK<br>GSK2857916 | Mock-up<br>PK_1 | Individual and Mean Cmax by Dose/Schedule and Day for Cycle 1 – Total Antibody (Arm B – GSK2857916 + Bor/Dex (Vd)) | See mock figure in Section 15.13 | IA [3], AAC [1] |

## 15.12.10. Biomarker Tables

| Bioma | arker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

| Bioma | Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

# 15.12.11. Biomarker Figures

| Bioma | Biomarker: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |

| Biomarker: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |

# 15.12.12. Patient Reported Outcomes Tables

| No. | Population | IDSL / Example | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| NO. | Population | Shell | Title | Programming Notes | [Priority] |
| PRO-C | TCAE | | | | |
| 6.001 | All Treated | PRO_MAX | Summary of Maximum Post-Baseline PRO-CTCAE Score (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Refer to mid205678 (primary_01) Table 8.0090 for guidance. For each selected item from PRO-CTCAE library: create summary table for maximum post-baseline PRO-CTCAE score for each of 3 attributes (frequency, severity and/or interference). Presence/Absence will only be listed. | [1] |
| 6.002 | All Treated | PRO_MAX | Summary of Maximum Post-Baseline PRO-CTCAE Score (Arm B – GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Refer to mid205678 (primary_01) Table 8.0090 for guidance. For each selected item from PRO-CTCAE library: create summary table for maximum post-baseline PRO-CTCAE score for each of 3 attributes (frequency, severity and/or interference). Presence/Absence will only be listed. | AAC [1] |
| OSDI | | | | | |
| 6.003 | All Treated | OSDI_CHG_TOT | Summary of Change in OSDI Total Scores from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Refer to mid205678 (primary_01) Table 8.00130 for guidance. | AAC [1] |
| 6.004 | All Treated | OSDI_CHG_TOT | Summary of Change in OSDI Total Scores from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Refer to mid205678 (primary_01) Table 8.00130 for guidance. | AAC [1] |

| Patien | Patient Reported Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.005 | All Treated | OSDI_CHG_SUB | Summary of Change in OSDI Subscale Scores from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Refer to mid205678 (primary_01) Table 8.00130 for guidance. | AAC [1] |
| | | | | Descriptive stats + frequencies of worsening >=12.5 (VRF). Refer to mid207503 (internal_02) Table 5.11 for guidance on VRF 12.5 worsening. | |
| 6.006 | All Treated | OSDI_CHG_SUB | Summary of Change in OSDI Subscale Scores from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Refer to mid205678 (primary_01) Table 8.00130 for guidance. | AAC [1] |
| | | | | Descriptive stats + frequencies of worsening >=12.5 (VRF). Refer to mid207503 (internal_02) Table 5.11 for guidance on VRF 12.5 worsening. | |

| Patien | Patient Reported Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.007 | All Treated | OSDI_DET | Summary of Patients with a 12.5 Point or Greater Deterioration from Baseline in the Visual Related Function Subscale Score (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Refer to mid205207 (primary_03) Table 6.0003for guidance. Include the following footnotes: (1) Improvement is defined as a decrease from the worst subscale score of at least 12.5 points. (2) Time to 12.5 point deterioration assessed only for those subjects experiencing a first worsening of at least one 12.5 unit as compared to the baseline score with complete onset date. (3) Duration is defined as time from the onset of first worsening of at least one 12.5 unit as compared to the baseline score to the first time of resolution based on 12.5 improvement from the first worst subscale score during the event. It requires at least one day gap between the resolution of worsening from first course to the onset of second course. | AAC [1] |

| Patien | Patient Reported Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.008 | All Treated | OSDI_DET | Summary of Patients with a 12.5 Point or Greater Deterioration from Baseline in the Visual Related Function Subscale Score (Arm B– GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Refer to mid205207 (primary_03) Table 6.0003 for guidance. Include the following footnotes: (1) Improvement is defined as a decrease from the worst subscale score of at least 12.5 points. (2) Time to 12.5 point deterioration assessed only for those subjects experiencing a first worsening of at least one 12.5 unit as compared to the baseline score with complete onset date. (3) Duration is defined as time from the onset of first worsening of at least one 12.5 unit as compared to the baseline score to the first time of resolution based on 12.5 improvement from the first worst subscale score during the event. It requires at least one day gap between the resolution of worsening from first course to the onset of second course. | AAC [1] |
| NEI-VFQ-25 | | | | | |
| 6.009 | All Treated | VFQ_CHG | Summary of Change in NEI-VFQ-25 Overall Composite Scores from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Timepoints includes EOT visit, last follow-up visit, and worst change from baseline. | AAC [1] |
| 6.010 | All Treated | VFQ_CHG | Summary of Change in NEI-VFQ-25 Overall Composite Scores from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Timepoints includes EOT visit, last follow-up visit, and worst change from baseline. | AAC [1] |
| Patien | Patient Reported Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.011 | All Treated | VFQ_CHG | Summary of Change in NEI-VFQ-25 Subscale Scores from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Timepoints includes EOT visit, last follow-up visit, and worst change from baseline. | AAC [1] |
| 6.012 | All Treated | VFQ_CHG | Summary of Change in NEI-VFQ-25 Subscale Scores from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Timepoints includes EOT visit, last follow-up visit, and worst change from baseline. | AAC [1] |
| EORT | C QLQ-C30 | | | | |
| 6.013 | All Treated | QLQ_CHG_DOM | Summary of Change in EORTC QLQ-C30 Domain Scores from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_01) Table 8.0020 for guidance. Including score for 15 domains and Improvement in EORTC QLQ-C30 domain score >=10 | AAC [1] |
| 6.014 | All Treated | QLQ_CHG_DOM | Summary of Change in EORTC QLQ-C30 Domain Scores from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_01) Table 8.0020 for guidance. Including score for 15 domains and Improvement in EORTC QLQ-C30 domain score >=10 | AAC [1] |
| EORT | C QLQ-MY20 | | | | |
| 6.015 | All Treated | QLQ_CHG_DOM | Summary of Change in EORTC QLQ-MY20 Domain Scores from Baseline (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_01) Table 8.0070 for guidance. Including score for 4 domains and Improvement in EORTC QLQ-MY20 domain score >=10 | AAC [1] |
| 6.016 | All Treated | QLQ_CHG_DOM | Summary of Change in EORTC QLQ-MY20 Domain Scores from Baseline (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_01) Table 8.0070 for guidance. Including score for 4 domains and Improvement in EORTC QLQ-MY20 domain score >=10 | AAC [1] |


| Patien | Patient Reported Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Compl | Compliance of PRO-CTCAE, OSDI, and EORTC QLQ-C30 | | | | |

| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.017 | All Treated | COMP1 | Summary of Compliance of PRO CTCAE, NEI-VFQ-25, and OSDI by Visit and Overall (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Refer to mid205678 (primary_07) Table 8.10010 for guidance. Include number and percentage of subjects for each assessment. Add "Overall" Compliance to bottom of table, representing compliance over all visits. Footnotes: Note: Percentage is calculated using # of subjects remaining in the study at given timepoint as denominator. Note: Subjects are counted as remaining in the study at last follow-up visit if they have at least one recorded follow-up visit. Note: Last Follow-up visit is not collected for PRO-CTCAE. Subjects who show corneal signs per the GSK scale at EOT will continue to receive only the OSDI and NEI-VFQ-25 assessments during follow-up for up to 1 year or until ocular exams are completed (whichever comes first). Note: The overall compliance rate is the number of subjects with an evaluable baseline score and at least one evaluable post-baseline score. | AAC [1] |

| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.018 | All Treated | COMP1 | Summary of Compliance of PRO CTCAE, NEI-VFQ-25, and OSDI by Visit and Overall (Arm B – GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Refer to mid205678 (primary_07) Table 8.10010 for guidance. Include number and percentage of subjects for each assessment. Add "Overall" Compliance to bottom of table, representing compliance over all visits. Footnote: Note: percentage is calculated using # of subject remaining in the study at given timepoint as denominator. | AAC [1] |
| 6.019 | All Treated | COMP2 | Summary of Compliance of EORTC QLQ-C30 and EORTC QLQ-MY20 by Visit and Overall (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_07) Table 8.10010 for guidance. Include number and percentage of subjects for each assessment. Add "Overall" Compliance to bottom of table, representing compliance over all visits. Footnote: Note: Percentage is calculated using # of subjects remaining in the study at given timepoint as denominator. Note: The overall compliance rate is the number of subjects with an evaluable baseline score and at least one evaluable post-baseline score. | AAC [1] |

| Patien | Patient Reported Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.020 | All Treated | COMP2 | Summary of Compliance of EORTC QLQ-C30 and EORTC QLQ-MY20 by Visit and Overall (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_07) Table 8.10010 for guidance. Include number and percentage of subjects for each assessment. Add "Overall" Compliance to bottom of table, representing compliance over all visits. Footnote: Note: percentage is calculated using # of subject remaining in the study at given timepoint as denominator. | AAC [1] |

# 15.12.13. Patient Reported Outcomes Figures

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PRO-CTC | AE | | | | |
| 6.021 | All Treated | PRO_STACK | Stacked Bar Chart of PRO-CTCAE Score by Attributes and Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Refer to mid205207 (primary_03) Figure 6.0001 for guidance. For each selected item from PRO-CTCAE library: create 5 sets of stacked bar charts per dose cohort for PRO-CTCAE score for each of 3 attributes (frequency, severity and/or interference). | AAC [1] |
| 6.022 | All Treated | PRO_STACK | Stacked Bar Chart of PRO-CTCAE Score by Attributes and Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Refer to mid205207 (primary_03) Figure 6.0001 for guidance. For each selected item from PRO-CTCAE library: create 5 sets of stacked bar charts per dose cohort for PRO-CTCAE score for each of 3 attributes (frequency, severity and/or interference). | AAC [1] |

| ratient h | Reported Outco | nnes: rigures | | | T |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| OSDI | | | | | |
| 6.023 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of OSDI<br>Total Score by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | Summarize by: dose level. Refer to mid205678 (primary_07) Figure 8.10023, 8.10024 & 8.10025 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, worst case post treatment and last follow-up visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note: Interval shown represents 95% confident limits around mean at each planned time. Note: BSLN = "Baseline", EOT = "End of Treatment", LFU = "Last Follow-Up", and WCPB = "Worst Case Post-Baseline". Note: Confidence Intervals are presented where n>=3. | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.024 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of OSDI Total Score by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Summarize by: dose level. Refer to mid205678 (primary_07) Figure 8.10023, 8.10024 & 8.10025 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, worst case post treatment and last follow-up visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| EORTC Q | LQ-C30 | | | | |
| 6.025 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Pain Domain Score by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_07) Figure 8.10037 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.026 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Pain Domain Score by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_07) Figure 8.10037 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient Ro | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.027 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Fatigue Domain Score by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_07) Figure 8.10038 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Post-baseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.028 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Fatigue Domain Score by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_07) Figure 8.10038 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.029 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Global Health Status / QoL Domain Score by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_07) Figure 8.10039 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.030 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Global Health Status / QoL Domain Score by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_07) Figure 8.10039 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | eported Outco | | | , | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.031 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Physical Functioning Domain Score by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_07) Figure 8.10037 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.032 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Physical Functioning Domain Score by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_07) Figure 8.10037 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.033 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Role Functioning Domain Score by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_07) Figure 8.10037 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.034 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-C30 Role Functioning Domain Score by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_07) Figure 8.10037 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | AAC [1] |

| Patient R | eported Outco | mes: Figures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| EORTC Q | LQ-MY20 | | | | |
| 6.035 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-MY20 Disease Symptom Domain Score by Visit (Arm A – GSK2857916 + Len/Dex (Rd)) | Refer to mid205678 (primary_07) Figure 8.10037 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | SAC [1] |

| Patient R | Patient Reported Outcomes: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.036 | All Treated | CFB_CI | Plot of Change from Baseline and Confidence Interval of EORTC QLQ-MY20 Disease Symptom Domain Score by Visit (Arm B – GSK2857916 + Bor/Dex (Vd)) | Refer to mid205678 (primary_07) Figure 8.10037 for guidance. Add a dashed line at y axis=0. In addition to treatment visits, also include end of treatment, and worst case post baseline visits. Add arrows showing direction of change from baseline: "deterioration" "improvement". Add the following footnotes: Note 1: Interval shown represents 95% confident limits around mean at each planned time. Note 2: "BSLN" represents "Baseline"; "EOT" represents "End of Treatment"; "WCPB" represents "Worst Case Postbaseline"; "LFU" represents "Last Follow-up". | SAC [1] |

### 15.12.14. ICH Listings

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.001 | All Treated | ES3 | Listing of Reasons for Study Withdrawal (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 Add footnotes: [1] y = years [2] Study Day is calculated as the number of days from the first dose date. | IA [2], SAC [1] |
| 1.002 | All Treated | ES3 | Listing of Reasons for Study Withdrawal (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |
| 1.003 | All Treated | SD2 | Listing of Reasons for Study Treatment Discontinuation (Arm A – GSK2857916 + Len/Dex (Rd)) | *Add a column for "Treatment" – see shell in Section 15.13 Add footnotes: [1] y = years [2] Study Day is calculated as the number of days from the first dose date. | IA [2], SAC [1] |
| 1.004 | All Treated | SD2 | Listing of Reasons for Study Treatment Discontinuation (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above | IA [1], IA [3],<br>SAC [1] |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protoco | l Deviations | | | | |
| 1.005 | All Treated | DV2 | Listing of Important Protocol Deviations (Arm A – GSK2857916 + Len/Dex (Rd)) | *Do not need last 3 columns titled "Deviation Requires Exclusion From" Add footnote: Note: Study Day is calculated as the number of days from the first dose date. | SAC [1] |
| 1.006 | All Treated | DV2 | Listing of Important Protocol Deviations (Arm B – GSK2857916 + Bor/Dex (Vd)) | *Do not need last 3 columns titled "Deviation Requires Exclusion From" Add footnote: Note: Study Day is calculated as the number of days from the first dose date. | IA [1],<br>SAC [1] |
| 1.007 | All Treated | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | RAPIDO DV at<br>SAC [1] |
| 1.008 | All Treated | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | RAPIDO DV at<br>SAC [1] |
| Demog | raphic and Basel | ine Character | istics | | |
| 1.009 | All Treated | DM2 | Listing of Demographic Characteristics (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.010 | All Treated | DM2 | Listing of Demographic Characteristics (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| Prior an | d Concomitant N | Medications | | | |
| 1.011 | All Treated | CM3 | Listing of Concomitant Medications (Arm A – GSK2857916 + Len/Dex (Rd)) | IDSL | SAC [1] |
| 1.012 | All Treated | CM3 | Listing of Concomitant Medications (Arm B – GSK2857916 + Bor/Dex (Vd)) | IDSL | SAC [1] |
| Exposu | re and Treatmen | t Compliance | | | |
| 1.013 | All Treated | OEX8A | Listing of Exposure Data (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 1.014 | All Treated | OEX8A | Listing of Exposure Data (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| Respon | se | | | | |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CI | | | | | |
| ı | | | | | |
| Adverse | e Events | r | | | |
| | | | | ICH E3 | |
| 1.017 | All Treated | AE8 | Listing of All Adverse Events (Arm A – GSK2857916 + Len/Dex (Rd)) | Add a footnote: - Time since 1st dose is the duration from the 1st dose of GSK2857916 to the start of the adverse event. Time since last dose is the duration since the latest dose taken (of any study treatment component) to the start of the adverse event. | IA [2], SAC [1] |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.018 | All Treated | AE8 | Listing of All Adverse Events (Arm B – GSK2857916 + Bor/Dex (Vd)) | Same as above Add an additional footnote: For IDs 2, 3, 6 (Arm B 2.5 mg/kg SINGLE) total number of adverse events may be overreported due to a site related unfixable non-standard logging of ongoing events. | IA [1], IA [3],<br>SAC [1] |
| 1.019 | All Treated | AE7 | Listing of Subject Numbers for Individual Adverse Events (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | RAPIDO DV at<br>SAC [1] |
| 1.020 | All Treated | AE7 | Listing of Subject Numbers for Individual Adverse Events (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | RAPIDO DV at<br>SAC [1] |
| Serious | Serious and Other Significant Adverse Events | | | | |
| 1.021 | All Treated | AE8 | Listing of Fatal Serious Adverse Events (Arm A – GSK2857916 + Len/Dex (Rd)) | | IA [2], SAC [1] |
| 1.022 | All Treated | AE8 | Listing of Fatal Serious Adverse Events (Arm B – GSK2857916 + Bor/Dex (Vd)) | | IA [1], IA [3],<br>SAC [1] |
| 1.023 | All Treated | AE8 | Listing of Non-Fatal Serious Adverse Events (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 1.024 | All Treated | AE8 | Listing of Non-Fatal Serious Adverse Events (Arm B – GSK2857916 + Bor/Dex (Vd)) | | SAC [1] |
| 1.025 | All Treated | AE14 | Listing of Reasons for Considering as a Serious Adverse Event (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 1.026 | All Treated | AE14 | Listing of Reasons for Considering as a Serious Adverse Event (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Labo | oratory | | | | |
| 1.027 | All Treated | LB5A | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 1.028 | All Treated | LB5A | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| 1.029 | All Treated | LB14 | Listing of Laboratory Data with Character Results (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | SAC [1] |
| 1.030 | All Treated | LB14 | Listing of Laboratory Data with Character Results (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | SAC [1] |
| 1.031 | All Treated | UR2 | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance (Arm A – GSK2857916 + Len/Dex (Rd)) | ICH E3 | RAPIDO DV at<br>SAC [1] |
| 1.032 | All Treated | UR2 | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance (Arm B – GSK2857916 + Bor/Dex (Vd)) | ICH E3 | RAPIDO DV at<br>SAC [1] |
| Death | | | | | |
| 1.033 | All Treated | DD2 | Listing of Subject Numbers for Specific Causes of Deaths (Arm A – GSK2857916 + Len/Dex (Rd)) | | SAC [1] |
| 1.034 | All Treated | DD2 | Listing of Subject Numbers for Specific Causes of Deaths (Arm B – GSK2857916 + Bor/Dex (Vd)) | | IA [3], SAC [1] |

### 15.12.15. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protocol Deviations | | | | | |
| 30.001 | All Treated | PAN7 | Listing of Visits Impacted by COVID-19 Pandemic (Arm A – GSK2857916 + Len/Dex (Rd)) | | RAPIDO DV at<br>SAC [1] |
| 30.002 | All Treated | PAN7 | Listing of Visits Impacted by COVID-19 Pandemic (Arm B – GSK2857916 + Bor/Dex (Vd)) | | RAPIDO DV at<br>SAC [1] |

| Non-ICH: List | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposure | | <u> </u> | | | 1 |
| 30.003 | All Treated | OEX9 | Summary Listing of Overall Exposure and Dose Modifications (Arm A – GSK2857916 + Len/Dex (Rd)) | *Add Site ID, Subject ID, Component, Time on Study Treatment, Dose Intensity, and Dose Modification Summary *We do not need the "X Missed Doses" category under "Dose Modification Summary" *Add footnotes (for correct order see annotated shells): [1] Dose intensity (units/interval) is the cumulative actual dose divided by duration of exposure, where interval is 4 weeks for SINGLE and SPLIT dosing, and 8 weeks for STRETCH dosing. For dose intensity, date of discontinuation is the date of last dose. For Arm A, each cycle is 4 weeks (28 days) No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE | IA [2], SAC [1] |

| Non-ICH: List | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 30.004 | All Treated | OEX9 | Summary Listing of Overall Exposure and Dose Modifications (Arm B – GSK2857916 + Bor/Dex (Vd)) | *Add Site D, Subject ID, Component, Time on Study Treatment, Dose Intensity, and Dose Modification Summary *We do not need the "X Missed Doses" category under "Dose Modification Summary" *Add footnotes (for correct order see annotated shells): [1] Dose intensity (units/interval) is the cumulative actual dose divided by duration of exposure, where interval is 3 weeks for SINGLE/SPLIT doses and 6 weeks for STRETCH and S/D STRETCH doses. [2] Dose Intensity for BOR and DEX calculated per day within a cycle for Bortezomib. For Arm B, each cycle is 3 weeks (21 days) No dose reduction of GSK2857916 allowed for 1.9 mg/kg STRETCH and SINGLE, and 2.5 mg/kg S/D STRETCH | IA [1], IA [3],<br>SAC [1] |
| Anti-Drug Ant | tibody | | | | • |
| 30.005 | All Treated | IMM5 | Listing of GSK2857916 Immunogenicity Results (Arm A – GSK2857916 + Len/Dex (Rd)) | | RAPIDO DV at AAC [1] |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 30.006 | All Treated | IMM5 | Listing of GSK2857916 Immunogenicity Results (Arm B – GSK2857916 + Bor/Dex (Vd)) | | RAPIDO DV at<br>AAC [1] |
| PK | | | | | |
| 30.007 | PK GSK2857916 | PK13 | Listing of GSK2857916 (ADC, Total Antibody, cys-mcMMAF) Pharmacokinetic Concentration-Time Data (Arm A – GSK2857916 + Len/Dex (Rd)) | Produce Listing by Treatment | AAC [1] |
| 30.008 | PK GSK2857916 | PK13 | Listing of GSK2857916 (ADC, Total Antibody, cys-mcMMAF) Pharmacokinetic Concentration-Time Data (Arm B – GSK2857916 + Bor/Dex (Vd)) | Produce Listing by Treatment | AAC [1] |
| 30.009 | PK Lenalidomide<br>25mg | PK13 | Listing of Lenalidomide Pharmacokinetic Concentration-Time<br>Data (Arm A – GSK2857916 + Len/Dex (Rd)) | Produce Listing by Treatment Can delete "dose number" from listing | AAC [1] |
| 30.010 | PK Lenalidomide<br>10mg | PK13 | Listing of Lenalidomide Pharmacokinetic Concentration-Time<br>Data (Arm A – GSK2857916 + Len/Dex (Rd)) | Produce Listing by Treatment Can delete "dose number" from listing | AAC [1] |
| 30.011 | PK Bortezomib | PK13 | Listing of Bortezomib Pharmacokinetic Concentration-Time<br>Data (Arm B – GSK2857916 + Bor/Dex (Vd)) | Produce Listing by Treatment Can delete "dose number" from listing Add column for "Route" | AAC [1] |

## 15.13. Appendix 13: Example Mock Shells for Data Displays

Mock shells will be available within a RAP Supportive Document. This RAP Supportive Document will contain the final templates applied for final SAC.

#### Signature Page for $\,207497\,TMF-16085540\,v1.0\,$

| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 25-Apr-2023 15:48:45 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 25-Apr-2023 16:02:53 GMT+0000 |

Signature Page for TMF-16085540 v1.0